

## STATISTICAL ANALYSIS PLAN

A PHASE 3, DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, PARALLEL-GROUP, 27-WEEK TRIAL TO EVALUATE THE EFFICACY, SAFETY, AND TOLERABILITY OF TWO FIXED DOSES OF TAVAPADON IN EARLY PARKINSON'S DISEASE (TEMPO-1 TRIAL)

Protocol Number: CVL-751-PD-001

**Compound: Tavapadon (CVL-751)** 

**Trial Phase: 3** 

Short Title: Fixed-Dose Trial in Early Parkinson's Disease

**Sponsor Name: Cerevel Therapeutics, LLC** 

**Protocol Version:** Version 4.0 Date: 06 Jul 2023

Version 3.0 03 Sep 2021 Version 2.0 29 Jun 2020

Original Version 1.0 Date: 07 Oct 2019

**Analysis Plan Version:** Final 1.0: 31 July 2024



# STATISTICAL ANALYSIS PLAN REVIEW AND APPROVAL

This Statistical Analysis Plan has been prepared in accordance with team reviewers' specifications.

| Prepared by: O2-Aug-2024 12:06 EDT Biostatistics PharPoint Research, Inc. Approved by: | | |
|---|---|---|
| Biostatistics PharPoint Research, Inc. | Prepared by: | |
| Biostatistics PharPoint Research, Inc. | | |
| Biostatistics PharPoint Research, Inc. | | |
| Biostatistics PharPoint Research, Inc. | | |
| Biostatistics PharPoint Research, Inc. | | |
| Biostatistics PharPoint Research, Inc. | | 02 40- 2024 12-06 507 |
| PharPoint Research, Inc. | | 02-AUG-2024 12:06 EDI |
| | Biostatistics | Date |
| Approved by: | PharPoint Research, Inc. | |
| Approved by: | | |
| | Approved by: | |



PharPoint Research, Inc.

Date

# Approved by:



Global Clinical Development Cerevel Therapeutics, LLC



Cerevel Therapeutics, LLC



# **TABLE OF CONTENTS**

| STATIST | TICAL ANALYSIS PLAN | 1 |
|---|---|---|
| STATIST | TICAL ANALYSIS PLAN REVIEW AND APPROVAL | 2 |
| TABLE ( | OF CONTENTS | 4 |
| LIST OF | TABLES | 9 |
| LIST OF | FIGURES | 10 |
| 1. | INTRODUCTION | 11 |
| 1.1. | Study Overview | 11 |
| 1.2. | Sample Size Considerations | 12 |
| 1.3. | Measures to Minimize Bias: Randomization and Blinding | 12 |
| 1.3.1. | Subject Assignment to Treatment | 12 |
| 1.3.2. | Blinding | 12 |
| 1.4. | Treatment Period | 12 |
| 2. | OBJECTIVES AND ENDPOINTS | 14 |
| 3. | KEY ASSESSMENTS AND DERIVATIONS | 15 |
| 3.1. | Efficacy Assessments | 15 |
| 3.1.1. | Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 15 |
| 3.1.1.1. | Part I Score | 15 |
| 3.1.1.2. | Part II Score | 15 |
| 3.1.1.3. | Part III Score | 15 |
| 3.1.1.4. | Handling of Missing Items from MDS-UPDRS | 15 |
| 3.1.1.5. | Part II + III Combined Score | 16 |
| 3.1.1.6. | Part I, Part II, and Part III Combined Score | 16 |
| 3.1.2. | Patient Global Impression of Change (PGIC) | |
| 3.1.3. | Clinical Global Impression – Severity of Illness (CGI-S) | 16 |
| 3.1.4. | Clinical Global Impression – Improvement (CGI-I) | 16 |
| 3.1.5. | 39-Item Parkinson's Disease Questionnaire (PDQ-39) Score | 17 |
| 3.1.6. | EuroQol 5 Dimension 5 Level | 17 |
| 3.1.7. | Schwab and England Activities of Daily Living (ADL) Scale | 18 |
| 3.2. | Safety Assessments | 18 |



| 3.2.1. | Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease Rating Scale (QUIP-RS) Scores | 18 |
|---|---|---|
| 3.2.2. | Epworth Sleepiness Scale (ESS) Total Score | 19 |
| 3.2.3. | Adverse Event (AE) | 19 |
| 3.2.3.1. | Adverse Event of Special Interest (AESI) | 19 |
| 3.2.3.2. | Treatment-emergent Adverse Event (TEAE) | |
| 3.2.4. | Clinical Safety Laboratory Assessments | 20 |
| 3.2.4.1. | Treatment-emergent Laboratory Abnormality and Toxicity | 20 |
| 3.2.5. | Columbia-Suicide Severity Rating Scale (C-SSRS) | 20 |
| 3.2.6. | Vital Signs | 21 |
| 3.2.7. | Electrocardiograms | 21 |
| 3.2.8. | Prior Medications, Concomitant Medications and Medications Taken Post Last Dose of IMP | 21 |
| 3.2.9. | Physical and Neurological Examinations | 22 |
| 3.2.10. | Eye Examinations | 22 |
| 3.3. | Pharmacokinetics | 22 |
| 4. | DATA CONVENTIONS AND VISIT WINDOWS | 23 |
| 4.1. | Data Conventions | 23 |
| 4.1.1. | Age | 23 |
| 4.1.2. | Day 1 | 23 |
| 4.1.3. | Endpoint | 23 |
| 4.1.4. | Study Day of an Event | 23 |
| 4.1.5. | Days on Study | 23 |
| 4.1.6. | Days on IMP | 23 |
| 4.1.7. | Baseline Value | 23 |
| 4.1.8. | Change from Baseline | 24 |
| 4.1.9. | Orthostatic Change | 24 |
| 4.1.10. | Duration of Titration Phase | 24 |
| 4.1.11. | Duration of Maintenance Phase | 24 |
| 4.1.12. | Average Dose of Titration Phase | 24 |
| 4.1.13. | Average Dose of Maintenance Phase | 24 |
| 4.1.14. | Compliance with Study Drug | 24 |



| 4.1.15. | Handling of Incomplete or Missing Dates Associated with an Event | 25 |
|---|---|---|
| 4.1.16. | Handling of Alphanumeric Data | 26 |
| 4.2. | Visit Windows | 27 |
| 5. | STATISTICAL ANALYSIS METHODS | 28 |
| 5.1. | General Considerations | 28 |
| 5.2. | Populations for Analyses | 28 |
| 5.3. | Statistical Hypotheses | 29 |
| 5.4. | Multiplicity Adjustment | 29 |
| 5.5. | Strata and Covariates | 30 |
| 5.6. | Subject Disposition, Demographic and Baseline Characteristics | 30 |
| 5.7. | Medical and Psychiatric History | 30 |
| 5.8. | Exposure to Treatment | 31 |
| 5.9. | Primary Efficacy Analysis | 31 |
| 5.9.1. | Primary Estimand | 31 |
| 5.9.2. | Main Analytical Approach | 32 |
| 5.9.3. | Sensitivity Analyses | 32 |
| 5.9.3.1. | Treatment Effect at Final Dose Levels | 32 |
| 5.9.3.2. | Treatment Effect based on Actual Treatment Received | 32 |
| 5.9.3.3. | Remote Assessments Excluded (treated as missing) | 32 |
| 5.9.3.4. | Impact of Missing Values Handling | 33 |
| 5.9.4. | Subgroup Analyses | 34 |
| 5.10. | Key Secondary Efficacy Analyses | 35 |
| 5.10.1. | Secondary Estimand 1 | 35 |
| 5.10.1.1. | Main Analytical Approach | 35 |
| 5.10.1.2. | Sensitivity Analyses | 36 |
| 5.10.1.3. | Subgroup Analyses | 36 |
| 5.10.2. | Secondary Estimand 2 | |
| 5.10.2.1. | Main Analytical Approach | 36 |
| 5.10.2.2. | Sensitivity Analyses | 37 |
| 5.10.2.3. | Subgroup Analyses | 37 |
| 5.11. | Summary of Primary and Key Secondary Efficacy Analyses | 38 |



| 5.12. | Other Efficacy Analyses | 39 |
|---|---|---|
| 5.13. | Interim and Final Analysis | 41 |
| 5.14. | Safety Analyses | 41 |
| 5.14.1. | Adverse Events | 41 |
| 5.14.2. | Epworth Sleepiness Scale (ESS) | 42 |
| 5.14.3. | Questionnaire for Impulsive-Compulsive Disorders in Parkinson Disease Rating Scale (QUIP-RS) | 42 |
| 5.14.4. | Non-IMP Medications and Non-Drug Therapy/Procedures | 43 |
| 5.14.5. | Clinical Laboratory Assessments | 43 |
| 5.14.6. | Vital Signs | 44 |
| 5.14.6.1. | Blood Pressure and Heart Rate | 44 |
| 5.14.6.2. | Body Weight | 46 |
| 5.14.6.3. | Temperature | 46 |
| 5.14.7. | Electrocardiograms (ECGs) | 46 |
| 5.14.8. | Physical and Neurological Examinations | 46 |
| 5.14.9. | Columbia-Suicide Severity Rating Scale (C-SSRS) | 47 |
| 5.14.10. | Eye Examinations | 47 |
| 5.15. | Pharmacokinetics | 47 |
| 5.15.1. | Pharmacokinetic Data Analysis | 47 |
| 5.16. | Protocol Deviations | 47 |
| 6. | CHANGES IN THE PLANNED ANALYSES | 48 |
| 7. | REVISION HISTORY | 49 |
| 8. | REFERENCES | 50 |
| 9. | APPENDICES | 51 |
| 9.1. | Schedule of Assessments | 52 |
| 9.2. | EQ-5D-5L Dimensions | 57 |
| 9.3. | Columbia-Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation and Suicidal Behavior Scores | 58 |
| 9.4. | Programming Conventions | 60 |
| 9.5. | MNAR Cases Identified Prior to Database Lock | 62 |
| 9.6. | Core Codes for imputation of MAR and MNAR | 64 |
| 9.6.1. | Imputation of Missing at Random (MAR) Cases | 64 |



| 9.6.2. | Imputation of Missing Not at Random (MNAR) Cases | 64 |
|--------|------------------------------------------------------------|-----|
| 9.7. | Randomization Stratum Errors | 65 |
| 9.8. | CTCAE Based Laboratory Test Results Grading Specifications | 66 |
| 9.9. | EQ-5D-5L Index Cross-walk Mapping | 90 |
| 9.10. | Abbreviations | 152 |



# LIST OF TABLES

| Table 1: | Tavapadon and Placebo Dosing Schedule | 13 |
|----------|---------------------------------------|----|
| Table 2: | Trial Objectives and Endpoints | 14 |
| Table 3: | Visit Windows | 27 |
| Table 4: | Populations for Analysis | 28 |
| Table 5: | Schedule of Assessments | 52 |



# **LIST OF FIGURES**

Final Statistical Analysis Plan



#### 1. INTRODUCTION

This document describes the statistical methods and data presentations planned for the analysis of the efficacy and safety data from Protocol CVL-751-PD-001. Background information is provided for the study designs and objectives. Further details of study conduct, and data collection are provided in the study protocol and electronic case report forms (eCRFs).

# 1.1. Study Overview

This is a prospective, Phase 3, multicenter, multinational, randomized, double blind, placebo controlled, parallel group, 27 week trial of the efficacy, safety, tolerability, and pharmacokinetics (PK) of 2 fixed doses of tavapadon (5 mg QD and 15 mg QD) in male and female subjects aged 40 to 80 years who have a diagnosis of Parkinson's disease (PD), consistent with the UK Parkinson's Disease Society Brain Bank diagnostic criteria; a modified Hoehn and Yahr stage of 1, 1.5, or 2; a Movement Disorder Society − Unified Parkinson's Disease Rating Scale (MDS UPDRS) Part II score ≥2 and Part III score ≥10; and are not receiving antiparkinsonian medication other than monoamine oxidase B (MAO B) inhibitors.

A total of 522 subjects are planned to be randomized in a 1:1:1 ratio to receive tavapadon 5 mg QD, tavapadon 15 mg QD, or placebo QD. The dose of tavapadon will be titrated to a target dose using a fixed titration scheme. Randomization will be stratified by concurrent use of allowed Parkinson's disease (PD) medications (MAO-B inhibitors) during the Treatment Period. The planned duration of treatment is 27 weeks, including the Titration and Maintenance Phases. The trial will include a Screening Period (maximum of 4 weeks), a 27 week Treatment Period, and a 4 week Safety Follow-up Period. Details of schedule of assessments are provided in Section 9.1.

The trial design is depicted in Figure 1.





MAC-B = monoamine oxidase B, PD = Parkinson's disease, MDS-UPDRS = Movement Disorder Society – Unified Parkinson's Disease Rating Scale, QD = once daily

Note: The change from baseline to endpoint in the MDS-UPDRS Parts II and III combined score is the primary endpoint.

Note: The change from baseline to endpoint in the MUS-OPDIGS Patts if and in combined score is the primary endpoint.

Adverse events and concomitant medications will be recorded. Nonserious adverse events will be followed through Week 31. Serious adverse events will be followed to resolution.



## 1.2. Sample Size Considerations

A sample size of 174 subjects per group will provide 90% power to detect a change in the primary outcome measure (change from baseline to endpoint in the MDS-UPDRS Parts II and III combined score) of 4 points, with a standard deviation of 9, 2-sided alpha level = 0.025, and assuming a 27% dropout rate.

In the event of higher than anticipated early terminations due to COVID-19 or other reasons, Cerevel may extend enrollment in order to maintain the planned statistical power.

# 1.3. Measures to Minimize Bias: Randomization and Blinding

#### 1.3.1. Subject Assignment to Treatment

All subjects will be centrally randomized in a 1:1:1 ratio to 1 of 3 treatment arms (tavapadon 5 mg QD, tavapadon 15 mg QD, or placebo) at the Baseline Visit via an Interactive Voice Response System/Interactive Web Response System (IVRS/IWRS), according to a computer-generated randomization scheme. Randomization will be stratified by concurrent use of allowed antiparkinsonian medication (MAO-B inhibitor).

#### 1.3.2. Blinding

The tavapadon and placebo tablets will be identical in appearance and will be packaged in identically appearing blister cards. All subjects will take 3 tablets once daily of IMP throughout the Treatment Period, either all tavapadon tablets, all placebo tablets, or a combination of tavapadon and placebo tablets. Tablets will be packaged to allow dosage adjustments to be made without breaking the trial blind.

Treatment assignments will be blinded to the investigators and other trial site personnel, the subjects, and all sponsor personnel who are involved in the conduct of the trial (including trial monitoring, data management, and data analysis). Access to the treatment codes will be restricted to personnel who are responsible for generating and maintaining the randomization code, packaging the IMPs, operating the IVRS/IWRS, analyzing the PK blood samples, or reporting serious adverse events (SAEs) or adverse events of special interest (AESI) to regulatory agencies.

Documentation of breaking the blind should be recorded in the subject's medical record and eCRFs, with the reason for breaking the blind, the date and time the blind was broken, and the names of the personnel involved. Once the blind is broken for a subject, treatment with the IMP may not be reinitiated for that subject.

#### 1.4. Treatment Period

The dose of tavapadon will be titrated to either 5 mg QD or 15 mg QD and then maintained for the duration of the 27-week Treatment Period. The titration schedule, as shown in Table 1, will be used for all subjects who are randomized to receive tavapadon. Subjects will take 3 tablets of investigational medicinal product (IMP), either all tavapadon tablets, all placebo tablets, or a combination of tavapadon and placebo tablets, throughout the trial to maintain the trial blind.



will be allowed. Titration of tavapadon No deviations in the titration schedule up through should be guided by absence of tolerability issues that are reported as AEs and that are of sufficient severity resulting in significant dysfunction or distress to the subject. Any questions regarding tolerability issues and titration should be directed to the medical monitor before adjustments are initiated. Subjects who cannot achieve or tolerate the dose at (5 mg QD) (10 mg QD) must be discontinued from the trial. Starting on Day 74, subjects who achieve but do not tolerate the dose at may go back to dose or will be permitted a one-time the dose at Subjects may remain at the dose if needed for symptomatic control. Subjects must receive rechallenge back to the dose for at least 7 days before a rechallenge to the who are unable to tolerate the dose upon rechallenge will be discontinued from the trial. Table 1: **Tavapadon and Placebo Dosing Schedule** 



## 2. OBJECTIVES AND ENDPOINTS

**Table 2:** Trial Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| To assess the efficacy of 2 fixed doses of tavapadon in subjects with early PD | <ul> <li>Primary Efficacy Endpoint</li> <li>Change from baseline to endpoint in the MDS-UPDRS Parts II and III combined score</li> <li>Key Secondary Efficacy Endpoints</li> <li>Change from baseline to endpoint in the MDS-UPDRS Part II score</li> <li>Percentage of responders at endpoint, defined as a score of "much improved" or "very much improved" on the PGIC</li> <li>Secondary Efficacy Endpoints (All Time Points)</li> <li>Change from baseline in the MDS-UPDRS Parts II and III combined score</li> <li>Change from baseline in the MDS-UPDRS Parts I, II, and III combined score</li> <li>Change from baseline in the MDS-UPDRS Part I, Part II, and Part III individual scores</li> <li>Change from baseline in the CGI-S score</li> <li>CGI-I score</li> <li>PGIC score</li> <li>Other Endpoints</li> <li>Change from baseline in PDQ-39 score</li> <li>Change from baseline in Schwab and England ADL score</li> <li>Change from baseline in the EQ-5D-5L index and VAS scores</li> </ul> |
| Secondary | |
| To assess the safety and tolerability of 2 fixed doses of tavapadon in subjects with early PD | <ul> <li>ESS</li> <li>QUIP-RS</li> <li>C-SSRS</li> <li>Nature, frequency, and temporality of TEAEs, including abuse-related AEs and AEs related to MHIs</li> <li>Clinical laboratory evaluations</li> <li>Vital signs</li> <li>Physical and neurological examinations</li> <li>ECGs</li> </ul> |
| Pharmacokinetic | |
| To evaluate the PK of tavapadon in this population | <ul> <li>Plasma concentrations of tavapadon and its major<br/>metabolite (if required) at baseline (Day 1) and<br/>Weeks 5, 11, 14, 22, and 27</li> </ul> |

Abbreviations: ADL = activities of daily living, AE = adverse event, CGI-I = Clinical Global Impression – Improvement, CGI-S = Clinical Global Impression – Severity of Illness, C-SSRS = Columbia-Suicide Severity Rating Scale, ECG = electrocardiogram, EQ-5D-5L = EuroQol 5 Dimension 5 Level, ESS = Epworth Sleepiness Scale, MDS-UPDRS = Movement Disorder Society-Unified Parkinson's Disease Rating Scale, MHIs = medication handling irregularities, PD = Parkinson's disease, PDQ-39 = 39-Item Parkinson's Disease Rating Scale, PGIC = Patient Global Impression of Change, PK = pharmacokinetic, QUIP-RS = Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale, TEAE = treatment-emergent adverse event, VAS = visual analog scale.



## 3. KEY ASSESSMENTS AND DERIVATIONS

## 3.1. Efficacy Assessments

# 3.1.1. Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS)

The MDS-UPDRS (Goetz et al, 2008) is a multidimensional scale that assesses the motor and nonmotor impacts of PD across 4 parts. The scale is completed using a combination of physician and patient assessments and a collection of information from the patient or caregiver. Each evaluation item is rated on a scale from 0 to 4 on which 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. This trial incorporates Part I, II, and III assessments for the specific trial population.

#### 3.1.1.1. Part I Score

Part I of the MDS-UPDRS focuses on the non-motor aspects of experiences of daily living. The MDS-UPDRS Part I score value for a given visit is obtained as the sum of all 13 evaluation items in the MDS-UPDRS Part I subscale, including the 6 items which are rated by the Physician. Valid values for the sum are integers from 0-52, with 0 being the least severe and 52 being the most severe.

#### **3.1.1.2. Part II Score**

Part II of the MDS-UPDRS focuses on the motor aspects of experiences of daily living. The MDS-UPDRS Part II score value for a given visit is obtained as the sum of all 13 evaluation items in the MDS-UPDRS Part II subscale. Valid values for the sum are integers from 0-52, with 0 being the least severe and 52 being the most severe.

#### 3.1.1.3. Part III Score

Part III of the MDS-UPDRS is the motor evaluation comprises 18 items that are assessed by the investigator (resulting in 33 scores by location and lateralization). Valid values for the sum are integers from 0-132, with 0 being the least severe and 132 being the most severe.

## 3.1.1.4. Handling of Missing Items from MDS-UPDRS

If individual items are missing from a given part of the MDS-UPDRS, the corresponding total score may be generated by prorating the response if the number of missing items is not excessive. For Part I and Part II assessments, only a single missing item score is allowable. For Part III, up to 7 missing item scores are allowable. To prorate the value, the following formula is utilized

$$P = \left(\frac{\sum_{i=1}^{n} j_{i}}{n}\right) U$$

Where n is the number of non-missing items,  $j_1$ - $j_n$  represents the n non-missing values reported by the subject for the given subscale, and U is the number of total items in the subscale. If more than the allowable items are missing, the total score will be treated as missing.

#### 3.1.1.5. Part II + III Combined Score

The MDS-UPDRS Part II + III Combined Score is defined as the sum of the total scores for Part II and Part III within a given assessment (i.e., to have a Part II + III Total score, the subject must have a non-missing Part II total score and a non-missing Part III total score on the same date). The Part II + III Combined Score will be derived after any imputation of missing values within each individual total score.

## 3.1.1.6. Part I, Part II, and Part III Combined Score

The MDS-UPDRS Part I, Part II, and Part III Combined Score is defined as the sum of the total scores for Parts I, II, and III within a given assessment (i.e., to have a Part I, Part II, and Part III Combined score, the subject must have a non-missing Part I total score, a non-missing Part II total score, and a non-missing Part III total score on the same date). The Part I, Part II, and Part III Combined Score will be derived after any imputation of missing values within each individual total score.

#### 3.1.2. Patient Global Impression of Change (PGIC)

The PGIC is the patient-reported outcome in a 7 point scale to rate how much the patient's illness has improved or worsened relative to the baseline state at the beginning of the intervention. The qualitative assessment of meaningful change is determined by the patient in response to the question, "Compared to your condition at the beginning of treatment, how much has your condition changed?" Scores are: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; and 7=very much worse.

## 3.1.3. Clinical Global Impression – Severity of Illness (CGI-S)

The CGI-S scale is a 7 point scale that requires the clinician to rate the severity of the patient's illness at the time of the assessment relative to the clinician's experience with patients who have the same diagnosis. Raters select one response based on the following question: "Considering your total clinical experience with this particular population, how ill is the patient at this time?" Scores are: 1=normal, not at all ill; 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=among the most extremely ill patients.

#### 3.1.4. Clinical Global Impression – Improvement (CGI-I)

The CGI-I is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to the baseline state at the beginning of the intervention. Raters select one response based on the following question, "Compared to your patient's condition at the beginning of treatment, how much has your patient changed?" Scores are: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; and 7=very much worse.

#### 3.1.5. 39-Item Parkinson's Disease Questionnaire (PDQ-39) Score

The 39-item Parkinson's Disease Questionnaire (PDQ-39) measures 39 items, which assess 8 domains of health: mobility (10 items), activities of daily living (6 items), emotional well being (6 items), stigma (4 items), social support (3 items), cognitions (4 items), communication (3 items), and bodily discomfort (3 items) (Peto et al, 1998). Each item is scored on the following scale: 0=never, 1=occasionally, 2=sometimes, 3=often, and 4=always. Items in each subscale and the total scale can be summarized into an index and transformed linearly to a scale from 0 (perfect health as assessed by the measure) to 100 (worst health as assessed by the measure).

A dimension score is calculated using the following formula:

$$d = \frac{1}{n*4} \sum_{j=1}^{n} t_{j}$$

where n is the number of items in the dimension, and  $t_j$  is the  $j^{th}$  item in the dimension. This transforms the scale linearly from 0 (perfect health as assessed by the measure) to 100 (worst health as assessed by the measure). If items are missing within a domain, the n in the above formula will be changed to the number of items in the dimension that the subject answered if at least half of the questions in the domain were answered. Otherwise, a domain and summary index will not be calculated.

A summary index called PDQ-39 SI, is calculated as the average of the 8-dimension scores.

#### 3.1.6. EuroQol 5 Dimension 5 Level

The EuroQol 5 Dimension 5 Level (EQ 5D 5L) is a patient-reported outcome that measures health in 5 dimensions. It is a widely used survey instrument for measuring economic preferences for health states, is applicable to a wide variety of health conditions and treatments, and provides a simple descriptive profile and a single index value for health status (Herdman et al, 2011). The EQ 5D 5L consists of a descriptive system and a visual analog scale (VAS).

The descriptive system comprises 5 dimensions: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The patient is asked to indicate his or her health state by ticking the box next to the most appropriate statement in each of the 5 dimensions (Section 9.2). This decision results if a 1 digit number that expresses the level that was selected for that dimension. The digits for the 5 dimensions are combined into a 5 digit number that describes the patient's health state. For example, 11122 would represent the health state for someone who has no problems with mobility, self-care, or usual activities, but who has slight pain or discomfort and slight anxiety or depression. For each subject and visit, the 5-digit health state will be converted into a single summary index, the EQ-5D Index, using the EQ-5D-5L Index calculator with US value set (van Hout, Janssen et al. 2012; Section 9.9).

Final Statistical Analysis Plan



The EQ VAS records the patient's self-rated health on a 20-cm vertical visual analogue scale (VAS). The VAS is numbered from 0 to 100 with 0 meaning 'the worst health you can imagine' and 100 meaning 'the best health you can imagine'. This information can be used as a quantitative measure of health outcome that reflects the patient's own judgement. The EQ-5D-5L asks respondents to simply 'mark an X on the scale to indicate how your health is TODAY' and then to 'write the number you marked on the scale in the box below'.

#### 3.1.7. Schwab and England Activities of Daily Living (ADL) Scale

The Schwab and England ADL scale is a method of assessing a person's ability to perform daily activities in terms of speed and independence through a percentage figure. The clinician determines the rating according to the following criteria, with 100% indicating total independence and 0% indicating a state of complete dependence:

- 100% Completely independent. Able to do all chores without slowness, difficulty, or impairment. Essentially normal. Unaware of any difficulty.
- 90% Completely independent. Able to do all chores with some degree of slowness, difficulty, and impairment. May take twice as long. Beginning to be aware of difficulty
- 80% Completely independent in most chores. Takes twice as long. Conscious of difficulty and slowness.
- 70% Not completely independent. More difficulty with some chores. Three to four times as long in some. May spend a large part of the day with chores.
- 60% Some dependency. Can do most chores, but exceedingly slowly and with much effort. Errors; some impossible.
- 50% More dependent. Help with half, slower, etc. Difficulty with everything.
- 40% Very dependent. Can assist with all chores, but few alone
- With effort, now and then does a few chores alone or begins alone. Much help needed
- 20% Nothing alone. Can be a slight help with some chores. Severe invalid
- 10% Totally dependent, helpless. Complete invalid.
- 0% Vegetative functions such as swallowing, bladder and bowel functions are not functioning. Bedridden.

# 3.2. Safety Assessments

# 3.2.1. Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease Rating Scale (QUIP-RS) Scores

The QUIP RS has 4 primary questions that pertain to commonly reported thoughts, urges/desires, and behaviors associated with impulse control disorders (ICDs), each of which is applied to 4 ICDs (compulsive gambling, buying, eating, sexual behavior) and 3 related disorders (medication use, punding, and hobbyism).



Each question is scored using a 5 point Likert scale (score, 0=never [not at all], 1=rarely [infrequently or 1 day/week], 2=sometimes, 3=often, 4=very often). Scores for each ICD and related disorder range from 0 to 16, with a higher score indicating greater severity (frequency) of symptoms.

The total QUIP-RS score for all ICDs and related disorders combined ranges from 0 to 112. In case of missing item scores, the missing value will be replaced by the average of non-missing scores at the same visit from the same subject. In case all item scores in any subcategory are missing, the total score will be set as missing.

## 3.2.2. Epworth Sleepiness Scale (ESS) Total Score

The ESS scale is used to determine the level of daytime sleepiness. There are 8 situations listed for which patients rate their likelihood of dozing or sleeping (0=no chance of dozing, 1=slight chance of dosing, 2=moderate chance of dosing, or 3=high chance of dozing). The total score is the sum of 8 item scores and can range between 0 and 24. The higher total score indicates the higher level of daytime sleepiness. A score of 10 or more is considered sleepy, and a score of 18 or more is very sleepy.

In case of missing item scores from the ESS, the missing value will be replaced by the average of non-missing scores at the same visit from the same subject. In case all item scores are missing, the total score will be set as missing.

## 3.2.3. Adverse Event (AE)

An AE is defined as any untoward medical occurrence in a patient or clinical trial subject, temporally associated with the use of trial intervention, whether considered related to the trial intervention. NOTE: Signs and symptoms and/or abnormal laboratory test result indicating a common underlying pathology/diagnosis should be reported as a single AE.

All adverse events will be recorded on the ADVERSE EVENTS eCRF. Adverse events with missing severity will have the severity imputed as 'Severe' for the AE tabulations. Adverse events with missing relationship to IMP will have the relationship imputed as 'Related' for the AE tabulations if the AE started on or after the first dose of IMP. However, in the data listings these missing severity and/or relationship will be presented as missing.

#### 3.2.3.1. Adverse Event of Special Interest (AESI)

For this study, any AEs related to abuse potential, AEs involving MHIs, abnormal liver function tests with a value  $>3 \times ULN$  for ALT or AST and  $>2 \times ULN$  for total bilirubin within the same visit, a value of  $>3 \times ULN$  for ALT or AST and clinical jaundice, an AE leading to the discontinuation of IMP or from the study will be considered AESIs. These events will be noted by the investigator in the ADVERSE EVENTS eCRF.

#### **3.2.3.2.** Treatment-emergent Adverse Event (TEAE)

Any event reported on the eCRF that occurs on or after the initiation of IMP until the end of AE reporting period per protocol is considered treatment emergent.



Additionally, it is assumed that an Adverse Event which was reported to have started on Day 1 without an associated onset time is assumed to be treatment emergent.

### 3.2.4. Clinical Safety Laboratory Assessments

The clinical laboratory tests as listed in the protocol will be performed in accordance with the laboratory manual and the Schedule of Assessments. All results, including repeats, will be included in the laboratory reports. The investigator must review the laboratory report, document this review, and record any clinically relevant changes occurring during the trial in the AE section of the eCRF.

#### 3.2.4.1. Treatment-emergent Laboratory Abnormality and Toxicity

A treatment-emergent laboratory abnormality is defined as value outside the normal range which occurs on or after the start of IMP and up to the last contact following discontinuation of IMP.

A treatment-emergent laboratory toxicity is defined as an increase of at least one abnormality severity grade (specifications in Section 9.8) from the baseline assessment at any post baseline visit which occurs after the first administration of IMP and through last test results of the study. If a laboratory assessment obtained on Day 1 with unknown collection times will be assumed to be an assessment prior to the initiation of IMP. If the relevant baseline assessments are missing for a given subject, any post-baseline severity grade at 1 or more is considered a treatment-emergent laboratory toxicity.

## 3.2.5. Columbia-Suicide Severity Rating Scale (C-SSRS)

Suicidality will be monitored during the trial using the C-SSRS. It was designed to quantify the severity of suicidal ideation and behavior.

This trial will use the "Baseline/Screening" and "Since Last Visit" versions of the scale. The "Baseline/Screening" version, which assesses the lifetime experience of the subject with suicide events and suicidal ideation and the occurrence of suicide events or ideation within a specified time period prior to entry into the trial, will be completed for all subjects at screening to determine eligibility and confirmed at baseline. Any subject with active suicidal ideation or suicidal behaviors within the last 6 months, suicidal behaviors within the last 2 years, or who in the clinical judgment of the investigator presents a serious risk of suicide should be excluded from the trial.

The "Since Last Visit" C-SSRS form will be completed at all visits after screening and baseline. The investigator will review the results of the "Since Last Visit" C-SSRS during the trial to determine whether it is safe for the subject to continue in the trial. If a subject demonstrates potential suicidal ideation associated with actual intent or method or plan as indicated by "YES" answers on item 4 or 5 of the C-SSRS, the investigator will evaluate whether a risk assessment by a qualified mental health professional (or the investigator alone if the investigator is a qualified mental health professional) is needed and whether the subject should continue in or be discontinued from the trial.

Details of C-SSR categories as well as definition of treatment emerging events are provided in Section 9.3.



## 3.2.6. Vital Signs

Vital signs include systolic and diastolic blood pressures, heart rate, and body temperature. Duplicate measurements of blood pressure and heart rate will be obtained supine (after 5 minutes of rest) and 1 measurement of blood pressure and heart rate will be obtained on standing (2 minutes after rising from supine to standing). The duplicate values will be individually recorded, and the values will be averaged by the sponsor for the time point assessment. Body temperature will be obtained once, at the time of the first blood pressure measurement.

## 3.2.7. Electrocardiograms

Single or triplicate 12 lead ECGs will be obtained during the trial. All ECG recordings be obtained after the subject has been supine and at rest for at least 5 minutes. A triplicate set of ECGs is 3 consecutive ECGs collected 1 to 2 minutes apart over a 5 minute period.

A single ECG will be obtained at the Screening Visit. For US sites, three sets of triplicate ECGs will be obtained during the 45 minutes before administration of the first dose of IMP on Day 1 (at -45, -30, and -15 minutes), and a single set of triplicate ECGs will be obtained ~1 hour after administration of the first dose of IMP on Day 1, just prior to the time of collection of the PK blood sample. One set of triplicate ECGs will be obtained at the Weeks 5, 11, 14, 22, and 27 clinic visits, just prior to the time of collection of the PK blood sample. The triplicate ECG information from US sites will be used in a C-QT analysis with results reported separately. For non-US sites, one set of triplicate ECGs will be obtained before administration of the first dose of IMP on Day 1, and a single ECG will be obtained ~1 hour after administration of the first dose of IMP on Day 1, just prior to the time of collection of the PK blood sample. Single ECGs will be obtained at the Weeks 5, 11, 14, 22, and 27 clinic visits, just prior to the time of collection of the PK blood sample. A central ECG service will be used for reading all ECGs to standardize interpretations for the safety analysis.

# 3.2.8. Prior Medications, Concomitant Medications and Medications Taken Post Last Dose of IMP

Prior medications are those medications taken prior and ended prior to the initiation of IMP. These medications will be captured in the CONCOMITANT MEDICATIONS eCRF.

Concomitant medications are those medications taken on or after the initiation of IMP. These medications include those medications started before the initiation of IMP and continuing post Day 1. Medications that start after the last dose of IMP until the end of protocol-specified reporting period will be classified as taken post last dose and will not be considered concomitant. These medications will be recorded in the eCRF. The investigator will record all medications and therapies (including vaccines, over-the-counter or prescription medicines, vitamins, and/or herbal supplements) that are used by the subject from 30 days before the informed consent form (ICF) is signed through the end of the Safety Follow-up Period (Week 31 or early termination). The investigator will also record all medications and therapies taken or received by a subject for treatment of an AE or that cause an AE through Week 31 or early termination.



#### 3.2.9. Physical and Neurological Examinations

A complete physical and neurological examinations will be conducted at screening and at the end of treatment visit (Visit 11 or early termination visit). Any condition present post-baseline physical or neurological examination that was not present at the baseline examination should be documented as an AE and followed to a satisfactory conclusion.



## 3.3. Pharmacokinetics

Blood samples for measurement of plasma concentrations of tavapadon and CVL-0000053, its major metabolite, will be collected ~1 hour after administration of the first dose of IMP on Day 1 and at the clinic visits at the end of Weeks 5, 11, 14, 22, and 27.

Drug concentration information will not be reported to investigative sites, clinical database or any blinded study personnel until the trial has been completed and unblinded.



#### 4. DATA CONVENTIONS AND VISIT WINDOWS

#### 4.1. Data Conventions

## 4.1.1. Age

Age is the age at the time of informed consent and is as captured on the eCRF (note: date of birth is not captured on the eCRF).

#### 4.1.2. Day 1

Day 1 is the day IMP is first initiated.

## 4.1.3. Endpoint

Endpoint as defined as the primary time point for the efficacy assessments is Week 26.

#### 4.1.4. Study Day of an Event

Study day of an event is defined relative to Day 1 as:

Study Day = event date – date of Day 1 (+ 1, if event date  $\geq$  date of Day 1).

This calculation will result in negative study days for an event occurring prior to the start of IMP and positive study days for an event on or after the start of IMP. There will be no Day 0 value to match the schedule of events.

#### 4.1.5. Days on Study

Days on Study is the number of days from Day 1 to the date of study completion or early termination as recorded on the END OF STUDY eCRF.

#### **4.1.6. Days on IMP**

Days on IMP is the number of days from Day 1 to the date of last dose of IMP as recorded on the EXPOSURE eCRF.

#### 4.1.7. Baseline Value

For purposes of analysis, the baseline value of a given assessment is defined as the last value obtained prior to initiation of IMP. Should the Day 1 visit value be obtained after the first dose of IMP or if this value is not available at Day 1, the most recent value obtained prior to the first dose of IMP will be used for the baseline value.

For US subjects with triplicate ECGs taken at 3 pre-dose timepoints, the baseline value will be defined as the average of the available pre-dose ECG values (i.e. triplicate ECGs at -45 minutes pre-dose, -30 minutes pre-dose, and -15 minutes pre-dose). For non-US subjects, the baseline value will be defined as the average of the available pre-dose ECG values. Scheduled records will be selected over unscheduled records if a tie breaker is needed.

For blood pressure and heart rate measurements, baseline is defined as the average of the duplicates at the last visit prior to the IMP administration. If no duplicate is available, the last non-missing value prior to the initiation of IMP will be used.

#### 4.1.8. Change from Baseline

Change from baseline for a given variable is defined as the value on a given Study Day (Time Point) minus the Baseline Value.

### 4.1.9. Orthostatic Change

Orthostatic change is calculated as the difference in the standing value from the supine value (i.e., supine value – standing value). If an average value is available at a given visit and date, it will be used for the calculation of orthostatic change. If an average value is not available, the individual record obtained on a given visit and date will be used.

#### 4.1.10. Duration of Titration Phase

The duration of the titration phase will be calculated as the days in schedule.

#### 4.1.11. **Duration of Maintenance Phase**

The duration of the maintenance phase will be calculated as the days in schedule.

#### **4.1.12.** Average Dose of Titration Phase

The average dose of the titration phase will be calculated as the sum of the milligrams of study drug taken in of the dosing schedule divided by the duration of days in the titration phase.

#### 4.1.13. Average Dose of Maintenance Phase

The average dose of the maintenance phase will be calculated as the sum of the milligrams of study drug taken in of the dosing schedule divided by the duration of days in the maintenance phase.

#### 4.1.14. Compliance with Study Drug

Accountability and compliance will be assessed through self-reporting by the subject and by tablet count at each clinic visit. For analysis purposes, evaluation of compliance will be based on the site assessment of compliance as recorded on the DRUG ACCOUNTABILITY eCRF. Compliance will be calculated as a percentage based on the total number of tablets taken relative to the total expected number of tablets based on days on study. If a kit was lost and return information was available, the return information will be used for the compliance calculation. If a kit was lost and no return information was available, it is assumed that the tablets were not taken for the compliance calculation. If return information is not available and the kit was not lost, it is assumed that the tablets were taken for the compliance calculation.

If a kit was redispensed and the number of tablets redispensed is not available, it is assumed that the number of tablets that were partially returned were redispensed for the compliance calculation.

#### 4.1.15. Handling of Incomplete or Missing Dates Associated with an Event

An incomplete date occurs when the exact date an event (e.g. an adverse event) occurred or ended cannot be obtained from a subject. The database contains data fields for month, day, and year. A date is incomplete if at least one of these three fields is not known.

For many of the planned analyses, a complete date is necessary to determine if the event should be included in the analysis (e.g. if the event is treatment-emergent) or to establish the duration of an event. In such cases, incomplete dates will be imputed as described below.

For the purposes of handling partially reported start and stop dates for an event the following algorithm will be applied:

- Missing start day, but month and year present:
   If the event occurs same month and year as the occurrence of IMP, then the start day of the event will be assigned to the day of first dose of IMP (i.e., Day 1).

   Otherwise the start day will be set to the first day of the month.
- Missing start day and month, but year present:
   If event occurs in the same year as IMP, then the start date of the event will be assigned to Day 1.
  - Otherwise the start day and month will be set to 01 January.
- In the unlikely event of a completely missing start date (year not present), the start date will be imputed as Day 1.
- Missing end day, but month and year present: The day will be set to the last day of the month.
- Missing end day and month, but year present:

  The end day and month will be set to the date of study completion. However, if study completion year is greater than the year of the event, then the day and month will be set to 31 December.
- Missing all components of an end date and the event is not marked as ongoing: The event will be considered as 'ongoing' and will be considered treatment-emergent if the start date is on or after Day 1.

If any imputed start date causes the start date to occur after the end date, the end date will be used for the imputation of the start date. If any imputed end date causes the end date to occur prior to the start date of the event, the start date of the event will be used for the imputation of the end date. If the imputed date is later than the date of study withdrawal, then the date of study withdrawal will be used to impute the date in question. In subject data listings, start and stop date of events will be displayed as reported on the eCRF without imputed dates.



For the purposes of handling partially reported diagnosis date of Parkinson's disease, the following algorithm will be applied to randomized subjects:

• Missing day, but month and year present:

If the diagnosis date occurs same month and year as the occurrence of the subject's screening date, then the day of the diagnosis date will be assigned to the day of the subject's screening date.

Otherwise the diagnosis day will be set to the first day of the month.

• Missing day and month, but year present:

If the diagnosis date occurs in the same year as the occurrence of the subject's screening date, then the diagnosis date will be assigned to the subject's screening date.

Otherwise the diagnosis day and month will be set to 01 January.

• In the event of missing year or a completely missing diagnosis date, the diagnosis date will be assigned to the subject's screening date.

In subject data listings, diagnosis dates will be displayed as reported on the eCRF without imputed dates. For screen failures, no imputation will be made to the date of diagnosis of Parkinson's disease.

## 4.1.16. Handling of Alphanumeric Data

Should there be instances where a clinical laboratory parameter is reported with imbedded non-numeric characters, as for example, "<0.1" or ">10", the data will be imputed as described below for quantitative summaries. The actual alphanumeric values as reported in the database will be presented in data listings.

- The values < LLN will be replaced with  $\frac{1}{2}$  the value of the lower limit. For example, "< 0.1" will be replaced with 0.05 if the LLN is 0.1.
- The values > ULN will be replaced by values of increased precision by one level. For example, ">0.1" will be imputed to "0.11" if the ULN is 0.1, and ">10" will be imputed to "10.1" if the ULN is 10.

Additionally, in the event of the upper limit of normal (ULN)/lower limit of normal (LLN) reported as alphanumeric (e.g., '<5', '>5', '>5', '>5'), the determination of the laboratory abnormality severity grade will be based on the convention on the ULN and LLN below:

• If the ULN is in the form of ≤5, only the numeric part will be used for determining the abnormality severity grade of the test results (i.e., the ULN is set to 5). If the ULN is in the form of <5, the numeric value of the ULN will be decreased by two levels of precision in the direction of the symbol (i.e., the ULN is set to 4.99).



• If the LLN is in the form of ≥5, only the numeric part will be used for determining the abnormality severity grade of the test results (i.e., the LLN is set to 5). If the LLN is in the form of >5, the numeric value of LLN will be increased by two levels of precision in the direction of the symbol (i.e., the LLN is set to 5.01).

#### 4.2. Visit Windows

Data collected longitudinally across visits will be summarized and analyzed by visit.

Laboratory data will be presented according to the nominal visit as collected from the eCRF or laboratory data unless the visit is an early termination or unscheduled visit. Early termination and unscheduled visits will be assigned visit windows based on the study day completed according to Table 3. Baseline will be determined per the baseline definition in Section 4.1.7. Other assessment data, including efficacy assessments data, will be mapped to the appropriate time point based on the window as defined in Table 3 from Baseline to Week 22 to appropriately captured time of assessment in cases of visit schedule variations. Due to the short interval between Visit 10 (Week 26) and Visit 11 (Week 27), data obtained at the nominal visit at this two time points will be used with the exception of early termination/unscheduled visits.

**Table 3: Visit Windows** 

| Analysis Visit | Analysis Visit Target Day | Analysis Visit Window |
|----------------|---------------------------|-----------------------|
| Baseline | 1 | ≤ 1 |
| Day 1* | 1 | 1 |
| Week 2 | 14 | 2 - 24 |
| Week 5 | 35 | 25 - 45 |
| Week 8 | 56 | 46 – 66 |
| Week 11 | 77 | 67 – 86 |
| Week 14 | 98 | 87 – 111 |
| Week 18 | 126 | 112 – 140 |
| Week 22 | 154 | 141 – 168 |
| Week 26 | 182 | 169 – 185 |
| Week 27 | 189 | 186 and higher |

<sup>\*</sup>Day 1 assessments are pre-IMP except ECG with a 60 minute post-dose assessment

If assessments are collected multiple times within a given visit window the result closest to the analysis visit target day will be used for summary presentations. If two measurements have the same distance to the target day, the later value will be used. If a subject has multiple non-missing values on the same date, the average record will be used (if applicable). If there are multiple average records on the same date, the average based on the scheduled measurements will be used. If no averages exist, the last record as determined by the time collected will be used.



#### 5. STATISTICAL ANALYSIS METHODS

#### **5.1.** General Considerations

Descriptive statistical methods will be used to summarize the data from this trial, with statistical testing performed for the efficacy endpoints. Unless stated otherwise, the term "descriptive statistics" refers to number of subjects (N), number of observations (n), arithmetic mean, median, standard deviation (SD), geometric mean and coefficient of variation (CV%) (for concentration data only), first quartile (Q1), third quartile (Q3), minimum, and maximum for continuous data, and frequencies and percentages for categorical data. Certain figure presentations will include the standard error of the mean (SE). The term "treatment group" refers to treatment assignment: placebo, tavapadon 5 mg, and tavapadon 15 mg. All data collected from subjects who sign the informed consent form, including screen failures, will be included in data listings. Unless otherwise noted, the data listings will be sorted first by treatment group and subject number and then by date within each subject number.

The number and proportion of missing visits and key assessments due to COVID-19 control measures and the frequency of remote assessments performed due to COVID-19 restrictions will be tabulated by treatment, visit, and assessment as well as the overall number and proportion of subjects with any such missing visits, assessments, or remote visits in each treatment group.

The statistical analyses will be conducted with the SAS® software package version 9.4 or higher.

# **5.2.** Populations for Analyses

The analysis populations are defined Table 4.

**Table 4: Populations for Analysis** 

| Population | Description | Analysis |
|---|---|---|
| ITT | All randomized subjects | Demographic and Baseline<br>Characteristics |
| FAS | All randomized subjects who receive at least 1 dose of IMP. This will be the safety analysis set. | Safety analysis |
| mITT | All randomized subjects who receive at least 1 dose of IMP and have a baseline and at least one postbaseline MDS-UPDRS assessment. | Primary analysis set for efficacy |
| Endpoint completers | All subjects in the mITT population who have an MDS-UPDRS assessment at baseline and endpoint | Sensitivity analysis set for efficacy |
| PK | All randomized subjects who receive at least 1 dose of tavapadon and have at least one measurable scheduled tavapadon (CVL751) concentration | PK analysis set |

Abbreviations: FAS = full analysis set, IMP = investigational medicinal product, ITT = intent-to-treat, mITT = modified intent-to-treat, PK = pharmacokinetic, MDS-UPDRS = Movement Disorder Society – Unified Parkinson's Disease Rating Scale.



# **5.3.** Statistical Hypotheses

The primary and key secondary hypotheses are summarized below. All will be tested based on 2-sided  $\alpha$ .

| Primary Endpoint | Tavapadon 15 mg QD vs Placebo | Tavapadon 5 mg QD vs Placebo |
|---|---|---|
| Change from baseline to endpoint in MDS-UPDRS Part II and III combined score | $H_1$ : $\mu_{active} = \mu_{placebo}$ vs $\mu_{active} \neq \mu_{placebo}$ | $H_2$ : $\mu_{active} = \mu_{placebo}$ vs $\mu_{active} \neq \mu_{placebo}$ |
| <b>Key Secondary Endpoints</b> | | |
| Change from baseline to endpoint | $H_3$ : $\mu_{\text{active}} = \mu_{\text{placebo}}$ | $H_5$ : $\mu_{\text{active}} = \mu_{\text{placebo}}$ |
| in the MDS-UPDRS Part II score | vs $\mu_{active} \neq \mu_{placebo}$ | vs $\mu_{active} \neq \mu_{placebo}$ |
| Proportion of responders on the | $H_4$ : $\pi_{\text{active}} = \pi_{\text{placebo}}$ | $H_6$ : $\pi_{\text{active}} = \pi_{\text{placebo}}$ |
| PGIC at endpoint | vs $\pi_{active} \neq \pi_{placebo}$ | vs $\pi_{ m active} eq \pi_{ m placebo}$ |

# 5.4. Multiplicity Adjustment

A graphical approach depicted below is utilized to illustrate the hierarchal multiple testing strategy planned for the hypotheses described above to control the overall Type I error rate. The primary endpoint of the tavapadon 15 mg QD will be compared with that of placebo ( $H_1$ ) with full  $\alpha$  of 0.05 and, if successful, the available  $\alpha$  will be passed along fully (r=1) to the comparison of the primary endpoint of tavapadon 5 mg QD with placebo ( $H_2$ ). If  $H_2$  is successful, the full  $\alpha$  will be available to the secondary hypothesis  $H_3$ . The sequence will continue until  $H_6$  or until the sequence breaks with no  $\alpha$  remaining available.



#### 5.5. Strata and Covariates

The randomization is stratified by concurrent use of MAO-B inhibitor. This factor is planned to be included as a covariate in the efficacy analyses. However, due to isolated administrative errors at a few sites during randomization through IRT system, 15 subjects were randomized to the incorrect strata (3 non-MAO-B inhibitor users were randomized to the MAO-B inhibitor use stratum and 12 MAO-B inhibitor users were randomized to the non-user stratum; details in Section 9.7). The actual MAO-B inhibitor use status, as recorded in eCRF, will be used as a covariate instead of the randomization strata in these cases.

The baseline value of each efficacy variable (if applicable) will also be included as a covariate in the efficacy analyses.

# 5.6. Subject Disposition, Demographic and Baseline Characteristics

Subject disposition will be based on the ITT population with tabulation of the number of subjects who complete the study and the number of discontinued and from the study and the reasons by treatment group. Additionally, the number of days on study will be summarized.

Tabulation of subject randomization by country and site will be presented for the ITT population and for completed subjects. A listing of randomization number, subject, treatment randomized, country, and site will be provided. Further tabulation by region (United States, Non-US) and country will also be presented. Subject disposition data will also be tabulated for all subjects screened to include the number of subjects screened, the number of screen failures, and the reason for screen failure.

Kaplan-Meier plots will be used to assess time to discontinuation of study treatment, time to discontinuation of treatment due to adverse events, and time to discontinuation of treatment due to subject withdrawal. The complete subjects or subjects discontinued treatment for reasons other than adverse events and withdrawal of consent will be censored at the time of end of treatment for the respective KM analyses. If a subject died without treatment discontinuation date information, date of death will be used as the time of discontinuation.

Number of subjects in each analysis population set will be summarized.

Demographic data and baseline characteristics including age, age categorical distribution, sex, childbearing potential, race, ethnicity, height at screening, weight at screening and at baseline, BMI at screening and at baseline, MAO-B inhibitor use at baseline, history of Parkinson's disease (including years from initial diagnosis), Montreal Cognitive Assessment (MoCA) total score, Modified Hoehn & Yahr assessment at screening, MDS-UPDRS (all parts, Part I + Part II + Part III combined, and Part II + III combined) score at baseline, and CGI-S at baseline will be summarized using descriptive statistics for the ITT population. Further tabulation by region and country will also be presented.

# 5.7. Medical and Psychiatric History

Medical and psychiatric history events will be mapped to a Medical Dictionary for Regulatory Activities (MedDRA) version 27.0 or higher preferred term and system organ class.



Medical and psychiatric history will be summarized by treatment group using preferred terms and system organ classes. All events will be listed.

# **5.8.** Exposure to Treatment

The number of days on study drug, reasons for premature discontinuation of IMP, treatment compliance, days in each phase (Titration and Maintenance), and average dose in each phase, will be summarized by treatment group for the FAS Population. Exposure data, including dose level as received, will be listed.

## 5.9. Primary Efficacy Analysis

## 5.9.1. Primary Estimand

The key research question for the primary endpoint will be addressed with an estimand based on the following attributes:

- 1) Treatments: treatments as randomized regardless of the actual treatment received or the final dose level achieved following the titration steps.
- 2) Target study population of interest: subjects in the modified intent-to-treat (mITT) population regardless the completion status of dose titration steps.
- 3) Endpoint (variable) of interest: change from baseline to Week 26 in the MDS-UPDRS Part II + III Combined Score.
- 4) Population level summary of interest: estimated mean difference between each tavapadon dose group and placebo group in the endpoint of interest.
- 5) Strategy for Intercurrent events (ICEs): a hypothetical strategy will be used to address intercurrent events (ICEs) of potential death, treatment discontinuations, missed visits/assessments, and start of prohibited concomitant Parkinson's disease medications. The data after treatment discontinuations or after the start of prohibited Parkinson's disease concomitant medications will be censored under the hypothetical strategy. Prohibited Parkinson's disease concomitant medications are defined as medications in ATC classifications of ADAMANTANE DERIVATIVES, DOPAMINE AGONISTS, MONOAMINE OXIDASE B INHIBITORS, OTHER ANTIPARKINSON DRUGS, OTHER DOPAMINERGIC AGENTS, or DOPA AND DOPA DERIVATIVES that are started after the first dose of IMP and prior to the last dose of IMP with duration of use 7 days or more. The hypothetical strategy allows the study to assess the effect of tavapadon treatment without the confounding effect of prohibited concomitant Parkinson's disease treatments.



#### 5.9.2. Main Analytical Approach

The change from baseline to each study visit in MDS-UPDRS Part II and III combined score will be summarized by visit and treatment group. A mixed model repeated measures (MMRM) analysis will be used to analyze the data from all post-randomization timepoints up to Week 27 with fixed effect of treatment group, visits, interaction between treatment group and visit, and baseline MAO-B inhibitor use. The baseline value of MDS-UPDRS Part II and III combined score will also be included as a covariate. Subject will be included as a random effect. An unstructured covariance structure will be used for the repeated measures. If the unstructured covariance matrix results in convergence issue, the heterogeneous Toeplitz covariance structure followed by the heterogeneous first-order autoregressive (AR(1)) structure will be used. The Kenward-Roger approximation will be used to estimate the denominator degrees of freedom. The difference between each active dose and placebo at the endpoint visit (Week 26) will be estimated based on the Least Squares Mean (LSMean) difference derived from the MMRM with the associated 95% confidence intervals (CI) and P-values. A Cohen's D value will also be derived as the ratio of the estimated difference to the population standard deviation at each visit estimated from the model (the square root of the diagonal elements of the estimated covariance matrix). The missing values, including missing due to missed visits or early termination due to COVID-19 control measures, are assumed to be missing at random (MAR) in the main MMRM analysis. Sensitivity analyses will be performed to assess the impact of deviation from MAR assumptions on the analysis results. Time curve plots will be presented for both raw Mean (SEM) and LSMean (SE).

#### **5.9.3.** Sensitivity Analyses

#### **5.9.3.1.** Treatment Effect at Final Dose Levels

To assess the treatment effect at the final dose level, a sensitivity analysis will be conducted on the mITT set using the MMRM analysis method described in Section 5.9.2 with treatment defined as the actual final dose level achieved. The final dose level is defined as the dose received at the Week 26 timepoint or at the time of early termination if the subject achieved a minimum of 5 mg prior to discontinuation.

#### 5.9.3.2. Treatment Effect based on Actual Treatment Received

Should a discrepancy between the study treatment received and the randomized treatment assignment occurred in 6 or more subjects, a sensitivity analysis may be conducted based on the study treatments that subjects actually received using the MMRM analysis method described in Section 5.9.2.

#### 5.9.3.3. Remote Assessments Excluded (treated as missing)

In addition, a sensitivity analysis excluding the MDS-UPDRS Part II + Part III combined score obtained remotely may be performed if such remote assessments are conducted due to COVID-19 restrictions. It should be noted that the study only has provision of remote assessments for Parts I & II of the MDS-UPDRS assessments, as the clinician administered motor examination required for Part III cannot be reliably completed remotely.



#### 5.9.3.4. Impact of Missing Values Handling

Whilst every effort will be made to prevent avoidable missing values during the study conduct (National Research Council, 2010), it is unrealistic to expect no missing values in clinical trials. The impact of missing values on the analysis results will be assessed by the sensitivity analyses described below.

#### Under Missing at Random (MAR) Assumption

Multiple imputation (MI) will be performed to replace each missing value with a set of plausible values that represent the uncertainty about the correct value to impute. The Markov chain (MCMC) method will be utilized for the mITT set. SAS PROC MI will be used to generate 27 possible imputed datasets: Each of these datasets will be analyzed using PROC MIXED in SAS using the MMRM model as described in Section 5.9.2. The results of the analyses of the datasets will be combined using PROC MIANALYZE to produce an inferential result.

#### Considerations of Data Potentially Missing Not at Random (MNAR)

A pattern mixture model (PMM) approach will be used to address potentially MNAR patterns. The following three patterns of subjects in the mITT set will be considered:

- 1) Subjects with no missing values from discontinuation or from initiation of prohibited Parkinson's disease concomitant mediation during treatment period.
- 2) Subjects with missing values from the types of ICEs below will be considered having MNAR
  - a. Subjects who discontinue due to reasons, as recorded on the eCRF, of lack of efficacy, adverse events associated with motor symptoms of Parkinson's disease, physician decision, and withdrawal by subject.
  - b. Subjects who initiated concomitant Parkinson's disease medications (ATC classifications of ADAMANTANE DERIVATIVES, DOPAMINE AGONISTS, MONOAMINE OXIDASE B INHIBITORS, OTHER ANTIPARKINSON DRUGS, OTHER DOPAMINERGIC AGENTS, or DOPA AND DOPA DERIVATIVES) after the first dose of IMP and prior to the last dose of IMP with a use duration of 7 days or more will be considered having a potential confounding ICE. The efficacy data post ICE will be treated as missing with the missing pattern of MNAR.

The MNAR cases will be identified and documented prior to database lock and unblinding (Section 9.5).

- 3) Subjects with missing values from the type of ICEs below will be considered as having MAR
  - a. Missing values after discontinuation due to reasons, as recorded on the eCRF, of death, pregnancy, loss to follow-up, adverse event unrelated to motor symptoms of Parkinson's disease, non-compliance, site termination, protocol deviation, failure to meet continuation criteria and other will be considered as MAR.

The MNAR pattern 2) above in the active treatment group will be imputed using the jump to reference (J2R) method (Cro et. al. 2020) by assuming that patients jump to behave like those in the placebo group following their last observed time point. However, such MNAR in the placebo group will still be imputed as MAR using the standard multiple imputation method.

The MAR patterns 3) will be imputed using the standard multiple imputation method described above.

Other missing values due to missed visits/assessments before endpoint or discontinuation will also be assumed as MAR and imputed using the standard multiple imputation method for all three patterns.

Core codes for MAR and MNAR imputations are provided in Section 9.6.

#### Under Missing Completely at Random (MCAR) Assumption

An additional sensitivity analysis will be conducted on the Endpoint (Week 26) Completer set using the MMRM analysis method described in Section 5.9.2.

#### 5.9.4. Subgroup Analyses

Subgroup analyses of the primary endpoint will be made based on the mITT set to assess consistency of the intervention effect across the following subgroups:

- Age group:  $< 65 \text{ vs} \ge 65 \text{ years}$
- Sex: female vs male
- Hoehn and Yahr Status at screening: 1 vs 1.5 vs 2
- Baseline MDS-UPDRS Part II score: ≤ baseline median vs > baseline median (median of the mITT set regardless of treatment group)
- Baseline MDS-UPDRS Part III score: ≤ baseline median vs > baseline median (median of the mITT set regardless of treatment group)
- Use of concomitant MAO-B inhibitor: yes vs no
- Years since initial diagnosis: (<1 year vs 1 to < 2 years vs 2 to < 3 years
- Race: white vs other
- Region: United States vs Non-US

If the number of subjects within a subgroup is too small (less than 10% of the mITT set), the subgroup categories may be redefined prior to unblinding the study or the specific subgroup analysis may not be performed. Provided that the sample sizes in the subgroups allow, the MMRM analysis method described in Section 5.9.2 will be applied to the subgroup analysis (excluding the covariate of MAO-B inhibitor use in the MAO-B subgroup models). The treatment effect across subgroups will be summarized by forest plots.

## 5.10. Key Secondary Efficacy Analyses

#### 5.10.1. Secondary Estimand 1

The key research question for the first secondary efficacy variable will be addressed with an estimand based on the following attributes:

- 1) Treatments: treatments as randomized regardless of the actual treatment received or the final dose level achieved following the titration steps.
- 2) Target study population of interest: subjects in the modified intent-to-treat (mITT) population regardless the completion status of dose titration steps.
- 3) Endpoint (variable) of interest: change from baseline to Week 26 in the MDS-UPDRS Part II Score.
- 4) Population level summary of interest: estimated mean difference between each tavapadon (CVL-751) dose group and placebo group in the endpoint of interest.
- 5) Strategy for Intercurrent events (ICEs): a hypothetical strategy will be used to address intercurrent events (ICEs) of potential death, treatment discontinuations, missed visits/assessments, and start of prohibited concomitant Parkinson's disease medications (see definitions in Section 5.9.1). The data after treatment discontinuations or after the start of prohibited concomitant Parkinson's disease treatments will be censored under the hypothetical strategy.

## 5.10.1.1. Main Analytical Approach

Similar to the analysis of the primary efficacy variable, the change from baseline to each study visit in MDS-UPDRS Part II score will be summarized by visit and treatment group. A mixed model repeated measures (MMRM) analysis will be used with fixed effect of treatment group, visits, and interaction between treatment group and visit, and MAO-B inhibitor use. The baseline value of MDS-UPDRS Part II score will be included as a covariate. Subject will be included as a random effect. An unstructured covariance structure will be used for the repeated measures. If the unstructured covariance matrix results in convergence issue, the heterogeneous Toeplitz covariance structure followed by the heterogeneous first-order autoregressive (AR(1)) structure will be used. The Kenward-Roger approximation will be used to estimate the denominator degrees of freedom. The difference between each active dose and placebo at the endpoint visit (Week 26) will be estimated based on the Least Squares Mean (LSMean) difference derived from the MMRM with the associated 95% confidence intervals (CI) and P-values. A Cohen's D value will also be derived as the ratio of the estimated difference to the population standard deviation at each visit estimated from the model (the square root of the diagonal elements of the estimated covariance matrix). The missing values, including missing due to missed visits or early termination due to COVID-19 control measures, are assumed to be missing at random (MAR) in the main MMRM analysis. Sensitivity analyses will be performed to assess the impact of deviation from MAR assumptions on the analysis results. Time curve plots will be presented for both raw Mean (SEM) and LSMean (SE).

#### 5.10.1.2. Sensitivity Analyses

The sensitivity analyses described in Section 5.9.3 for the primary estimand will also be performed for the secondary efficacy estimand 1.

#### 5.10.1.3. Subgroup Analyses

The subgroup analyses described in Section 5.9.4 for the primary estimand will also be performed for the secondary efficacy estimand 1.

## 5.10.2. Secondary Estimand 2

The key research question for the second secondary efficacy variable will be addressed with an estimand based on the following attributes:

- 1) Treatments: treatments as randomized regardless of the actual treatment received or the final dose level achieved following the titration steps.
- 2) Target study population of interest: subjects in the modified intent-to-treat (mITT) population regardless the completion status of dose titration steps.
- 3) Endpoint (variable) of interest: proportion of responders, defined as subjects with a score of "much improved" or "very much improved" on the PGIC, at Week 26.
- 4) Population level summary of interest: : estimated difference expressed as odds ratio between each tavapadon (CVL-751) dose group and placebo group in achieving response.
- 5) Strategy for Intercurrent events (ICEs): a hypothetical strategy will be used to address intercurrent events (ICEs) of potential death, treatment discontinuations, missed visits/assessments, and start of prohibited concomitant Parkinson's disease medications (see definitions in Section 5.9.1). The data after treatment discontinuations or after the start of prohibited concomitant Parkinson's disease treatments will be censored under the hypothetical strategy.

#### 5.10.2.1. Main Analytical Approach

The number and percentage of responders will be summarized by visit and treatment group. The binomial repeated measures up to Week 27 will be analyzed using a generalized linear mixed model with logit link (SAS® GLIMMIX procedure). The treatment group, MAO-B inhibitor use, visits, and interaction between treatment group and visit will be included as fixed effect. An unstructured covariance structure will be used for the repeated measures. If the model does not converge with the unstructured covariance structure, the heterogeneous Toeplitz structure will be used. The odds ratio of each active dose to placebo at the endpoint visit will be estimated based on the Least Squares Mean difference in logit between the treatment groups from the GLIMMIX model with the associated 95% confidence intervals (CI) and P-values. The missing values are assumed to be missing at random, including missing due to missed visits or early termination due to COVID-19 control measures. Sensitivity analyses will be performed to assess the impact of deviation from MAR assumptions on the analysis results.


# 5.10.2.2. Sensitivity Analyses

The sensitivity analyses described in Section 5.9.3 for the primary estimand will also be performed for the secondary efficacy estimand 2 except for the sensitivity analyses to assess the impact of missing value handling. For the secondary efficacy estimand 2, the case of potential MNAR will be imputed as "non-responder" for the sensitivity analysis. No additional sensitivity analysis under the MAR assumption using multiple imputations will be performed. In addition, a sensitivity analysis excluding the PGIC score obtained remotely may be performed if such remote assessments are conducted due to COVID-19 restrictions.

# 5.10.2.3. Subgroup Analyses

The subgroup analyses described in Section 5.9.4 for the primary estimand will also be performed for the secondary efficacy estimand 2: proportion of responders at Week 26.



# 5.11. Summary of Primary and Key Secondary Efficacy Analyses

| ICE Strategy | Primary Analysis | Sensitivity Analysis | Subgroup Analysis |
|---|---|---|---|
| Primary Endpoint | : Change from baselin | e in the MDS UPDRS Part II + III c | ombined score at Week 26 |
| Hypothetical strategy with data after treatment discontinuations or after the start of prohibited concomitant medications censored | <ul> <li>mITT population</li> <li>Treatment as randomized</li> <li>MMRM described in Section 5.9.2</li> </ul> | Treatment effect at final dose levels Treatment effect based on actual treatment received, if applicable Missing values imputation using multiple imputations (MI) Missing values imputation using pattern mixture model (PMM) Endpoint completer analysis Analysis with remote assessments excluded (treated as missing) | <ul> <li>Age</li> <li>Sex</li> <li>Hoehn&amp;Yahr Status</li> <li>MAO-B inhibitor use</li> <li>Baseline MDS-UPDRS Part II and Part III baseline</li> <li>Years since diagnosis</li> <li>Race</li> <li>Region</li> </ul> |
| Key Secondary En | dpoint 1: Change from | n baseline in the MDS UPDRS Part | II score at Week 26 |
| Hypothetical strategy with data after treatment discontinuations or after the start of prohibited concomitant medications censored | <ul> <li>mITT population</li> <li>Treatment as<br/>randomized</li> <li>MMRM described<br/>in Section 5.9.2</li> </ul> | Treatment effect at final dose levels Treatment effect based on actual treatment received, if applicable Missing values imputation using multiple imputations (MI) Missing values imputation using pattern mixture model (PMM) Endpoint completer analysis Analysis with remote assessments excluded (treated as missing) | Age Sex Hoehn&Yahr Status MAO-B inhibitor use Baseline MDS-UPDRS Part II and Part III baseline Years since diagnosis Race Region |
| Key Secondary En | dpoint 2: Proportion | of PGIC responders at Week 26 | |
| Hypothetical<br>strategy with data<br>after treatment<br>discontinuations<br>or after the start<br>of prohibited<br>concomitant<br>medications<br>censored | <ul> <li>mITT population</li> <li>Treatment as randomized</li> <li>GLIMMIX model described in Section 5.10.2.1</li> </ul> | Treatment effect at final dose levels Treatment effect based on actual treatment received, if applicable Potential MNAR missing values treated as non-responders Endpoint completer analysis Analysis with remote assessments excluded (treated as missing) | Age Sex Hoehn&Yahr Status MAO-B inhibitor use Baseline MDS-UPDRS Part II and Part III baseline Years since diagnosis Race Region |



# **5.12.** Other Efficacy Analyses

| Endpoint | Analysis<br>Population | ICE Strategy | Analysis Method | Subgroup Analysis |
|---|---|---|---|---|
| | • | Seconda | ry Endpoints | |
| Change from<br>baseline in the MDS<br>UPDRS Part II + III<br>combined score (all<br>time points) | mITT | Hypothetical | MMRM described in Section 5.9.2 | <ul> <li>Age</li> <li>Sex</li> <li>Hoehn&amp;Yahr Status</li> <li>MAO-B inhibitor use</li> <li>Baseline MDS-UPDRS Part II and Part III baseline</li> <li>Years since diagnosis</li> <li>Race</li> <li>Region</li> </ul> |
| Change from<br>baseline in the MDS<br>UPDRS Part I,<br>Part II, and Part III<br>combined score (all<br>time points) | mITT | Hypothetical | MMRM described in Section 5.9.2 | <ul> <li>Age</li> <li>Sex</li> <li>Hoehn&amp;Yahr Status</li> <li>MAO-B inhibitor use</li> <li>Baseline MDS-UPDRS Part II and Part III baseline</li> <li>Years since diagnosis</li> <li>Race</li> <li>Region</li> </ul> |
| Change from<br>baseline in the MDS<br>UPDRS Part I score<br>(all time points) | mITT | Hypothetical | MMRM described in Section 5.9.2 | <ul> <li>Age</li> <li>Sex</li> <li>Hoehn&amp;Yahr Status</li> <li>MAO-B inhibitor use</li> <li>Baseline MDS-UPDRS Part II and Part III baseline</li> <li>Years since diagnosis</li> <li>Race</li> <li>Region</li> </ul> |
| Change from<br>baseline in the MDS<br>UPDRS Part II<br>score (all time<br>points) | mITT | Hypothetical | MMRM described in Section 5.9.2 | <ul> <li>Age</li> <li>Sex</li> <li>Hoehn&amp;Yahr Status</li> <li>MAO-B inhibitor use</li> <li>Baseline MDS-UPDRS Part II and Part III baseline</li> <li>Years since diagnosis</li> <li>Race</li> <li>Region</li> </ul> |



| Endpoint | Analysis<br>Population | ICE Strategy | Analysis Method | Subgroup Analysis |
|---|---|---|---|---|
| Change from<br>baseline in the MDS<br>UPDRS Part III<br>score (all time<br>points) | mITT | Hypothetical | MMRM described in Section 5.9.2 | <ul> <li>Age</li> <li>Sex</li> <li>Hoehn&amp;Yahr Status</li> <li>MAO-B inhibitor use</li> <li>Baseline MDS-UPDRS Part II and Part III baseline</li> <li>Years since diagnosis</li> <li>Race</li> <li>Region</li> </ul> |
| Change from<br>baseline in the<br>CGI-S score (all<br>time points) | mITT | Hypothetical | MMRM described in Section 5.9.2 | <ul> <li>Age</li> <li>Sex</li> <li>Hoehn&amp;Yahr Status</li> <li>MAO-B inhibitor use</li> <li>Baseline MDS-UPDRS Part II and Part III baseline</li> <li>Years since diagnosis</li> <li>Race</li> <li>Region</li> </ul> |
| CGI-I score (all time points) | mITT | Hypothetical | MMRM described in Section 5.9.2 | <ul> <li>Age</li> <li>Sex</li> <li>Hoehn&amp;Yahr Status</li> <li>MAO-B inhibitor use</li> <li>Baseline MDS-UPDRS Part II and Part III baseline</li> <li>Years since diagnosis</li> <li>Race</li> <li>Region</li> </ul> |
| PGIC score (all time points) | mITT | Hypothetical | MMRM described in Section 5.9.2 | <ul> <li>Age</li> <li>Sex</li> <li>Hoehn&amp;Yahr Status</li> <li>MAO-B inhibitor use</li> <li>Baseline MDS-UPDRS Part II and Part III baseline</li> <li>Years since diagnosis</li> <li>Race</li> <li>Region</li> </ul> |



| Endpoint | Analysis<br>Population | ICE Strategy | Analysis Method | Subgroup Analysis |
|---|---|---|---|---|
| Other Endpoints | | | | |
| Change from baseline in the PDQ 39 score | mITT | Hypothetical | MMRM described in Section 5.9.2 | None |
| Change from<br>baseline in the<br>Schwab and<br>England ADL score | mITT | Hypothetical | MMRM described in Section 5.9.2 | None |
| Change from baseline in the EQ-5D-5L index score | mITT | Hypothetical | MMRM described in Section 5.9.2 | None |
| Change from<br>baseline in<br>EQ-5D-5L VAS<br>score | mITT | Hypothetical | MMRM described in Section 5.9.2 | None |

Cohen's D effect size by time point will be derived for MDS-UPDRS Part II+III and MDS-UPDRS Part II only. Time curve plots will be presented for LSMean (SE) of change from baseline for MDS-UPDRS Part II+III, Part I+II+III, individual Part I, II and III, CGI-S, and Schwab and England ADL scores as well as for LSMean (SE) of CGI-I and PGIC over time.

# 5.13. Interim and Final Analysis

A final analysis will be conducted once the last subject completes or discontinues the study, and the resulting clinical database has been cleaned, quality checked, and the database has been locked.

No interim analysis is planned.

# 5.14. Safety Analyses

All safety analyses will be performed on the full analysis set (FAS). Should any subjects receive a treatment other than their randomized treatment, the treatment as received will be used in the safety presentation.

#### **5.14.1.** Adverse Events

Adverse events will be mapped to a Medical Dictionary for Regulatory Activities (MedDRA) version 27.0 or higher preferred term and system organ class. If a subject experiences multiple events that map to a single preferred term, the greatest severity and strongest investigator assessment of relation to IMP will be assigned to the preferred term for the appropriate summaries. Events with missing severity or relationship will be classified as outlined in Section 3.2. Missing onset dates will be imputed as previously outlined in Section 4.1 as required to determine treatment-emergent events.



Summaries of treatment-emergent AEs will include any AEs reported beginning with the initiation of study drug on Day 1 through end of reporting period specified in the protocol post the last dose of IMP. The occurrence of TEAEs will be summarized by treatment group using preferred terms, system organ classes, and severity. The TEAEs by subgroup of MAO-B inhibitor use will be summarized by treatment, organ class, and preferred term. Separate summaries of treatment-emergent serious adverse events (TESAEs), TEAEs related to IMP, AESIs (including AEs related to abuse potential and AEs involving medication handling irregularities), events leading to the discontinuation of IMP, and AESIs that did not result in discontinuation of IMP or study will be generated respectively. A summary of AEs by treatment phase and by dose at event onset will also be presented. Adverse events leading to the discontinuation of IMP by preferred term and phase at onset will be prepared. All adverse events reported will be listed for individual subjects showing both verbatim and preferred terms. All adverse events that occurred prior to the initiation of study treatment or after the protocol-specified reporting period post the last dose of IMP will be excluded from the summary tables but will be included in the listings.

In addition, TEAEs rate per 100 person-years of exposure (PYE) will be summarized by treatment group using system organ class and preferred term. TEAEs with  $\geq$ 2% incidence in either tavapadon dose group and a greater incidence than the placebo group will be summarized by treatment group using preferred term in descending order of the incidence in the tavapadon15 mg group followed by that in the tavapadon 5 mg group. The most common TEAEs, defined as an incidence  $\geq$ 5% in either tavapadon dose group and greater than 2 times of the incidence in the placebo group, will also be summarized by treatment group using preferred term in descending order of the incidence in the tavapadon15 mg group followed by that in the tavapadon 5 mg group.

## **5.14.2.** Epworth Sleepiness Scale (ESS)

The ESS individual questions and total score and corresponding changes from baseline will be summarized by treatment group and study visit. The percentage of subjects with sleepy (10 or more) and very sleepy (18 or more) scores will also be summarized. ESS individual question score as well as the total score will be presented in a listing. The ESS total score will also be analyzed using the same method (MMRM analysis) describer in Section 5.9.2 to explore any treatment difference in sleepiness. Time curve plot will be presented for LSMean (SE) of change from baseline.

# 5.14.3. Questionnaire for Impulsive-Compulsive Disorders in Parkinson Disease Rating Scale (QUIP-RS)

The QUIP-RS component scores (Gambling, Sex, Buying, Eating, Hobbyism-Punding, PD Medication Use), total ICD score, and total score and corresponding changes from baseline will be summarized by treatment group and study visit. QUIP-RS individual data will be presented in a listing. The total ICD score will also be analyzed using the same method (MMRM analysis) describer in Section 5.9.2 to explore any treatment difference in impulsive-compulsive behaviors. Time curve plots will be presented for LSMean (SE) of change from baseline.



### 5.14.4. Non-IMP Medications and Non-Drug Therapy/Procedures

The use of non-IMP medications will be coded using the World Health Organization (WHO) drug dictionary (WHODrug) (Version: Global B3 September 2019 or later). Concomitant medications, with start date on or after the date of the first IMP through the last IMP dose date, will be summarized by treatment group, frequency of drug classification, and generic drug name. Medications with start date after the last dose of IMP through the end of protocol-defined reporting period, will also be summarized. Prior medications use will be similarly summarized. All prior, concomitant, and post IMP medications will be presented in a data listing.

The use of non-drug therapy/procedures will be coded using MedDRA Version 27.0 or higher. Concomitant and post-IMP non-drug therapy/procedures will be summarized by treatment group, frequency of system organ class and preferred term. All non-drug therapy/procedures will be presented in a data listing.

#### **5.14.5.** Clinical Laboratory Assessments

Descriptive summaries of selected (quantitative) clinical laboratory results will be presented by treatment group and study visit. Laboratory values outside the normal range for each systematically collected hematology, blood chemistry, and urinalysis parameter will be identified. Each subject's hematology, blood chemistry, and quantitative urinalysis values will be flagged as "low" (below the lower limit of normal/LLN), "normal" (within the normal range), or "high" (above the upper limit of normal/ULN) relative to the normal ranges of the central laboratory. Each subject's qualitative urinalysis results will be flagged as "normal" or "abnormal". In addition, the severity of laboratory abnormality will be graded based on toxicity criteria specified in Section 9.8 in reference to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. The result of each laboratory test for individual subjects will be presented in a listing with the normal range defined by the central laboratory, the status relative to the normal range, and the toxicity grade.

Shift table will be used to summarize shifts from baseline toxicity grades to greatest (worst) treatment-emergent laboratory toxicity grade. For hematology and, blood chemistry, and quantitative urinalysis parameters that toxicity grade was not defined, a shift table for each laboratory test will be based on the shift from baseline high/normal/low status to the status of the maximum post-baseline value and the minimum post-baseline value (including test results from unscheduled visits, if any). Similarly, for qualitative urinalysis parameters, shifts from baseline normal/abnormal status to the worst post-baseline status will be summarized.

The number and percentage of subjects who have post-baseline elevations in liver transaminase (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]) or bilirubin abnormalities in relation to fold above the upper limit of normal will be summarized according to the Food and Drug Administration's Premarketing Clinical Evaluation on Drug-Induced Liver Injury Guidance for Industry (FDA 2009). Abnormal hepatic laboratory values will be categorized and evaluated for any occurrence among all post-baseline assessments (where "and" in the bulleted list below indicates elevations occurring at the same visit). Within each laboratory parameter grouping, a subject may be counted once per elevation criteria using the worst-case result.

That is, a subject with a worst case ALT elevation  $> 5 \times$  the ULN would be counted once in the ALT  $> 3 \times$  ULN category and once in the ALT  $> 5 \times$  ULN category, regardless of how many ALT elevations the subject had that met the  $> 3 \times$  ULN and  $> 5 \times$  ULN elevation criteria.

- ALT and/or AST  $> 3 \times ULN$  and total bilirubin > 1.5 or  $2 \times ULN$
- AST  $> 3, 5, 10, 20 \times ULN$
- ALT  $> 3, 5, 10, 20 \times ULN$
- Total bilirubin  $> 1.5, 2 \times ULN$
- Alkaline phosphatase (ALP)  $> 1.5 \times ULN$

In addition, an eDISH plot, a shift plot showing liver safety panel tests over time (baseline vs. post-baseline), and distribution plots of ALT, AST, ALP, and bilirubin over time will be produced to aid identification of any potential cases (Merz M. et. al. 2014). The plots to be included are the scatter plot of maximum transaminase versus maximum bilirubin, the liver test safety panel over time, and the distribution of ALT by time. The distribution plots for AST, ALP, and bilirubin will use the same format as used for ALT.

### **5.14.6. Vital Signs**

Vital signs include systolic and diastolic blood pressures, heart rate, and body temperature. Supine (after 5 minutes of rest) and standing (2 minutes after rising from supine to standing) measurements will be obtained for blood pressure and heart rate. Duplicate readings of supine blood pressure and heart rate will be taken. The duplicate values will be individually recorded, and the values will be averaged by the sponsor for the time point assessment. Orthostatic changes will be derived using standing and supine values. Body temperature will be obtained once, at the time of the first blood pressure measurement.

#### **5.14.6.1.** Blood Pressure and Heart Rate

Blood pressure and heart rate measurements and corresponding changes from baseline will be summarized by treatment group, position (if applicable), and visit using descriptive statistics. The distribution of diastolic and systolic blood pressure over time will be evaluated using box plots. Average records will be used for the analysis where available.

Number and percent of subjects with at least one of the out-of-range value in blood pressure and heart rate will be summarized by treatment group based on the following criteria:

Supine Systolic Blood Pressure (mmHg)

- < 80 mmHg
- < 90 mmHg
- > 140 mmHg
- > 160 mmHg
- > 200 mmHg



Change from Baseline in Supine Systolic Blood Pressure (mmHg)

- < -20 mmHg
- < -10 mmHg
- > 10 mmHg
- > 20 mmHg

Orthostatic Systolic Blood Pressure (mmHg)

- $\geq$  20 mmHg decrease upon standing compared with supine position
- $\geq$  20 mmHg increase upon standing compared with supine position

Supine Diastolic Blood Pressure (mmHg)

- < 50 mmHg
- > 90 mmHg
- > 100 mmHg
- > 120 mmHg

Change from Baseline in Supine Diastolic Blood Pressure (mmHg)

- < -15 mmHg
- < -10 mmHg
- > 10 mmHg
- > 25 mmHg

Orthostatic Diastolic Blood Pressure (mmHg)

- $\geq 10$  mmHg decrease upon standing compared with supine position
- $\geq$  10 mmHg increase upon standing compared with supine position

Supine Heart Rate (beats/min)

- < 50 bpm
- < 60 bpm
- > 100 bpm and  $\le 120$  bpm
- > 120 bpm

The number and percentage of the out-of-range values will also be summarized by treatment phase (titration and maintenance phase). For supine measurements, the average of the duplicate will be used to determined out-of-range status, unless in isolated cases where only a single measurement was taken.

### **5.14.6.2. Body Weight**

Body weight measurements at baseline and at the end of treatment with corresponding changes from baseline will be summarized by treatment group using descriptive statistics.

Number and percent of subjects with out-of-range body weight changes will be summarized based on the following criteria:

- Decrease from Baseline 7% or more (i.e. change from baseline  $\leq$  -7%)
- Increase from baseline 7% or more (i.e. change from baseline  $\geq$ 7%)

# **5.14.6.3. Temperature**

Temperature and corresponding changes from baseline will be summarized by treatment group, and visit using descriptive statistics. Number and percent of subjects with out-of-range temperature will be summarized based on the following criteria:

- >38.0 °C
- <36.0 °C

# 5.14.7. Electrocardiograms (ECGs)

Single or triplicate 12 lead ECGs will be obtained during the trial. All ECG recordings will be obtained after the subject has been supine and at rest for at least 5 minutes. A triplicate set of ECGs is 3 consecutive ECGs collected 1 to 2 minutes apart over a 5 minute period. Any values taken in triplicate will be averaged for analysis. ECGs and corresponding changes from baseline will be summarized by treatment group and visit using descriptive statistics. Average records will be used for the analysis where available.

The number and percentage of subjects who experience any post-baseline occurrence of potentially clinically significant corrected QT values using Fridericia's method (QTcF) will be summarized by treatment group. These presentations will include QTcF values > 450 to  $\leq$  480, > 480 to  $\leq$  500, and > 500 msec; or changes of > 30 to  $\leq$  60 or > 60 msec (FDA, 2005). For this categorization, the average of triplicate values will be utilized rather than the individual values comprising the triplicate measurement. An out-of-range categorical tabulation will also be presented for the subgroup of U.S subjects.

Additionally, a distribution plot of QTcF over time will be presented as an aid in identification of any possible time trend and outliers.

A substudy to evaluate the effect of tavapadon on the QT interval using C-QT modelling is also included in this trial. Matched triplicate ECGs and plasma tavapadon concentrations that are collected at preselected sites will be used to characterize the effects of tavapadon on the QT interval. The analysis plan is summarized separately.

#### **5.14.8.** Physical and Neurological Examinations

Physical and Neurological examination data will be listed.

### 5.14.9. Columbia-Suicide Severity Rating Scale (C-SSRS)

The maximum post-baseline results from the C-SSRS will be summarized. The maximum of each subscale (suicidal ideation [Categories 1-5], suicidal behavior [Categories 6-10], suicidal ideation or behavior [Categories 1-10], and self-injurious behavior without suicidal intent) will be presented. The number of patients with suicide-related treatment-emergent events, treatment-emergent suicidal ideation, and suicidal behavior, based on a comparison of the C-SSRS at baseline and/or previous lifetime experience to maximum C-SSRS scores across all post-baseline assessments will be provided. All C-SSRS elements will be reflected in a listing.

#### 5.15. Pharmacokinetics

Plasma concentrations of tavapadon and CV-0000053 (metabolite) will be determined using a validated LC-MS/MS method. PK data listings will be presented for the PK population. PK summary tables and mean figures will be presented using the PK analysis set.

# 5.15.1. Pharmacokinetic Data Analysis

Plasma concentrations of tavapadon and CV-0000053 (metabolite) will be summarized separately using descriptive statistics by visit. Plasma concentrations of tavapadon and CV-0000053 that are <LLOQ will be reported as 'BLQ' in the data listings. Plasma concentrations that are BLQ will be treated as 0 for calculation of descriptive statistics. The geometric mean, however, will be calculated by imputing BLQ values as ½ LLOQ. If the calculated mean concentration is below the limit of quantitation, the mean will be reported as BLQ and the SD and CV% shall be reported as not determined (ND). Mean plasma concentrations (SD) of tavapadon and CV-0000053 will also be plotted versus time (in both linear and semi-logarithmic scale) based on nominal visit.

### **5.16.** Protocol Deviations

All protocol deviations will be reviewed by the project team prior to database lock and unblinding to identify subjects with important protocol deviations. The number and percentage of subjects with important deviations will be tabulated by treatment and further tabulated by category and treatment. All deviations from the protocol will be listed by category along with a description and any additional comments.



# 6. CHANGES IN THE PLANNED ANALYSES

Should any deviations from the analyses specified in the final approved (prior to database lock and unblinding) statistical analysis plan arise, such deviations will be documented in the final clinical study report.



# 7. REVISION HISTORY

| Date | Revision | Rationale |
|------|----------|-----------|



#### 8. REFERENCES

Cro S, Morris TP, Kenward MG, Carpenter JR. Sensitivity analysis for clinical trials with missing continuous outcome data using controlled multiple imputation: A practical guide. Statistics in Medicine. 2020;39:2815–2842.

Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, et al. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008;15;23(15):2129-70.

Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, et al. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011; 20(10):1727–36.

Merz M, Lee KR, Kullak-Ublick GA, Brueckner A, Watkins PB. Methodology to Assess Clinical Liver Safety Data. Drug Saf (2014) 37 (Suppl 1):S33–S45

National Research Council. The Prevention and Treatment of Missing Data in Clinical Trials; 2010.

Peto V, Jenkinson C, Fitzpatrick R. PDQ-39: a review of the development, validation and application of a Parkinson's disease quality of life questionnaire and its associated measures. J Neurol. 1998 May;245 Suppl 1:S10-4.

US Food and Drug Administration (FDA). Guidance for Industry: Drug-Induced Liver Injury: Premarketing Clinical Evaluation; 2009.

US Food and Drug Administration (FDA). Guidance for Industry: E14 Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs, 2005.

van Hout B, Janssen MF, Feng YS, Kohlmann T, Busschbach J, Golicki D, Lloyd A, Scalone L, Kind P, Pickard AS. Interim scoring for the EQ-5D-5L: mapping the EQ-5D-5L to EQ-5D-3L value sets. Value Health. 2012 Jul-Aug;15(5):708-15.



# 9. APPENDICES



# 9.1. Schedule of Assessments

# **Table 5:** Schedule of Assessments

| Trial Period: | Screen | Baseline | | | | | Treatn | nent | | | | Safety<br>Follow-up <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Week: | -4 to -1 | 1 | 2 | 5 | 8 | 11 | 14 | 18 | 22 | 26 | 27 <sup>b</sup> | 31 |
| Trial Day: | -31 to -1 | 1 | 14±3 | 35±3 | 56±3 | 77±3 | 98±3 | 126±3 | 154±3 | 182±3 | 189±3 | 217±3 |
| Visit/Contact: | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 | Visit 10 | Visit 11<br>(EOT/ET) | Telephone <sup>c</sup> |
| Entrance and History | l | | | | | | | | | l | <u>'</u> | |
| Informed consent <sup>d</sup> | X | | | | | | | | | | | |
| Eligibility criteria | X | X | | | | | | | | | | |
| Demography | X | | | | | | | | | | | |
| Psychiatric history <sup>e</sup> | <b>←</b> | | | | | | | | | | | |
| Medical history <sup>e</sup> | ← | | | | | | | | | | | |
| Alcohol/illicit drug use inquiry | X | | | | | | | | | | | |
| Modified Hoehn and Yahr stage | X | | | | | | X | | | X | X | |
| MoCA | X | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | |
| Efficacy and Other Endpoint Assessme | ents | | | | | | | | | | | |
| MDS-UPDRS <sup>f</sup> | X | X | | X | X | X | X | X | X | X | X | |
| CGI-S | | X | | X | X | X | X | X | X | X | X | |
| CGI-I <sup>g</sup> | | | | X | X | X | X | X | X | X | X | |
| PGIC <sup>g</sup> | | | | X | X | X | X | X | X | X | X | |
| PDQ-39 | | X | | | | | | | | X | X | |
| Schwab and England ADL | | X | | X | X | X | X | X | X | X | X | |
| EQ-5D-5L | | X | | | | | X | | | X | X | |
| Safety Assessments | I . | | | | | | | ı | ı | ı | ı l | |
| ESS | | X | X | X | X | X | X | X | X | X | X | |



| Trial Period: | Screen | Baseline | | | | | Treatn | nent | | | | Safety<br>Follow-up <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Week: | -4 to -1 | 1 | 2 | 5 | 8 | 11 | 14 | 18 | 22 | 26 | 27 <sup>b</sup> | 31 |
| Trial Day: | -31 to -1 | 1 | 14±3 | 35±3 | 56±3 | 77±3 | 98±3 | 126±3 | 154±3 | 182±3 | 189±3 | 217±3 |
| Visit/Contact: | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 | Visit 10 | Visit 11<br>(EOT/ET) | Telephone <sup>c</sup> |
| QUIP-RS | | X | X | X | X | X | X | X | X | X | X | |
| C-SSRS <sup>h</sup> | X | X | X | X | X | X | X | X | X | X | X | |
| Physical/neurological examination <sup>i</sup> | X | | | | | | | | | | X | |
| Weight | X | X | | | | | | | | | X | |
| Vital signs <sup>j</sup> | X | X | X | X | X | X | X | X | X | X | X | |
| 12-Lead ECGs | | | | | | | | | | | | |
| US sites | | | | | | | | | | | | |
| Single ECG | X | | | | | | | | | | | |
| Three sets of triplicate ECGs <sup>k</sup> (-45, -30, and -15 min prior to first dose of IMP) | | X | | | | | | | | | | |
| One set of triplicate ECGs <sup>k,l</sup> | | X | | X | | X | X | | X | | X | |
| Non-US sites | | | | | | | | | | | | |
| Single ECG <sup>l</sup> | X | X | | X | | X | X | | X | | X | |
| One set of triplicate ECGs <sup>k,l</sup><br>prior to first dose of IMP | | X | | | | | | | | | | |
| Eye examination | | | | | | X <sup>v</sup> | | | | | Xw | |
| Prior/concomitant medications | <b>←</b> | | | | | | | | | | | → |
| Adverse events <sup>m</sup> | | <b>←</b> | | | | | | | | | | <del>-</del> |
| Laboratory <sup>n</sup> | • | | | | | | | | | | | |
| Safety laboratory blood sample | X | X | | | | X | | | X | | X | |
| Prolactin level | | X <sup>u</sup> | | | | | | | | | X <sup>u</sup> | |
| Serology (HIV, HbsAg, and HCV) | X | | | | | | | | | | | |
| Dipstick urinalysis <sup>o</sup> | X | X | | | | X | | | X | | X | |

| Trial Period: | Screen | Baseline | Baseline Treatment | | | | | | | Safety<br>Follow-up <sup>a</sup> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Week: | -4 to -1 | 1 | 2 | 5 | 8 | 11 | 14 | 18 | 22 | 26 | 27 <sup>b</sup> | 31 |
| Trial Day: | -31 to -1 | 1 | 14±3 | 35±3 | 56±3 | 77±3 | 98±3 | 126±3 | 154±3 | 182±3 | 189±3 | 217±3 |
| Visit/Contact: | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 | Visit 10 | Visit 11<br>(EOT/ET) | Telephone <sup>c</sup> |
| Serum pregnancy test <sup>p</sup> | X | | | | | | | | | | | |
| Urine dipstick pregnancy test <sup>p</sup> | | ← | | | | | | | | | | |
| Urine drug screen <sup>q</sup> | X | ← | | | | | | | | | X | |
| Plasma PK sample <sup>r</sup> | | X | | X | | X | X | | X | | X | |
| Future biospecimen research blood sample <sup>s</sup> | | X | | | | | | | | | | |
| IMP Administration and Compliance <sup>t</sup> | | | | | | | | | | | | |
| Dispense IMP | | X | X | X | X | X | X | X | X | X | | |
| Assess IMP compliance | | | X | X | X | X | X | X | X | X | X | |

Abbreviations: ADL = activities of daily living, CGI-I = Clinical Global Impression – Improvement, CGI-S = Clinical Global Impression – Severity of Illness, C-SSRS = Columbia-Suicide Severity Rating Scale, ECG = electrocardiogram, eCRF = electronic case report form, EQ-5D-5L = EuroQol 5 Dimension 5 Level, ESS = Epworth Sleepiness Scale, EOT = end of treatment, ET = early termination, HbsAg = hepatitis B surface antigen, HCV = hepatitis C virus, HIV = human immunodeficiency virus, IMP = investigational medicinal product , MDS-UPDRS = Movement Disorder Society – Unified Parkinson's Disease Rating Scale, MoCA = Montreal Cognitive Assessment, PDQ-39 = 39-Item Parkinson's Disease Questionnaire, PGIC = Patient Global Impression of Change, PK = pharmacokinetic, QUIP-RS = Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale.

- a. Subjects who prematurely discontinue from the trial or who are not eligible for or choose not to participate in the open-label extension trial (Protocol CVL-751-PD-004) are to participate in the 4-week Safety Follow-Up Period. Subjects who proceed into the open-label extension trial will go directly into that trial and will not complete the Safety Follow-Up Period.
- b. The assessments scheduled for the Week 27 visit are to be performed for any subject who prematurely discontinues from the trial.
- c. Contact with subjects via telephone call or other means of communication to check on their status.
- d. Informed consent must be obtained before any trial-related procedures are performed.
- e. Medical occurrences that begin before the start of IMP dosing but after obtaining informed consent will be recorded as medical and/or psychiatric history.
- f. MDS-UPDRS Parts I, II, and III will be conducted before the first dose of IMP at the Baseline Visit and at ~2 to ~6 hours after dosing (at home) at clinic visits during the Treatment Period.
- g. All responses will be relative to the subject's condition at the Baseline Visit (Day 1) before the first dose of IMP.
- h. The "Baseline/Screening" C-SSRS form will be completed at the Screening Visit to determine eligibility. The "Since Last Visit" C-SSRS form will be completed at the Baseline Visit to ensure that the subject continues to qualify for the trial and at all visits after the Baseline Visit.
- i. Full physical and neurological examinations should be completed at the Screening Visit and at Week 27. The physical examination should include height at the Screening Visit only. Physical and/or neurological examinations can be done at any time point during the trial at the investigator's discretion.

Confidential Page 54 of 154 Version 1.0: 31 July 2024



| Trial Period: | Screen | Baseline | | Treatment | | | | | | | Safety<br>Follow-up <sup>a</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Week: | -4 to -1 | 1 | 2 | 2 5 8 11 14 18 22 26 27 <sup>b</sup> | | | | | | 31 | | |
| Trial Day: | -31 to -1 | 1 | 14±3 | 14±3 35±3 56±3 77±3 98±3 126±3 154±3 182±3 189±3 | | | | | | 217±3 | | |
| Visit/Contact: | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 | Visit 10 | Visit 11<br>(EOT/ET) | Telephone <sup>c</sup> |

- j. Duplicate measurements of blood pressure and heart rate will be obtained in supine (after 5 minutes of rest) and 1 measurement of blood pressure and heart rate will be obtained on standing (2 minutes after rising from supine to standing).
- k. A triplicate set of ECGs is 3 consecutive ECGs collected 1 to 2 minutes apart over a 5-minute period.
- 1. The postdose ECGs (triplicate set for US sites at all visits and single for non-US sites at all visits) will be obtained at ~1 hour after administration of the first dose of IMP at the Baseline Visit just prior to the time of collection of the PK blood sample. ECGs at all postbaseline visits will be obtained just prior to the time of collection of the PK blood sample.
- m. All adverse events that are observed by trial personnel or volunteered by the subject in response to open-ended questioning will be recorded from the first dose of IMP through the end of the Safety Follow-up Period. Serious adverse events will be followed until resolution.
- n. Individual sites may require subjects to have COVID-19 testing done prior to randomization. COVID-19 testing may be performed after randomization per the principal investigator's discretion.
- o. Dipstick urinalysis results are not to be recorded on the eCRFs; any clinically significant abnormality should be captured as an adverse event.
- p. For women of childbearing potential only. All positive urine dipstick pregnancy tests must be confirmed by a serum test. Pregnancy tests can be performed at any time during the trial at the discretion of the investigator. Female subjects with exclusively the same sex partners may not be required to have pregnancy tests per investigator discretion; confirmation with the medical monitor is required.
- q. A urine drug screen is required at screening (see exclusion criteria for exclusions based on the urine drug screen) and may be obtained at other times, at investigator discretion, if use of prohibited drugs is suspected.
- r. PK samples will be collected ~1 hour after administration of the first dose (Day 1) and at the clinic visits at the end of Weeks 5, 11, 14, 22, and 27 just after ECG acquisition at each time point. The date and time of the most recent dose, the dose amount, and the time of the blood draw will be recorded.
- s. Future biospecimen research sample is optional and is to only be collected if signed consent is obtained from the subject.
- t. The first dose of IMP (at the Baseline Visit) will be taken in the clinic; all other doses will be taken on an outpatient basis. Subjects will be instructed to bring their IMP to each clinic visit. Compliance will be assessed through self-reporting by the subject and by tablet count.
- u. Prolactin results will be blinded.



| Trial Period: | Screen | Baseline | | Treatment | | | | | | | Safety<br>Follow-up <sup>a</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trial Week: | -4 to -1 | 1 | 2 | 5 | 8 | 11 | 14 | 18 | 22 | 26 | 27 <sup>b</sup> | 31 |
| Trial Day: | -31 to -1 | 1 | 14±3 | 35±3 | 56±3 | 77±3 | 98±3 | 126±3 | 154±3 | 182±3 | 189±3 | 217±3 |
| Visit/Contact: | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 | Visit 10 | Visit 11<br>(EOT/ET) | Telephone <sup>c</sup> |



# 9.2. EQ-5D-5L Dimensions

# EQ-5D-5L Dimensions (UK English Sample Version)

| Dimensions | Item | Coded Value |
|---|---|---|
| Mobility | I have no problems in walking about | 1 |
| | I have slight problems in walking about | 2 |
| | I have moderate problems in walking about | 3 |
| | I have severe problems in walking about | 4 |
| | I am unable to walk about | 5 |
| Self-care | I have no problems washing or dressing myself | 1 |
| | I have slight problems washing or dressing myself | 2 |
| | I have moderate problems washing or dressing myself | 3 |
| | I have severe problems washing or dressing myself | 4 |
| | I am unable to wash or dress myself | 5 |
| Usual activities | I have no problems doing my usual activities | 1 |
| (e.g., work, study, housework, family | I have slight problems doing my usual activities | 2 |
| or leisure activities) | I have moderate problems doing my usual activities | 3 |
| | I have severe problems doing my usual activities | 4 |
| | I am unable to do my usual activities | 5 |
| Pain/discomfort | I have no pain or discomfort | 1 |
| | I have slight pain or discomfort | 2 |
| | I have moderate pain or discomfort | 3 |
| | I have severe pain or discomfort | 4 |
| | I have extreme pain or discomfort | 5 |
| Anxiety/depression | I am not anxious or depressed | 1 |
| | I am slightly anxious or depressed | 2 |
| | I am moderately anxious or depressed | 3 |
| | I am severely anxious or depressed | 4 |
| | I am extremely anxious or depressed | 5 |

# 9.3. Columbia-Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation and Suicidal Behavior Scores

The C-SSRS is comprised of 10 categories with binary responses. The 10 categories include:

Category 1 – Wish to be Dead

Category 2 – Non-specific Active Suicidal Thoughts

Category 3 – Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act

Category 4 – Active Suicidal Ideation with Some Intent to Act, without Specific Plan

Category 5 – Active Suicidal Ideation with Specific Plan and Intent

Category 6 – Preparatory Acts or Behavior

Category 7 – Aborted Attempt

Category 8 – Interrupted Attempt

Category 9 – Actual Attempt (non-fatal)

Category 10 – Completed Suicide

Categories 1-5 represent Suicidal Ideation and categories 6-10 represent Suicidal Behavior. Each category is scored as 1 if there is a positive response in the category and a 0 if there are no positive responses in the category.

• Self-Injurious Behavior Without Suicidal Intent During Treatment

A subject will be categorized as having self-injurious behavior without suicidal intent if there is an occurrence of non-suicidal self-injurious behavior on the C-SSRS – Since Last Visit eCRF at any post-baseline visit.

• Baseline C-SSRS Score

Baseline represents the pre-treatment assessment of recent history, with elements of suicidal ideation assessed over the prior 6 months and elements of suicidal behavior assessed over the prior 2 years. It is scaled from 0 (no suicidal ideation or behavior) to 10 (completed suicide)

• Treatment-Emergent Suicide-Related Event

A subject will be categorized as having a treatment-emergent suicide-related event if at least one post-baseline suicidal ideation or suicidal behavior score is greater than 0.

• Treatment-Emergent Suicidal Ideation Compared to Recent History

A subject will be categorized as having treatment-emergent suicidal ideation compared to recent history when there is at least one post-baseline suicidal ideation score > 0 and is an increase from baseline. Lifetime scores are not considered for baseline suicidal ideation responses.

• Treatment-Emergent Serious Suicidal Ideation Compared to Recent History

A subject will be categorized as having treatment-emergent serious suicidal ideation compared to recent history if the baseline score was < 4 and the post-baseline suicidal ideation score increases to 4 or 5. Lifetime scores are not considered for baseline suicidal ideation responses.



• Emergence of Serious Suicidal Ideation Compared to Recent History

A subject will be categorized as having emergence of serious suicidal ideation compared to recent history if baseline score was 0 (no suicidal ideation) and post-baseline C-SSRS suicidal ideation score is either 4 or 5. Lifetime scores are not considered for baseline suicidal ideation responses.

• Emergence of Suicidal Behavior Compared to all Prior History

A subject will be categorized as having emergence of suicidal behavior compared to all prior history if there had been no suicidal behavior in Categories 6-10 reported at any pre-treatment assessment, including responses to lifetime history questions, and there is at least one positive post-baseline C-SSRS assessment in Categories 6-10. 'All Prior History' represents lifetime history.



# 9.4. Programming Conventions

- <u>Page orientation, margins, and fonts</u>: Summary tables, listings, and figures will appear in landscape orientation. There should be a 1.0" boundary on the left and right edges. The top and bottom margins are 1.0" for tables and listings, but may vary for figures. Output should be printed in Courier New with a point size of 8.
- <u>Identification of analysis population</u>: Every summary table, listing, and figure will clearly specify the analysis population being summarized/listed. Listings will be prepared for all subjects randomized.
- <u>Group headers:</u> In the summary tables, the group headers will identify the within-group sample size for the indicated analysis population. Of note, the header's sample size does not necessarily equal the number of subjects actually summarized within any given summary module; some subjects in the analysis population may have missing values and thus may not be summarized.
- <u>Suppression of percentages corresponding to null categories:</u> When count data are presented as category frequencies and corresponding percentages, the percent should be suppressed when the count is zero in order to draw attention to the non-zero counts.
- <u>Presentation of sample sizes:</u> Summary modules should indicate, in one way or another, the number of subjects actually contributing to the summary statistics presented in any given summary module. As mentioned above, this may be less than the number of subjects in the analysis population.
  - ♦ In the quantitative modules describing continuous variables (and thus presenting sample size, means, and standard deviations), the sample size should be the number of non-missing observations
  - ♦ For categorical variables that are presented in frequency tables, the module should present the total count in addition to the count in each category. Percentages should be calculated using this total as the denominator, and the percentage corresponding to the sum itself (that is, 100%) should be presented so as to indicate clearly to a reviewer the method of calculation.
- <u>Sorting:</u> Listings will be sorted by treatment, subject number and date, if applicable. If a listing is sorted in a different manner, it will be indicated on the listing shells.
- <u>General formatting rules:</u> Rounding for all variables will occur only as the last step, immediately prior to presentation in listings, tables, and figures. No intermediate rounding will be performed on derived variables. The standard rounding practice of rounding numbers ending in 0-4 down and numbers ending in 5-9 up will be employed.
- The presentation of numerical values will adhere to the following guidelines (exceptions may be necessary in some circumstances for derived analysis variables to allow readability):
  - Raw measurements will be reported to the number of significant digits as captured electronically or on the eCRFs.





- Standard deviations will be reported to two decimal places beyond the number of decimal places the original parameter is presented. EQ-5D-5L Index Score summaries will use 4 decimal places for standard deviation.
- Means medians, and quartiles will be reported to one decimal place beyond the number of decimal places the original parameter is presented.
- will be reported to the one decimal place beyond the number of decimal places the original parameter is presented.
- Calculated percentages will be reported with one decimal place.
- Coefficient of variation will be reported to the same number of decimal places as the standard deviation.
- ♦ P-values will be reported to 4 decimal places
- Dates will be formatted as DDMMMYYYY. Partial dates will be presented on data listings as recorded on eCRFs.
- Time will be presented according to the 24-hour clock (HH:MM).
- <u>Verification of Results</u>: All analyses will be subject to formal verification procedures. Specifically, results will be verified utilizing independent programming prior to issuance of the draft statistical report. All documents will be verified by the lead statistician to ensure accuracy and consistency of analyses.



# 9.5. MNAR Cases Identified Prior to Database Lock

| Site | Subject<br>ID | IMP Start<br>Date | IMP End Date | Intercurrent Event | Prohibited PD<br>Medication<br>Start Date |
|---|---|---|---|---|---|
| | | | | PHYSICIAN DECISION | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | ADVERSE EVENT | • |
| | | | | ADVERSE EVENT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | ADVERSE EVENT | |
| | | | | WITHDRAWAL BY SUBJECT | • |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | • |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | ADVERSE EVENT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | PROHIBITED MEDICATION | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | LACK OF EFFICACY | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | LACK OF EFFICACY | |
| | | | | LACK OF EFFICACY | |



| Site | Subject<br>ID | IMP Start<br>Date | IMP End Date | Intercurrent Event | Prohibited PD<br>Medication<br>Start Date |
|---|---|---|---|---|---|
| | | | | WITHDRAWAL BY SUBJECT | • |
| | | | | WITHDRAWAL BY SUBJECT | • |
| | | | | ADVERSE EVENT | • |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | • |
| | | | | WITHDRAWAL BY SUBJECT | • |
| | | | | WITHDRAWAL BY SUBJECT | • |
| | | | | LACK OF EFFICACY | • |
| | | | | ADVERSE EVENT | • |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | • |
| | | | | WITHDRAWAL BY SUBJECT | • |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | WITHDRAWAL BY SUBJECT | |
| | | | | ADVERSE EVENT | |
| | | | | LACK OF EFFICACY | |



# 9.6. Core Codes for imputation of MAR and MNAR

# 9.6.1. Imputation of Missing at Random (MAR) Cases

SAS PROC MI will be used to generate 27 possible imputed datasets using the following SAS code:

```
proc mi data=mcmc1 seed=SEED1 nimpute=27 out=Out1X; mcmc chain=multiple displayinit initial=em(itprint); var TRT y0 y1 y2 ... yn; run;
```

Here, TRT is an indicator variable representing treatment with values of 'CVL-751 5 mg', CVL-751 15 mg', or 'Placebo',  $Y_1$  -  $Y_N$  represent the response variable (e.g., MDS-UPDRS Part II+III score) for each visit,  $Y_0$  is the baseline score, and SEED1 is a random number.

Each of these datasets will be analyzed using PROC MIXED in SAS using the MMRM model. The results of the analyses of the datasets will be combined using PROC MIANALYZE to produce an inferential result.

#### 9.6.2. Imputation of Missing Not at Random (MNAR) Cases

The MNAR cases are imputed using reference based imputation (J2R) method. The five macros; SAS code for reference based multiple imputation [https://www.lshtm.ac.uk/research/centresprojects-groups/missing-data#dia-working-group] will be used to generate 27 possible imputed datasets using the following sample SAS code:

```
%include "&Path\part1A_33.sas";
%include "&Path\part1B_47.sas";
%include "&Path\part2A 40.sas";
%include "&Path\part2B_31.sas";
%include "&Path\part3_55.sas";
%include "&Path\plotter_7.sas";
%include "&Path\plotter_7.sas";
%part1A(Jobname=X, Data=XX, Subject=usubjid, Response=aval, Time=avisitn, Treat=Tr t01pn, cov=BASE, Catcov=MAOBINHI, covgroup=trt01pn, Debug=1);
%part1b(Jobname=X, Ndraws=27, thin=350, seed=s, Debug=1);
%part2a(Jobname=X J2R, inname=XX, method=J2R, ref=0, Debug=1);
%part2b(Jobname=X J2R, seed=s, Debug=1);
```

Each of these datasets will be analyzed using PROC MIXED in SAS using the MMRM model. The results of the analyses of the datasets will be combined using PROC MIANALYZE to produce an inferential result.



# 9.7. Randomization Stratum Errors

| Site | Subject | Confirmed Status of MAO-<br>B Inhibitor Use | IRT Randomization Stratum of MAO-B Inhibitor Use |
|---|---|---|---|
| | | No | Yes |
| | | No | Yes |
| | | No | Yes |
| | | Yes | No |



# 9.8. CTCAE Based Laboratory Test Results Grading Specifications

#### Lab Test = Albumin

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Hypoalbuminemia | <lln -="" 3="" dl;<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL; &lt;30 - 20 g/L</td><td>&lt;2 g/dL; &lt;20 g/L</td><td>Life-threatening<br/>consequences; urgent<br/>intervention<br/>indicated</td><td>Death</td></lln></lln> | <3 - 2 g/dL; <30 - 20 g/L | <2 g/dL; <20 g/L | Life-threatening<br>consequences; urgent<br>intervention<br>indicated | Death |

Albumin will have grades 1-3,

- Grade 1 being any values from the LLN to 3 g/dL,
- Grade 2 from 2 to < 3 g/dL and
- Grade 3 < 2 g/dL

#### Lab Test = Amylase

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Serum amylase<br>increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN; >2.0 - 5.0<br>x ULN and asymptomatic | >2.0 - 5.0 x ULN with signs<br>or symptoms; >5.0 x ULN<br>and asymptomatic | >5.0 x ULN and with signs or symptoms | - |

Amylase will have Grades 1, 2 and 3:

- Grade 1 being any values from the ULN to 1.5 x ULN
- Grade 2 from >1.5 to 5.0 x ULN
- Grade 3 from>5 x ULN

Lab Test = Alkaline Phosphatase

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Alkaline<br>phosphatase<br>increased | baseline was normal; | >2.5 - 5.0 x ULN if baseline<br>was normal; >2.5 - 5.0 x<br>baseline if baseline was<br>abnormal | >5.0 - 20.0 x ULN if baseline<br>was normal; >5.0 - 20.0 x<br>baseline if baseline was<br>abnormal | >20.0 x ULN if<br>baseline was normal;<br>>20.0 x baseline if<br>baseline was<br>abnormal | - |

Alkaline Phosphatase will have grades 1-4 and grading is based ULN only.

- Grade 1 being any values from the ULN to 2.5 x ULN
- Grade 2 from >2.5 to 5.0 x ULN
- Grade 3 from >5.0 to 20.0 x ULN
- Grade 4 from>20.0 x ULN

#### Lab Test = Alanine Aminotransferase

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Alanine<br>aminotransferase<br>increased | baseline was normal; | >3.0 - 5.0 x ULN if baseline<br>was normal; >3.0 - 5.0 x<br>baseline if baseline was<br>abnormal | >5.0 - 20.0 x ULN if baseline<br>was normal; >5.0 - 20.0 x<br>baseline if baseline was<br>abnormal | >20.0 x ULN if<br>baseline was normal;<br>>20.0 x baseline if<br>baseline was<br>abnormal | - |

ALT will have grades 1-4 and grading is based ULN only.

- Grade 1 being any values from the ULN to 3.0 x ULN
- Grade 2 from >3.0 to 5.0 x ULN
- Grade 3 from >5.0 to 20.0 x ULN
- Grade 4 from>20.0 x ULN



Lab Test = Aspartate Aminotransferase

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Aspartate<br>aminotransferase<br>increased | baseline was normal; | >3.0 - 5.0 x ULN if baseline<br>was normal; >3.0 - 5.0 x<br>baseline if baseline was<br>abnormal | >5.0 - 20.0 x ULN if baseline<br>was normal; >5.0 - 20.0 x<br>baseline if baseline was<br>abnormal | >20.0 x ULN if<br>baseline was normal;<br>>20.0 x baseline if<br>baseline was<br>abnormal | - |

AST will have grades 1-4 and grading is based ULN only.

- Grade 1 being any values from the ULN to 3.0 x ULN
- Grade 2 from >3.0 to 5.0 x ULN
- Grade 3 from >5.0 to 20.0 x ULN
- Grade 4 from>20.0 x ULN



#### Lab Test = Bilirubin

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Blood bilirubin increased | baseline was normal; | , | >3.0 - 10.0 x ULN if baseline<br>was normal; >3.0 - 10.0 x<br>baseline if baseline was<br>abnormal | >10.0 x ULN if<br>baseline was normal;<br>>10.0 x baseline if<br>baseline was<br>abnormal | - |

Bilirubin will have grades 1-4 and grading is based ULN only

- Grade 1 being any values from the ULN to 1.5 x ULN
- Grade 2 from >1.5 to 3.0 x ULN
- Grade 3 from >3.0 to 10.0 x ULN
- Grade 4 from>10.0 x ULN



Lab Test = Corrected Serum Calcium

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Hypocalcemia | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" ionized="" l;="" l<="" mg="" mmol="" td=""><td>Corrected serum calcium of<br/>&lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75<br/>mmol/L; Ionized calcium<br/>&lt;1.0 - 0.9 mmol/L;<br/>symptomatic</td><td>Corrected serum calcium of &lt;7.0 - 6.0 mg/dL; &lt;1.75 - 1.5 mmol/L; Ionized calcium &lt;0.9 - 0.8 mmol/L; hospitalization indicated</td><td>Corrected serum calcium<br/>of &lt;6.0 mg/dL; &lt;1.5<br/>mmol/L; Ionized<br/>calcium &lt;0.8 mmol/L;<br/>life-threatening<br/>consequences</td><td>Death</td></lln> | Corrected serum calcium of<br><8.0 - 7.0 mg/dL; <2.0 - 1.75<br>mmol/L; Ionized calcium<br><1.0 - 0.9 mmol/L;<br>symptomatic | Corrected serum calcium of <7.0 - 6.0 mg/dL; <1.75 - 1.5 mmol/L; Ionized calcium <0.9 - 0.8 mmol/L; hospitalization indicated | Corrected serum calcium<br>of <6.0 mg/dL; <1.5<br>mmol/L; Ionized<br>calcium <0.8 mmol/L;<br>life-threatening<br>consequences | Death |
| Hypercalcemia | Corrected serum<br>calcium of >ULN -<br>11.5 mg/dL; >ULN -<br>2.9 mmol/L; Ionized<br>calcium >ULN - 1.5<br>mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; Ionized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 - 13.5 mg/dL; >3.1 - 3.4 mmol/L; Ionized calcium >1.6 - 1.8 mmol/L; hospitalization indicated | Corrected serum calcium<br>of >13.5 mg/dL; >3.4<br>mmol/L; Ionized<br>calcium >1.8 mmol/L;<br>life-threatening<br>consequences | Death |

Calcium will have to be corrected for albumin using Payne's formula:

Corrected calcium = measured Ca (mg/dL) +  $0.8 \times (4.0 \text{ g/dL} - \text{patient albumin (g/dL)})$ .

(NOTE: It should be confirmed with the lab whether or not the correction has already been applied).

The grading is in both directions High and Low. Both directions are graded in 4 categories as Hypercalcemia

- Grade 1 being any values from the ULN to 11.5 mg/dL,
- Grade 2 from >11.5 to 12.5 mg/dL,
- Grade 3 from >12.5 to 13.5 mg/dL,
- Grade 4 >13.5 mg/dL

#### Hypocalcemia

- Grade 1 being any values from the LLN to 8.0 mg/dL,
- Grade 2 from 7.0 to <8.0 mg/dL,</li>
- Grade 3 from 6.0 to <7.0 mg/dL,
- Grade 4 < 6.0 mg/dL



#### Lab Test = Cholesterol

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Cholesterol high | >ULN - 300 mg/dL;<br>>ULN - 7.75<br>mmol/L | >300 - 400 mg/dL; >7.75 -<br>10.34 mmol/L | >400 - 500 mg/dL; >10.34 -<br>12.92 mmol/L | >500 mg/dL; >12.92<br>mmol/L | - |

Cholesterol will have grades 1-4,

- Grade 1 being any values from the ULN to 300 mg/dL,
- Grade 2 from >300 to 400 mg/dL,
- Grade 3 from >400 to 500 mg/dL,
- Grade 4 > 500 mg/dL

#### Lab Test = Creatine Kinase

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| CPK increased | >ULN - 2.5 x ULN | >2.5 x ULN - 5 x ULN | >5 x ULN - 10 x ULN | >10 x ULN | - |

Creatine Kinase will have grades 1-4,

- $\bullet$   $\;$  Grade 1 being any values from the ULN to 2.5 x ULN ,
- Grade 2 from >2.5 to 5 x ULN,
- Grade 3 from >5 to 10 x ULN ,
- Grade 4 > 10 ULN



#### Lab Test = Creatinine

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Creatinine increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x baseline; >1.5 - 3.0 x ULN | >3.0 x baseline; >3.0 - 6.0 x<br>ULN | >6.0 x ULN | - |

# Creatinine will have grades 1-4

- Grade 1 being any values from the ULN to 1.5 x ULN,
- Grade 2 from >1.5 to 3.0 x ULN or >1.5 3.0 x baseline,
- Grade 3 from >3.0 to 6.0 x ULN or >3.0 x baseline,
- Grade 4 > 6.0 x ULN


Lab Test = Fibrinogen

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Fibrinogen<br>decreased | <1.0 - 0.75 x LLN; if<br>abnormal, <25%<br>decrease from<br>baseline | <0.75 - 0.5 x LLN; if<br>abnormal, 25 - <50%<br>decrease from baseline | <0.5 - 0.25 x LLN; if<br>abnormal, 50 - <75%<br>decrease from baseline | <0.25 x LLN; if<br>abnormal, 75%<br>decrease from<br>baseline; absolute<br>value <50 mg/dL | - |

Fibrinogen will have Grades 1-4:

- Grade 1 < 1.0 0.75 x LLN
- Grade 2 < 0.75 0.5 x LLN</li>
- Grade 3 < 0.5 0.25 x LLN</li>
- Grade 4 < 0.25 x LLN</li>

Lab Test = Gamma-Glutamyl Transpeptidase

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| GGT increased | baseline was normal; | >2.5 - 5.0 x ULN if baseline<br>was normal; >2.5 - 5.0 x<br>baseline if baseline was<br>abnormal | >5.0 - 20.0 x ULN if baseline<br>was normal; >5.0 - 20.0 x<br>baseline if baseline was<br>abnormal | >20.0 x ULN if<br>baseline was normal;<br>>20.0 x baseline if<br>baseline was<br>abnormal | - |

Gamma-Glutamyl Transpeptidase will have grades 1-4 and based on ULN only

- Grade 1 being any values from the ULN to 2.5 x ULN,
- Grade 2 from >2.5 to 5.0 x ULN
- Grade 3 from >5.0 to 20.0 x ULN
- Grade 4 from>20.0 x ULN

### Lab Test = Glucose

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Hyperglycemia | Abnormal glucose<br>above baseline with<br>no medical<br>intervention | Change in daily management<br>from baseline for a diabetic;<br>oral antiglycemic agent<br>initiated; workup for diabetes | Insulin therapy initiated;<br>hospitalization indicated | Life-threatening<br>consequences; urgent<br>intervention<br>indicated | Death |
| Hypoglycemia | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 - 40 mg/dL; &lt;3.0 - 2.2<br/>mmol/L</td><td>&lt;40 - 30 mg/dL; &lt;2.2 - 1.7 mmol/L</td><td>&lt;30 mg/dL; &lt;1.7<br/>mmol/L; life-<br/>threatening<br/>consequences;<br/>seizures</td><td>Death</td></lln></lln> | <55 - 40 mg/dL; <3.0 - 2.2<br>mmol/L | <40 - 30 mg/dL; <2.2 - 1.7 mmol/L | <30 mg/dL; <1.7<br>mmol/L; life-<br>threatening<br>consequences;<br>seizures | Death |

Hypoglycemia will have grades 1-4,

- Grade 1 being any values from the LLN to 55 mg/dL,
- Grade 2 from 40 to <55 mg/dL,
- Grade 3 from 30 to <40 mg/dL,</li>
- Grade 4 < 30 mg/dL

Hyperglycemia will have one grade using the WHO criterion below

• Grade 1 >200 mg/dL;



Lab Test = Lipase

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Serum lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN; >2.0 - 5.0<br>x ULN and asymptomatic | >2.0 - 5.0 x ULN with signs<br>or symptoms; >5.0 x ULN<br>and asymptomatic | >5.0 x ULN and with signs or symptoms | - |

Lipase will have Grades 1, 2 and 3:

- Grade 1 being any values from the ULN to 1.5 x ULN
- Grade 2 from >1.5 to 5.0 x ULN
- Grade 3 from>5 x ULN

Lab Test = Magnesium

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23<br>mmol/L | • | >3.0 - 8.0 mg/dL; >1.23 - 3.30 mmol/L | >8.0 mg/dL; >3.30<br>mmol/L; life-<br>threatening<br>consequences | Death |
| Hypomagnesemia | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL; &lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 - 0.7 mg/dL; &lt;0.4 - 0.3 mmol/L</td><td>&lt;0.7 mg/dL; &lt;0.3<br/>mmol/L; life-<br/>threatening<br/>consequences</td><td>Death</td></lln></lln> | <1.2 - 0.9 mg/dL; <0.5 - 0.4 mmol/L | <0.9 - 0.7 mg/dL; <0.4 - 0.3 mmol/L | <0.7 mg/dL; <0.3<br>mmol/L; life-<br>threatening<br>consequences | Death |

Hypermagnesemia will have grades 1, 3, and 4,

- Grade 1 being any values from the ULN to 3.0 mg/dL,
- Grade 3 from >3.0 to 8.0 mg/dL,
- Grade 4 from>8.0 mg/dL

Hypomagnesemia will have grades 1 - 4,

- Grade 1 being any values from the LLN to 1.2 mg/dL,
- Grade 2 from 0.9 to <1.2 mg/dL,
- Grade 3 from 0.7 to <0.9 mg/dL,
- Grade 4 < 0.7 mg/dL</li>

### Lab Test = Potassium

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L;<br>intervention initiated | >6.0 - 7.0 mmol/L;<br>hospitalization indicated | >7.0 mmol/L; life-<br>threatening<br>consequences | Death |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td>Symptomatic with <lln -<br="">3.0 mmol/L; intervention<br/>indicated</lln></td><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-<br/>threatening<br/>consequences</td><td>Death</td></lln> | Symptomatic with <lln -<br="">3.0 mmol/L; intervention<br/>indicated</lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated | <2.5 mmol/L; life-<br>threatening<br>consequences | Death |

Hyperkalemia will have grades 1-4,

- Grade 1 being any values from the ULN to 5.5 mmol/L,
- Grade 2 from >5.5 to 6.0 mmol/L,
- Grade 3 from >6.0 to 7.0 mmol/L,
- Grade 4 from>7.0 mmol/L

Hypokalemia will have grades 1, 3, and 4,

- Grade 1 being any values from the LLN to 3.0 mmol/L,
- Grade 3 from >2.5 to 3.0 mmol/L,
- Grade 4 <2.5 mmol/L</li>

### Lab Test = Sodium

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L;<br>intervention initiated | >155 - 160 mmol/L;<br>hospitalization indicated | >160 mmol/L; life-<br>threatening<br>consequences | Death |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>125-129 mmol/L and asymptomatic</td><td>125-129 mmol/L<br/>symptomatic; 120-124<br/>mmol/L regardless of<br/>symptoms</td><td>&lt;120 mmol/L; life-<br/>threatening<br/>consequences</td><td>Death</td></lln> | 125-129 mmol/L and asymptomatic | 125-129 mmol/L<br>symptomatic; 120-124<br>mmol/L regardless of<br>symptoms | <120 mmol/L; life-<br>threatening<br>consequences | Death |

Hypernatremia will have grades 1-4,

- Grade 1 being any values from the ULN to 150 mmol/L,
- Grade 2 from >150 to 155 mmol/L,
- Grade 3 from >155 to 160 mmol/L,
- Grade 4 from>160 mmol/L

Hyponatremia will have grades 1-4,

- Grade 1 being any values from the LLN to 130 mmol/L,
- Grade 2 from 125 to <130 mmol/L,
- Grade 3 from 120 to <125 mmol/L,
- Grade 4 <120 mmol/L</li>



Lab Test = Triglycerides

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Hypertriglyceridemia | 150 mg/dL - 300<br>mg/dL; 1.71<br>mmol/L - 3.42<br>mmol/L | >300 mg/dL - 500 mg/dL;<br>>3.42 mmol/L - 5.7 mmol/L | >500 mg/dL - 1000 mg/dL;<br>>5.7 mmol/L - 11.4 mmol/L | >1000 mg/dL; >11.4<br>mmol/L; life-<br>threatening<br>consequences | Death |

Triglycerides will have grades 1-4,

- Grade 1 being any values from the 150 to 300 mg/dL,
- Grade 2 from >300 to 500 mg/dL,
- Grade 3 from >500 to 1000 mg/dL,
- Grade 4 from>1000 mmol/L

# Lab Test = Uric Acid

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Hyperuricemia | >ULN without physiologic consequences | - | >ULN with physiologic consequences | Life-threatening consequences | Death |

Uric Acid will not be CTCAE graded.

Lab Test = Bicarbonate or CO2

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Blood bicarbonate decreased | <lln and="" initiated<="" intervention="" no="" td=""><td>•</td><td>•</td><td>-</td><td>-</td></lln> | • | • | - | - |

Bicarbonate or CO2 will not be CTCAE graded.

Lab Test = Phosphorus or Phosphate

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Hypophosphatemia | Laboratory finding<br>only and<br>intervention not<br>indicated | Oral replacement therapy indicated | Severe or medically<br>significant but not<br>immediately life-threatening;<br>hospitalization or<br>prolongation of existing<br>hospitalization indicated | Life-threatening consequences | Death |
| Hyperphosphatemia | Laboratory finding<br>only and<br>intervention not<br>indicated | Noninvasive intervention indicated | Severe or medically<br>significant but not<br>immediately life-threatening;<br>hospitalization or<br>prolongation of existing<br>hospitalization indicated | Life-threatening<br>consequences;<br>urgent intervention<br>indicated (e.g.,<br>dialysis) | Death |

Phosphorus or Phosphate will not be CTCAE graded.



Lab Test = Serum pH [This is not urine pH]

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Acidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 | Life-threatening consequences | - |
| Alkalosis | pH >normal, but<br><=7.5 | - | pH >7.5 | Life-threatening consequences | - |

Serum pH will be graded in both directions with Grades 1 and 3 only.

Acidosis Grade 1 .<LLN, but >=7.3 Grade 3, pH < 7.3

Alkaosis Grade 1 .>ULN, but <=7.5 Grade 3, pH < 7.5



Lab Test = Activated Partial Thromboplastin Time

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Activated partial thromboplastin time prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; bleeding | • | - |

APTT will be graded in Grade 1-3

- Grade 1 being any values from the >ULN to 1.5 x ULN,
- Grade 2 from >1.5 to 2.5 x ULN,
- Grade 3 from >2.5 x ULN,

#### Lab Test = International Normalized Ratio

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| INR increased | >1.2 - 1.5; >1 - 1.5 x<br>baseline if on<br>anticoagulation;<br>monitoring only<br>indicated | >1.5 - 2.5; >1.5 - 2.5 x<br>baseline if on<br>anticoagulation; dose<br>adjustment indicated | >2.5; >2.5 x baseline if on anticoagulation; bleeding | - | - |

INR will be graded in Grade 1-3 without baseline factor

- Grade 1 being any values from the >1.2 to 1.5,
- Grade 2 from >1.5 to 2.5,
- Grade 3 from >2.5,



Lab Test = Eosinophils

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Eosinophilia | >ULN and >Baseline | - | Steroids initiated | - | - |

Eosinophils will not be CTCAE graded

Lab Test = Hemoglobin

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Anemia | Hemoglobin (Hgb)<br><lln -="" 10.0="" dl;<br="" g=""><lln -="" 6.2="" l;<br="" mmol=""><lln -="" 100="" g="" l<="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL; &lt;6.2 - 4.9 mmol/L; &lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL; &lt;4.9 mmol/L; &lt;80 g/L; transfusion indicated</td><td>Life-threatening<br/>consequences; urgent<br/>intervention<br/>indicated</td><td>Death</td></lln></lln></lln> | Hgb <10.0 - 8.0 g/dL; <6.2 - 4.9 mmol/L; <100 - 80g/L | Hgb <8.0 g/dL; <4.9 mmol/L; <80 g/L; transfusion indicated | Life-threatening<br>consequences; urgent<br>intervention<br>indicated | Death |
| Hemoglobin<br>Increased | Increase in > 0-2 | Increase in >2-4g/dL | Increase > 4 g/DL | • | Death |

Decreased Hemoglobin will have grades 1-3, with

- Grade 1 being any values from the LLN to 10 g/DL,
- Grade 2 from 8 to < 10 g/DL and
- Grade 3 < 8 g/DL

Increased Hemoglobin will not be graded.



Lab Test = CD4 Lymphocytes

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| CD4 lymphocytes<br>decreased | <lln -="" 500="" mm3;<br=""><lln -="" 0.5="" 10e9<br="" x="">/L</lln></lln> | <500 - 200/mm3; <0.5 - 0.2<br>x 10e9 /L | <200 - 50/mm3; <0.2 x 0.05 - 10e9 /L | <50/mm3; <0.05 x<br>10e9 /L | - |

Decreased CD4 count will have grades 1-4, with

- Grade 1 being any values from the LLN to 500/mm3,
- Grade 2 from <500 to 200/mm3 and</li>
- Grade 3 from <200 to 50/mm3 and
- Grade 4 < 50/mm3



Lab Test = Lymphocytes

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Lymphocyte count decreased | <lln -="" 800="" mm3;<br=""><lln -="" 0.8="" 10e9="" l<="" td="" x=""><td>&lt;800 - 500/mm3; &lt;0.8 - 0.5<br/>x 10e9 /L</td><td>&lt;500 - 200/mm3; &lt;0.5 - 0.2 x<br/>10e9 /L</td><td>&lt;200/mm3; &lt;0.2 x<br/>10e9 /L</td><td>Lymphocyte count decreased</td></lln></lln> | <800 - 500/mm3; <0.8 - 0.5<br>x 10e9 /L | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200/mm3; <0.2 x<br>10e9 /L | Lymphocyte count decreased |
| Lymphocyte count increased | - | >4000/mm3 - 20,000/mm3 | >20,000/mm3 | - | Lymphocyte count increased |

Decreased Lymphocytes will have grades 1-4, with

- Grade 1 being any values from the LLN to 800/mm3,
- Grade 2 from <800 to 500/mm3 and</li>
- Grade 3 from <500 to 200/mm3 and
- Grade 4 < 200/mm3

Increase Lymphocytes will have grades 2 and 3 only, with

- Grade 2 from >4000 to 20,000/mm3 and
- Grade 3 >20,000/mm3

Lab Test = Neutrophils

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Neutrophil count decreased | <lln -="" 1500="" mm3;<br=""><lln -="" 1.5="" 10e9<br="" x="">/L</lln></lln> | <1500 - 1000/mm3; <1.5 -<br>1.0 x 10e9 /L | <1000 - 500/mm3; <1.0 - 0.5<br>x 10e9 /L | <500/mm3; <0.5 x<br>10e9 /L | - |

Neutrophils will have grades 1-4, with

- Grade 1 being any values from the LLN to 1500/mm3,
- Grade 2 from 1000 to <1500/mm3 and</li>
- Grade 3 from 500 to <1000/mm3 and
- Grade 4 < 500/mm3

# Lab Test = Platelets

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Platelet count<br>decreased | <lln -<br="">75,000/mm3; <lln<br>- 75.0 x 10e9 /L</lln<br></lln> | <75,000 - 50,000/mm3;<br><75.0 - 50.0 x 10e9 /L | <50,000 - 25,000/mm3; <50.0<br>- 25.0 x 10e9 /L | <25,000/mm3; <25.0<br>x 10e9 /L | - |

Platelet count will not be CTCAE graded



### Lab Test = WBC

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| White blood cell<br>decreased | <lln -="" 3000="" mm3;<br=""><lln -="" 10e9<br="" 3.0="" x="">/L</lln></lln> | <3000 - 2000/mm3; <3.0 -<br>2.0 x 10e9 /L | <2000 - 1000/mm3; <2.0 -<br>1.0 x 10e9 /L | <1000/mm3; <1.0 x<br>10e9 /L | - |
| Leukocytosis | - | - | >100,000/mm3 | Clinical<br>manifestations of<br>leucostasis; urgent<br>intervention<br>indicated | Death |

Decreased WBC will have grades 1-4, with

- Grade 1 being any values from the LLN to 3000/mm3,
- Grade 2 from 2000 to <3,000/mm3 and
- Grade 3 from 1000 to <2,000/mm3 and
- Grade 4 < 1000/mm3

High WBC will have grade 1, with

• Grade 1 >11,000/mm3 (https://www.aafp.org/afp/2000/1101/p2053 html),



# Lab Test = Urine Glucose

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|------------|---------|---------|---------|---------|---------|
| Glucosuria | Present | - | - | - | - |

Urine Glucose will have grades 1,

• Grade 1 if not negative or trace

# Lab Test = Urine Protein

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Proteinuria | 1+ proteinuria;<br>urinary protein<br>≥ULN - <1.0 g/24<br>hrs | Adult: 2+ and 3+ proteinuria; urinary protein 1.0 - <3.5 g/24 hrs; Pediatric: Urine P/C (Protein/Creatinine) ratio 0.5 - 1.9 | Adult: Urinary protein >=3.5 g/24 hrs; 4+ proteinuria; Pediatric: Urine P/C (Protein/Creatinine) ratio >1.9 | - | - |

Urine Protein will have grades 1-3, with

- Grade 1 = 1+,
- Grade 2 = 2 + to 3 +
- Grade 3 = 4+



Lab Test: Urine RBCs/Blood

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| Hematuria | Asymptomatic;<br>clinical or<br>diagnostic<br>observations only;<br>intervention not<br>indicated | Symptomatic; urinary<br>catheter or bladder<br>irrigation indicated;<br>limiting instrumental<br>ADL | Gross hematuria;<br>transfusion, IV<br>medications, or<br>hospitalization<br>indicated; elective<br>invasive intervention<br>indicated; limiting self<br>care ADL | Life-threatening<br>consequences;<br>urgent invasive<br>intervention<br>indicated | Death |

Urine blood will not be CTCAE graded

### Lab Test: eGFR or CrCl

| CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|---|---|---|---|---|---|
| eGFR<br>decreased/CrCL<br>decreased | eGFR (estimated<br>Glomerular Filtration<br>Rate) or CrCl<br>(creatinine clearance)<br><lln -="" 60<br="">ml/min/1.73 m2 or<br/>proteinuria 2+ present;<br/>urine protein/creatinine<br/>&gt;0.5</lln> | eGFR or CrCl 59 - 30<br>ml/min/1.73 m2 | eGFR or CrCl 29 - 15<br>ml/min/1.73 m2 | eGFR or CrCl <15<br>ml/min/1.73 m2;<br>dialysis or renal<br>transplant indicated | Death |

Values will be graded using the CTCAE values noted above with Grade 1 – Grade 4 values.

eGFR/CrCL:

Grade 1:  $\leq$  LLN - 60 ml/min/1.73 m2

Grade 2: 30 - < 60 ml/min/1.73 m2

Grade 3: 15 - < 30 ml/min/1.73 m2

Grade 4: < 15 ml/min/1.73



# 9.9. EQ-5D-5L Index Cross-walk Mapping

US Value Set

| Health State (5L profile) | US |
|---------------------------|-------|
| 11111 | 1.000 |
| 11112 | 0.876 |
| 11113 | 0.844 |
| 11114 | 0.700 |
| 11115 | 0.550 |
| 11121 | 0.861 |
| 11122 | 0.820 |
| 11123 | 0.809 |
| 11124 | 0.669 |
| 11125 | 0.524 |
| 11131 | 0.827 |
| 11132 | 0.806 |
| 11133 | 0.800 |
| 11134 | 0.661 |
| 11135 | 0.517 |
| 11141 | 0.682 |
| 11142 | 0.663 |
| 11143 | 0.659 |
| 11144 | 0.544 |
| 11145 | 0.426 |
| 11151 | 0.463 |
| 11152 | 0.450 |
| 11153 | 0.446 |
| 11154 | 0.369 |
| 11155 | 0.289 |
| 11211 | 0.888 |
| 11212 | 0.846 |
| 11213 | 0.835 |
| 11214 | 0.695 |
| 11215 | 0.550 |
| 11221 | 0.832 |
| 11222 | 0.796 |
| 11223 | 0.786 |
| 11224 | 0.654 |
| 11225 | 0.517 |
| 11231 | 0.818 |
| 11232 | 0.783 |
| 11233 | 0.774 |
| 11234 | 0.644 |
| 11235 | 0.508 |
| 11241 | 0.676 |
| 11242 | 0.647 |
| 11243 | 0.640 |
| 11244 | 0.532 |
| 11245 | 0.421 |
| 11251 | 0.463 |
| 11201 | 0.103 |



| Health State (5L profile) | US |
|---------------------------|----------------|
| 11252 | 0.443 |
| 11253 | 0.437 |
| 11254 | 0.365 |
| 11255 | 0.289 |
| 11311 | 0.860 |
| 11312 | 0.839 |
| 11313 | 0.833 |
| 11314 | 0.694 |
| 11315 | 0.550 |
| 11321 | 0.825 |
| 11322 | 0.790 |
| 11323 | 0.781 |
| 11324 | 0.650 |
| 11325 | 0.515 |
| 11331 | 0.816 |
| 11332 | 0.778 |
| 11333 | 0.768 |
| 11334 | 0.639 |
| 11335 | 0.506 |
| 11341 | 0.675 |
| 11342 | 0.643 |
| 11343 | 0.635 |
| 11343 | 0.529 |
| 11345 | 0.329 |
| 11343 | 0.463 |
| 11351 | 0.441 |
| 11352 | 0.435 |
| 11353 | 0.363 |
| 11354 | 0.303 |
| 11411 | 0.783 |
| 11411 | 0.763 |
| 11412 | 0.764 |
| 11413 | |
| 11414 | 0.641<br>0.518 |
| 11415 | |
| | 0.751 |
| 11422 | 0.721 |
| 11423 | 0.713 |
| 11424 | 0.601 |
| 11425 | 0.485 |
| 11431 | 0.742 |
| 11432 | 0.710 |
| 11433 | 0.701 |
| 11434 | 0.591 |
| 11435 | 0.477 |
| 11441 | 0.618 |
| 11442 | 0.591 |
| 11443 | 0.584 |
| 11444 | 0.490 |
| 11445 | 0.393 |
| 11451 | 0.431 |
| 11452 | 0.412 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 11453 | 0.406 |
| 11454 | 0.338 |
| 11455 | 0.266 |
| 11511 | 0.626 |
| 11512 | 0.613 |
| 11513 | 0.609 |
| 11514 | 0.532 |
| 11515 | 0.452 |
| 11521 | 0.599 |
| 11522 | 0.579 |
| 11523 | 0.574 |
| 11524 | 0.501 |
| 11525 | 0.425 |
| 11531 | 0.592 |
| 11532 | 0.571 |
| 11533 | 0.565 |
| 11534 | 0.493 |
| 11535 | 0.418 |
| | 0.501 |
| 11541 | |
| 11542 | 0.483 |
| 11543 | 0.478 |
| 11544 | 0.410 |
| 11545 | 0.339 |
| 11551 | 0.365 |
| 11552 | 0.352 |
| 11553 | 0.348 |
| 11554 | 0.285 |
| 11555 | 0.220 |
| 12111 | 0.854 |
| 12112 | 0.815 |
| 12113 | 0.805 |
| 12114 | 0.665 |
| 12115 | 0.520 |
| 12121 | 0.802 |
| 12122 | 0.765 |
| 12123 | 0.756 |
| 12124 | 0.623 |
| 12125 | 0.486 |
| 12131 | 0.789 |
| 12132 | 0.753 |
| 12133 | 0.743 |
| 12134 | 0.613 |
| 12134 | 0.478 |
| 12133 | 0.478 |
| 12141 | 0.617 |
| 12142 | 0.607 |
| 12144 | 0.502 |
| 12145 | 0.390 |
| 12151 | 0.433 |
| 12152 | 0.413 |
| 12153 | 0.408 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 12154 | 0.335 |
| 12155 | 0.259 |
| 12211 | 0.828 |
| 12212 | 0.792 |
| 12213 | 0.782 |
| 12214 | 0.650 |
| 12215 | 0.513 |
| 12221 | 0.778 |
| 12222 | 0.731 |
| 12223 | 0.719 |
| 12224 | 0.595 |
| 12225 | 0.467 |
| 12231 | 0.765 |
| 12232 | 0.716 |
| 12233 | 0.703 |
| 12234 | 0.581 |
| 12235 | 0.455 |
| 12241 | 0.630 |
| 12242 | 0.587 |
| 12243 | 0.576 |
| 12244 | 0.477 |
| 12245 | 0.374 |
| 12251 | 0.426 |
| 12252 | 0.393 |
| 12253 | 0.385 |
| 12254 | 0.320 |
| 12255 | 0.252 |
| 12311 | 0.822 |
| 12312 | 0.786 |
| 12312 | 0.776 |
| 12313 | 0.646 |
| 12314 | 0.511 |
| 12313 | 0.772 |
| 12321 | 0.723 |
| 12322 | 0.723 |
| 12323 | 0.710 |
| 12325 | 0.462 |
| 12331 | 0.759 |
| 12332 | 0.707 |
| 12333 | 0.693 |
| 12334 | 0.574 |
| 12335 | 0.449 |
| 12341 | 0.625 |
| 12342 | 0.580 |
| 12343 | 0.568 |
| 12344 | 0.471 |
| 12345 | 0.370 |
| 12351 | 0.424 |
| 12352 | 0.388 |
| 12353 | 0.379 |
| 12354 | 0.316 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 12355 | 0.250 |
| 12411 | 0.748 |
| 12412 | 0.717 |
| 12413 | 0.709 |
| 12414 | 0.597 |
| 12415 | 0.482 |
| 12421 | 0.703 |
| 12422 | 0.659 |
| 12423 | 0.648 |
| 12424 | 0.545 |
| 12425 | 0.438 |
| 12431 | 0.692 |
| 12432 | 0.645 |
| 12433 | 0.632 |
| 12434 | 0.531 |
| 12435 | 0.427 |
| 12441 | 0.573 |
| 12442 | 0.533 |
| 12443 | 0.522 |
| 12444 | 0.437 |
| 12445 | 0.348 |
| 12451 | 0.395 |
| 12452 | 0.364 |
| 12453 | 0.356 |
| 12454 | 0.295 |
| 12455 | 0.230 |
| 12511 | 0.596 |
| 12512 | 0.576 |
| 12512 | 0.571 |
| 12513 | 0.498 |
| 12514 | 0.422 |
| 12513 | 0.562 |
| 12522 | 0.529 |
| 12523 | 0.521 |
| 12524<br>12525 | 0.456 |
| | 0.388 |
| 12531 | 0.554 |
| 12532 | 0.518 |
| 12533 | 0.508 |
| 12534 | 0.445 |
| 12535 | 0.380 |
| 12541 | 0.466 |
| 12542 | 0.437 |
| 12543 | 0.429 |
| 12544 | 0.368 |
| 12545 | 0.304 |
| 12551 | 0.335 |
| 12552 | 0.315 |
| 12553 | 0.310 |
| 12554 | 0.251 |
| 12555 | 0.190 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 13111 | 0.825 |
| 13112 | 0.803 |
| 13113 | 0.797 |
| 13114 | 0.658 |
| 13115 | 0.514 |
| 13121 | 0.790 |
| 13122 | 0.754 |
| 13123 | 0.745 |
| 13124 | 0.614 |
| 13125 | 0.479 |
| 13131 | 0.781 |
| 13132 | 0.742 |
| 13133 | 0.732 |
| 13134 | 0.603 |
| 13135 | 0.470 |
| 13141 | 0.640 |
| 13142 | 0.608 |
| 13143 | 0.599 |
| 13144 | 0.493 |
| 13145 | 0.383 |
| 13151 | 0.363 |
| 13152 | 0.427 |
| 13153 | 0.400 |
| 13154 | 0.328 |
| 13155 | 0.328 |
| 13133 | |
| | 0.816 |
| 13212 | 0.781 |
| 13213 | 0.771 |
| 13214 | 0.641 |
| 13215 | 0.505 |
| 13221 | 0.767 |
| 13222 | 0.718 |
| 13223 | 0.705 |
| 13224 | 0.583 |
| 13225 | 0.456 |
| 13231 | 0.755 |
| 13232 | 0.702 |
| 13233 | 0.689 |
| 13234 | 0.569 |
| 13235 | 0.444 |
| 13241 | 0.620 |
| 13242 | 0.575 |
| 13243 | 0.563 |
| 13244 | 0.466 |
| 13245 | 0.364 |
| 13251 | 0.418 |
| 13252 | 0.383 |
| 13253 | 0.374 |
| 13254 | 0.311 |
| 13255 | 0.244 |
| 13311 | 0.814 |
| 15511 | 0.011 |



| Health State (5L profile) | US |
|---------------------------|----------------|
| 13312 | 0.775 |
| 13313 | 0.765 |
| 13314 | 0.636 |
| 13315 | 0.503 |
| 13321 | 0.761 |
| 13322 | 0.709 |
| 13323 | 0.695 |
| 13324 | 0.575 |
| 13325 | 0.451 |
| 13331 | 0.748 |
| 13332 | 0.693 |
| 13333 | 0.678 |
| 13334 | 0.560 |
| 13335 | 0.438 |
| 13341 | 0.615 |
| 13342 | 0.567 |
| 13343 | 0.554 |
| 13344 | 0.459 |
| 13345 | 0.360 |
| 13351 | 0.416 |
| 13352 | 0.378 |
| 13353 | 0.368 |
| 13354 | 0.306 |
| 13355 | 0.242 |
| 13411 | 0.740 |
| 13412 | 0.707 |
| 13413 | 0.699 |
| 13414 | 0.589 |
| 13415 | 0.474 |
| 13421 | 0.693 |
| 13422 | 0.647 |
| 13423 | 0.635 |
| 13424 | 0.533 |
| 13425 | 0.333 |
| 13423 | 0.682 |
| 13431 | 0.632 |
| 13432 | 0.619 |
| 13434 | 0.519 |
| 13434 | 0.319 |
| 13433 | 0.416 |
| 13441 | 0.564 |
| 13442 | |
| | 0.510 |
| 13444 | 0.426<br>0.339 |
| 13445 | |
| 13451 | 0.387 |
| 13452 | 0.355 |
| 13453 | 0.346 |
| 13454 | 0.286 |
| 13455 | 0.223 |
| 13511 | 0.590 |
| 13512 | 0.569 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 13513 | 0.563 |
| 13514 | 0.491 |
| 13515 | 0.416 |
| 13521 | 0.555 |
| 13522 | 0.519 |
| 13523 | 0.510 |
| 13524 | 0.447 |
| 13525 | 0.381 |
| 13531 | 0.546 |
| 13532 | 0.507 |
| 13533 | 0.497 |
| 13534 | 0.436 |
| 13535 | 0.372 |
| 13541 | 0.459 |
| 13542 | 0.427 |
| 13543 | 0.419 |
| 13544 | 0.359 |
| 13545 | 0.297 |
| 13551 | 0.329 |
| 13552 | 0.308 |
| 13553 | 0.302 |
| 13554 | 0.244 |
| 13555 | 0.184 |
| 14111 | 0.753 |
| 14112 | 0.733 |
| 14113 | 0.728 |
| 14114 | 0.604 |
| 14115 | 0.475 |
| 14121 | 0.720 |
| 14122 | 0.688 |
| 14123 | 0.680 |
| 14124 | 0.563 |
| 14125 | 0.442 |
| 14131 | 0.712 |
| 14132 | 0.677 |
| 14133 | 0.668 |
| 14134 | 0.553 |
| 14135 | 0.434 |
| 14141 | 0.583 |
| 14142 | 0.554 |
| 14143 | 0.546 |
| 14144 | 0.450 |
| 14145 | 0.349 |
| 14151 | 0.388 |
| 14152 | 0.369 |
| 14153 | 0.364 |
| 14154 | 0.294 |
| 14155 | 0.221 |
| 14211 | 0.746 |
| 14212 | 0.715 |
| 14213 | 0.706 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 14214 | 0.590 |
| 14215 | 0.469 |
| 14221 | 0.701 |
| 14222 | 0.656 |
| 14223 | 0.644 |
| 14224 | 0.536 |
| 14225 | 0.423 |
| 14231 | 0.690 |
| 14232 | 0.641 |
| 14233 | 0.629 |
| 14234 | 0.523 |
| 14235 | 0.412 |
| 14241 | 0.567 |
| 14242 | 0.525 |
| 14243 | 0.514 |
| 14244 | 0.426 |
| 14245 | 0.333 |
| 14251 | 0.382 |
| 14251 | 0.350 |
| 14253 | 0.342 |
| 14254 | 0.280 |
| 14255 | 0.215 |
| 14311 | 0.745 |
| 14312 | 0.710 |
| 14313 | 0.701 |
| 14314 | 0.586 |
| 14315 | 0.467 |
| 14321 | 0.696 |
| 14322 | 0.648 |
| 14323 | 0.635 |
| 14324 | 0.529 |
| 14325 | 0.419 |
| 14331 | 0.684 |
| 14332 | 0.633 |
| 14333 | 0.619 |
| 14334 | 0.515 |
| 14335 | 0.407 |
| 14341 | 0.563 |
| 14342 | 0.518 |
| 14343 | 0.506 |
| 14344 | 0.420 |
| 14345 | 0.330 |
| 14343 | 0.380 |
| 14351 | 0.346 |
| 14353 | 0.337 |
| 14354 | 0.337 |
| 14355 | 0.213 |
| 14333 | 0.213 |
| 14411 | 0.651 |
| 14412 | 0.631 |
| 14414 | 0.544 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 14415 | 0.440 |
| 14421 | 0.638 |
| 14422 | 0.595 |
| 14423 | 0.584 |
| 14424 | 0.492 |
| 14425 | 0.397 |
| 14431 | 0.627 |
| 14432 | 0.581 |
| 14433 | 0.569 |
| 14434 | 0.479 |
| 14435 | 0.386 |
| 14441 | 0.517 |
| 14442 | 0.478 |
| 14443 | 0.468 |
| 14444 | 0.390 |
| 14445 | 0.310 |
| 14451 | 0.353 |
| 14452 | 0.324 |
| 14453 | 0.316 |
| 14454 | 0.257 |
| 14455 | 0.196 |
| 14511 | 0.551 |
| 14512 | 0.532 |
| 14513 | 0.527 |
| 14514 | 0.457 |
| 14515 | 0.384 |
| 14521 | 0.518 |
| 14521 | 0.486 |
| 14523 | 0.478 |
| 14524 | 0.416 |
| 14525 | 0.351 |
| 14525 | 0.510 |
| 14531 | 0.475 |
| | 0.473 |
| 14533 | |
| 14534 | 0.406 |
| 14535 | 0.343 |
| 14541 | 0.425 |
| 14542 | 0.396 |
| 14543 | 0.389 |
| 14544 | 0.331 |
| 14545 | 0.270 |
| 14551 | 0.297 |
| 14552 | 0.278 |
| 14553 | 0.273 |
| 14554 | 0.217 |
| 14555 | 0.160 |
| 15111 | 0.529 |
| 15112 | 0.516 |
| 15113 | 0.512 |
| 15114 | 0.435 |
| 15115 | 0.355 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 15121 | 0.503 |
| 15122 | 0.482 |
| 15123 | 0.477 |
| 15124 | 0.404 |
| 15125 | 0.328 |
| 15131 | 0.496 |
| 15132 | 0.474 |
| 15133 | 0.468 |
| 15134 | 0.396 |
| 15135 | 0.321 |
| 15141 | 0.405 |
| 15142 | 0.386 |
| 15143 | 0.381 |
| 15144 | 0.313 |
| 15145 | 0.242 |
| 15151 | 0.268 |
| 15152 | 0.255 |
| 15153 | 0.251 |
| 15154 | 0.188 |
| 15155 | 0.123 |
| 15211 | 0.529 |
| 15212 | 0.509 |
| 15212 | 0.503 |
| 15213 | 0.303 |
| 15214 | 0.450 |
| 15215 | 0.496 |
| 15222 | 0.463 |
| 15223 | 0.403 |
| 15225 | 0.389 |
| 15224 | 0.389 |
| 15225 | 0.321 |
| 15231 | 0.457 |
| 15232 | 0.432 |
| 15235 | 0.442 |
| | 0.379 |
| 15235 | |
| 15241 | 0.400 |
| 15242 | 0.370 |
| 15243 | 0.362 |
| 15244 | 0.301 |
| 15245 | 0.237 |
| 15251 | 0.268 |
| 15252 | 0.248 |
| 15253 | 0.242 |
| 15254 | 0.184 |
| 15255 | 0.123 |
| 15311 | 0.529 |
| 15312 | 0.507 |
| 15313 | 0.501 |
| 15314 | 0.429 |
| 15315 | 0.354 |
| 15321 | 0.494 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 15322 | 0.458 |
| 15323 | 0.449 |
| 15324 | 0.385 |
| 15325 | 0.319 |
| 15331 | 0.485 |
| 15332 | 0.446 |
| 15333 | 0.436 |
| 15334 | 0.374 |
| 15335 | 0.310 |
| 15341 | 0.398 |
| 15342 | 0.366 |
| 15343 | 0.358 |
| 15344 | 0.298 |
| 15345 | 0.235 |
| 15351 | 0.268 |
| 15352 | 0.246 |
| 15353 | 0.240 |
| 15354 | 0.183 |
| 15355 | 0.123 |
| 15411 | 0.497 |
| 15412 | 0.478 |
| 15413 | 0.472 |
| 15414 | 0.403 |
| 15415 | 0.332 |
| 15421 | 0.464 |
| 15422 | 0.434 |
| 15423 | 0.426 |
| 15424 | 0.364 |
| 15425 | 0.299 |
| 15431 | 0.456 |
| 15432 | 0.423 |
| 15433 | 0.414 |
| 15434 | 0.354 |
| 15435 | 0.291 |
| 15441 | 0.372 |
| 15442 | 0.344 |
| 15443 | 0.337 |
| 15444 | 0.279 |
| 15445 | 0.219 |
| 15451 | 0.245 |
| 15452 | 0.226 |
| 15453 | 0.221 |
| 15454 | 0.167 |
| 15455 | 0.110 |
| 15511 | 0.431 |
| 15512 | 0.418 |
| 15513 | 0.414 |
| 15514 | 0.351 |
| 15515 | 0.286 |
| 15521 | 0.404 |
| 15522 | 0.384 |



| Health State (5L profile) | US |
|---------------------------|----------------|
| 15523 | 0.379 |
| 15524 | 0.320 |
| 15525 | 0.260 |
| 15531 | 0.397 |
| 15532 | 0.376 |
| 15533 | 0.370 |
| 15534 | 0.313 |
| 15535 | 0.253 |
| 15541 | 0.318 |
| 15542 | 0.300 |
| 15543 | 0.295 |
| 15544 | 0.241 |
| 15545 | 0.186 |
| 15551 | 0.199 |
| 15552 | 0.186 |
| 15553 | 0.182 |
| 15554 | 0.134 |
| 15555 | 0.084 |
| 21111 | 0.880 |
| 21112 | 0.840 |
| 21113 | 0.830 |
| 21114 | 0.690 |
| 21115 | 0.544 |
| 21121 | 0.826 |
| 21122 | 0.790 |
| 21123 | 0.780 |
| 21123 | 0.648 |
| 21125 | 0.511 |
| 21123 | 0.813 |
| 21131 | 0.777 |
| 21132 | 0.768 |
| 21133 | 0.638 |
| 21134 | 0.502 |
| 21133 | 0.502 |
| 21142<br>21143 | 0.641<br>0.634 |
| 21144 | 0.526 |
| 21145 | 0.415 |
| 21151 | 0.457 |
| 21152 | 0.437 |
| 21153 | 0.432 |
| 21154 | 0.359 |
| 21155 | 0.283 |
| 21211 | 0.853 |
| 21212 | 0.816 |
| 21213 | 0.807 |
| 21214 | 0.675 |
| 21215 | 0.538 |
| 21221 | 0.803 |
| 21222 | 0.756 |
| 21223 | 0.744 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 21224 | 0.620 |
| 21225 | 0.491 |
| 21231 | 0.790 |
| 21232 | 0.741 |
| 21233 | 0.728 |
| 21234 | 0.606 |
| 21235 | 0.480 |
| 21241 | 0.655 |
| 21242 | 0.612 |
| 21243 | 0.601 |
| 21244 | 0.502 |
| 21245 | 0.398 |
| 21251 | 0.451 |
| 21252 | 0.418 |
| 21253 | 0.409 |
| 21254 | 0.344 |
| 21255 | 0.276 |
| 21311 | 0.846 |
| 21312 | 0.810 |
| 21312 | 0.801 |
| 21313 | 0.671 |
| 21314 | 0.536 |
| 21313 | 0.797 |
| 21321 | 0.797 |
| 21322 | 0.748 |
| 21323 | 0.735 |
| 21325 | 0.486 |
| 21331 | 0.785 |
| 21332 | 0.732 |
| 21333 | 0.719 |
| 21334 | 0.599 |
| 21335 | 0.474 |
| 21341 | 0.651 |
| 21342 | 0.605 |
| 21343 | 0.593 |
| 21344 | 0.495 |
| 21345 | 0.394 |
| 21351 | 0.449 |
| 21352 | 0.413 |
| 21353 | 0.404 |
| 21354 | 0.340 |
| 21355 | 0.274 |
| 21411 | 0.772 |
| 21412 | 0.741 |
| 21413 | 0.733 |
| 21414 | 0.622 |
| 21415 | 0.507 |
| 21421 | 0.728 |
| 21422 | 0.684 |
| 21423 | 0.673 |
| 21424 | 0.569 |



| Health State (5L profile) | US |
|---------------------------|--------------------|
| 21425 | 0.462 |
| 21431 | 0.717 |
| 21432 | 0.670 |
| 21433 | 0.658 |
| 21434 | 0.556 |
| 21435 | 0.451 |
| 21441 | 0.598 |
| 21442 | 0.558 |
| 21443 | 0.547 |
| 21444 | 0.462 |
| 21445 | 0.373 |
| 21451 | 0.420 |
| 21452 | 0.389 |
| 21453 | 0.381 |
| 21454 | 0.319 |
| 21455 | 0.255 |
| 21511 | 0.620 |
| 21512 | 0.600 |
| 21513 | 0.595 |
| 21514 | 0.522 |
| 21515 | 0.446 |
| 21515 | 0.586 |
| 21521 | 0.554 |
| 21522 | 0.546 |
| 21525 | 0.346 |
| 21524 | 0.480 |
| 21531 | 0.578 |
| 21532 | 0.543 |
| 21533 | 0.534 |
| 21534 | 0.470 |
| 21535 | 0.404 |
| 21541 | 0.491 |
| 21542 | 0.462 |
| 21543 | 0.454 |
| 21544 | 0.392 |
| 21545 | 0.329 |
| 21551 | 0.359 |
| 21552 | 0.339 |
| 21553 | 0.334 |
| 21554 | 0.276 |
| 21555 | 0.215 |
| 22111 | 0.823 |
| 22112 | 0.786 |
| 22113 | 0.777 |
| 22114 | 0.645 |
| 22115 | 0.507 |
| 22121 | 0.772 |
| 22122 | 0.725 |
| 22122 | 0.713 |
| 22123 | 0.589 |
| 22124 | 0.389 |
| 22123 | V. <del>T</del> U1 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 22131 | 0.760 |
| 22132 | 0.710 |
| 22133 | 0.697 |
| 22134 | 0.575 |
| 22135 | 0.449 |
| 22141 | 0.624 |
| 22142 | 0.581 |
| 22143 | 0.570 |
| 22144 | 0.471 |
| 22145 | 0.368 |
| 22151 | 0.420 |
| 22152 | 0.387 |
| 22153 | 0.379 |
| 22154 | 0.314 |
| 22155 | 0.246 |
| 22211 | 0.799 |
| 22212 | 0.751 |
| 22213 | 0.739 |
| 22214 | 0.616 |
| 22215 | 0.487 |
| 22221 | 0.738 |
| 22222 | 0.678 |
| 22223 | 0.662 |
| 22224 | 0.547 |
| 22225 | 0.427 |
| 22231 | 0.723 |
| 22232 | 0.659 |
| 22233 | 0.643 |
| 22234 | 0.530 |
| 22235 | 0.412 |
| 22241 | 0.594 |
| 22241 | 0.537 |
| 22242 | 0.523 |
| 22243 | 0.432 |
| 22244 | 0.432 |
| 22251 | 0.338 |
| 22251 | 0.354 |
| 22252 | 0.334 |
| 22253 | 0.342 |
| 22255 | 0.283 |
| 22311 | 0.793 |
| 22312 | 0.743 |
| 22313 | 0.730 |
| 22314 | 0.609 |
| 22315 | 0.483 |
| 22321 | 0.729 |
| 22322 | 0.666 |
| 22323 | 0.649 |
| 22324 | 0.536 |
| 22325 | 0.419 |
| 22331 | 0.714 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 22332 | 0.647 |
| 22333 | 0.629 |
| 22334 | 0.518 |
| 22335 | 0.403 |
| 22341 | 0.587 |
| 22342 | 0.527 |
| 22343 | 0.511 |
| 22344 | 0.422 |
| 22345 | 0.330 |
| 22351 | 0.396 |
| 22352 | 0.346 |
| 22353 | 0.333 |
| 22354 | 0.278 |
| 22355 | 0.221 |
| 22411 | 0.724 |
| 22412 | 0.680 |
| 22413 | 0.668 |
| 22414 | 0.565 |
| 22415 | 0.459 |
| 22421 | 0.666 |
| 22422 | 0.608 |
| 22423 | 0.593 |
| 22424 | 0.498 |
| 22425 | 0.400 |
| 22431 | 0.652 |
| 22431 | 0.590 |
| 22433 | 0.574 |
| 22434 | 0.482 |
| 22435 | 0.386 |
| 22441 | 0.540 |
| 22442 | 0.485 |
| 22442 | 0.483 |
| 22443 | |
| | 0.394 |
| 22445 | 0.314 |
| 22451 | 0.372 |
| 22452 | 0.327 |
| 22453 | 0.316 |
| 22454 | 0.262 |
| 22455 | 0.207 |
| 22511 | 0.583 |
| 22512 | 0.550 |
| 22513 | 0.542 |
| 22514 | 0.477 |
| 22515 | 0.409 |
| 22521 | 0.537 |
| 22522 | 0.490 |
| 22523 | 0.478 |
| 22524 | 0.421 |
| 22525 | 0.362 |
| 22531 | 0.525 |
| 22532 | 0.475 |



| Health State (5L profile) |
|---|
| 22534 0.407 22535 0.351 22541 0.444 22542 0.401 22543 0.390 22544 0.337 22545 0.282 22551 0.322 22552 0.289 22553 0.281 22554 0.230 22555 0.178 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.569 23144 0.615 23145 0.557 23146 0.557 23 |
| 22535 0.351 22541 0.444 22542 0.401 22543 0.390 22544 0.337 22545 0.282 22551 0.322 22552 0.289 22553 0.281 22554 0.230 22555 0.178 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.499 23141 0.615 23142 0.569 23141 0.615 23142 0.569 23143 0.569 23144 |
| 22541 0.444 22542 0.401 22543 0.390 22544 0.337 22545 0.282 22551 0.322 22552 0.289 22553 0.281 22554 0.230 22555 0.178 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.499 23141 0.615 23142 0.569 23143 0.569 23144 0.606 23145 0.359 23151 0.413 |
| 22542 0.401 22543 0.390 22544 0.337 22545 0.282 22551 0.322 22552 0.289 22553 0.281 22554 0.230 22555 0.178 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.569 23144 0.605 23145 0.359 23145 0.359 23151 0.413 |
| 22543 0.390 22544 0.337 22545 0.282 22551 0.322 22552 0.289 22553 0.281 22554 0.230 22555 0.178 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 22544 0.337 22545 0.282 22551 0.322 22552 0.289 22553 0.281 22554 0.230 22555 0.178 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.615 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 22545 0.282 22551 0.322 22552 0.289 22553 0.281 22554 0.230 22555 0.178 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.60 23145 0.359 23147 0.460 23148 0.359 23151 0.413 |
| 22551 0.322 22552 0.289 22553 0.281 22554 0.230 22555 0.178 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23121 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.557 23145 0.359 23151 0.413 |
| 22552 0.289 22553 0.281 22554 0.230 22555 0.178 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.400 23145 0.359 23151 0.413 |
| 22553 0.281 22554 0.230 22555 0.178 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 22554 0.230 22555 0.178 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 22555 0.178 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23111 0.811 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23112 0.775 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23113 0.766 23114 0.635 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23114 0.635 23121 0.500 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23115 0.500 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23121 0.761 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23122 0.712 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23123 0.699 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23124 0.577 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23125 0.451 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23131 0.749 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23132 0.696 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23133 0.683 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23134 0.563 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23135 0.439 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23141 0.615 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23142 0.569 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23143 0.557 23144 0.460 23145 0.359 23151 0.413 |
| 23144 0.460 23145 0.359 23151 0.413 |
| 23145 0.359<br>23151 0.413 |
| 23151 0.413 |
| 72157 |
| 23153 0.368 |
| 23154 0.305 |
| 23155 0.239 |
| 23211 0.788 |
| 23212 0.738 |
| 23213 0.726 |
| 23214 0.604 |
| 23215 0.477 |
| 23221 0.725 |
| 23222 0.662 |
| 23223 0.645 |
| 23224 0.532 |
| 23225 0.414 |
| 23231 0.709 |
| 23232 0.643 |
| 23233 0.626 |



| TIIdl. Co. 4 (#T | TIO |
|---------------------------|-------|
| Health State (5L profile) | US |
| 23234 | 0.514 |
| 23235 | 0.399 |
| 23241 | 0.582 |
| 23242 | 0.522 |
| 23243 | 0.507 |
| 23244 | 0.418 |
| 23245 | 0.326 |
| 23251 | 0.390 |
| 23252 | 0.341 |
| 23253 | 0.328 |
| 23254 | 0.273 |
| 23255 | 0.216 |
| 23311 | 0.782 |
| 23312 | 0.729 |
| 23313 | 0.716 |
| 23314 | 0.596 |
| 23315 | 0.472 |
| 23321 | 0.716 |
| 23322 | 0.649 |
| 23323 | 0.632 |
| 23324 | 0.521 |
| 23325 | 0.405 |
| 23323 | 0.700 |
| 23332 | 0.630 |
| 23332 | 0.611 |
| 23334 | 0.502 |
| 23335 | 0.389 |
| 23333 | 0.574 |
| 23341 | 0.574 |
| 23343 | 0.494 |
| 23344 | 0.408 |
| 23345 | 0.318 |
| 23351 | 0.385 |
| 23352 | 0.332 |
| 23353 | 0.319 |
| 23354 | 0.266 |
| 23355 | 0.211 |
| 23411 | 0.714 |
| 23412 | 0.667 |
| 23413 | 0.655 |
| 23414 | 0.554 |
| 23415 | 0.449 |
| 23421 | 0.654 |
| 23422 | 0.593 |
| 23423 | 0.577 |
| 23424 | 0.484 |
| 23425 | 0.388 |
| 23431 | 0.639 |
| 23432 | 0.574 |
| 23433 | 0.558 |
| 23434 | 0.467 |
| 25.51 | 0.107 |


| Haalda CA-4- (#T Pl.) | TIC |
|---------------------------|---------------------|
| Health State (5L profile) | US |
| 23435 | 0.373 |
| 23441 | 0.528 |
| 23442 | 0.471 |
| 23443 | 0.456 |
| 23444 | 0.381 |
| 23445 | 0.303 |
| 23451 | 0.362 |
| 23452 | 0.315 |
| 23453 | 0.303 |
| 23454 | 0.251 |
| 23455 | 0.197 |
| 23511 | 0.576 |
| 23512 | 0.540 |
| 23513 | 0.531 |
| 23514 | 0.468 |
| 23515 | 0.402 |
| 23521 | 0.527 |
| 23522 | 0.477 |
| 23523 | 0.464 |
| 23524 | 0.409 |
| 23525 | 0.352 |
| 23525 | 0.532 |
| 23531 | 0.313 |
| 23532 | 0.462 |
| | 0.395 |
| 23534 | |
| 23535 | 0.340 |
| 23541 | 0.435 |
| 23542 | 0.389 |
| 23543 | 0.377 |
| 23544 | 0.325 |
| 23545 | 0.272 |
| 23551 | 0.315 |
| 23552 | 0.279 |
| 23553 | 0.270 |
| 23554 | 0.221 |
| 23555 | 0.170 |
| 24111 | 0.741 |
| 24112 | 0.709 |
| 24113 | 0.701 |
| 24114 | 0.584 |
| 24115 | 0.463 |
| 24121 | 0.695 |
| 24122 | 0.650 |
| 24123 | 0.638 |
| 24124 | 0.530 |
| 24125 | 0.418 |
| 24131 | 0.684 |
| 24132 | 0.636 |
| 24132 | 0.623 |
| 24133 | 0.023 |
| 24134 | 0.317 |
| L 24133 | U. <del>4</del> U / |



| Health State (5L profile) | US |
|---------------------------|-------|
| 24141 | 0.561 |
| 24142 | 0.519 |
| 24143 | 0.508 |
| 24144 | 0.420 |
| 24145 | 0.328 |
| 24151 | 0.376 |
| 24152 | 0.344 |
| 24153 | 0.336 |
| 24154 | 0.274 |
| 24155 | 0.210 |
| 24211 | 0.722 |
| 24212 | 0.677 |
| 24213 | 0.665 |
| 24214 | 0.557 |
| 24215 | 0.444 |
| 24221 | 0.663 |
| 24222 | 0.604 |
| 24223 | 0.589 |
| 24224 | 0.489 |
| 24225 | 0.385 |
| 24231 | 0.648 |
| 24232 | 0.586 |
| 24233 | 0.570 |
| 24234 | 0.472 |
| 24235 | 0.371 |
| 24241 | 0.532 |
| 24242 | 0.477 |
| 24243 | 0.462 |
| 24244 | 0.382 |
| 24245 | 0.299 |
| 24251 | 0.357 |
| 24252 | 0.312 |
| 24253 | 0.301 |
| 24254 | 0.247 |
| 24255 | 0.191 |
| 24311 | 0.717 |
| 24312 | 0.669 |
| 24313 | 0.656 |
| 24314 | 0.550 |
| 24315 | 0.440 |
| 24321 | 0.655 |
| 24322 | 0.593 |
| 24323 | 0.577 |
| 24324 | 0.479 |
| 24325 | 0.377 |
| 24331 | 0.640 |
| 24332 | 0.574 |
| 24333 | 0.557 |
| 24334 | 0.461 |
| 24335 | 0.362 |
| 24341 | 0.525 |



| TIId. Co. (#T | TIC |
|---------------------------|-------|
| Health State (5L profile) | US |
| 24342 | 0.466 |
| 24343 | 0.451 |
| 24344 | 0.373 |
| 24345 | 0.292 |
| 24351 | 0.353 |
| 24352 | 0.305 |
| 24353 | 0.292 |
| 24354 | 0.240 |
| 24355 | 0.186 |
| 24411 | 0.659 |
| 24412 | 0.616 |
| 24413 | 0.604 |
| 24414 | 0.513 |
| 24415 | 0.418 |
| 24421 | 0.602 |
| 24422 | 0.545 |
| 24423 | 0.531 |
| 24424 | 0.447 |
| 24425 | 0.361 |
| 24431 | 0.588 |
| 24432 | 0.528 |
| 24433 | 0.512 |
| 24434 | 0.431 |
| 24435 | 0.431 |
| 24443 | 0.347 |
| 24441 | 0.483 |
| 24443 | 0.418 |
| 24444 | 0.349 |
| 24445 | 0.277 |
| 24451 | 0.331 |
| 24452 | 0.288 |
| 24453 | 0.277 |
| 24454 | 0.226 |
| 24455 | 0.173 |
| 24511 | 0.539 |
| 24512 | 0.507 |
| 24513 | 0.499 |
| 24514 | 0.437 |
| 24515 | 0.372 |
| 24521 | 0.494 |
| 24522 | 0.448 |
| 24523 | 0.437 |
| 24524 | 0.383 |
| 24525 | 0.327 |
| 24531 | 0.483 |
| 24532 | 0.434 |
| 24533 | 0.421 |
| 24534 | 0.369 |
| 24535 | 0.315 |
| 24533 | 0.404 |
| 24541 | 0.362 |
| ムオノオム | 0.302 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 24543 | 0.351 |
| 24544 | 0.301 |
| 24545 | 0.248 |
| 24551 | 0.286 |
| 24552 | 0.254 |
| 24553 | 0.245 |
| 24554 | 0.197 |
| 24555 | 0.148 |
| 25111 | 0.523 |
| 25112 | 0.503 |
| 25113 | 0.498 |
| 25114 | 0.425 |
| 25115 | 0.349 |
| 25121 | 0.490 |
| 25122 | 0.457 |
| 25123 | 0.449 |
| 25124 | 0.383 |
| 25125 | 0.315 |
| 25131 | 0.481 |
| 25132 | 0.446 |
| 25133 | 0.437 |
| 25134 | 0.373 |
| 25135 | 0.307 |
| 25141 | 0.394 |
| 25142 | 0.365 |
| 25143 | 0.357 |
| 25144 | 0.295 |
| 25145 | 0.232 |
| 25151 | 0.262 |
| 25151 | 0.242 |
| 25153 | 0.237 |
| 25155 | 0.179 |
| 25154 | 0.118 |
| 25133 | 0.517 |
| 25211 | 0.484 |
| 25212 | 0.475 |
| 25213 | 0.473 |
| 25214 | 0.342 |
| | 0.342 |
| 25221<br>25222 | 0.470 |
| 25223 | 0.412 |
| 25224 | 0.355 |
| 25225 | 0.296 |
| 25231 | 0.459 |
| 25232 | 0.409 |
| 25233 | 0.397 |
| 25234 | 0.342 |
| 25235 | 0.284 |
| 25241 | 0.377 |
| 25242 | 0.335 |
| 25243 | 0.324 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 25244 | 0.270 |
| 25245 | 0.215 |
| 25251 | 0.255 |
| 25252 | 0.223 |
| 25253 | 0.214 |
| 25254 | 0.164 |
| 25255 | 0.111 |
| 25311 | 0.515 |
| 25312 | 0.479 |
| 25313 | 0.470 |
| 25314 | 0.406 |
| 25315 | 0.340 |
| 25321 | 0.465 |
| 25322 | 0.416 |
| 25323 | 0.403 |
| 25324 | 0.348 |
| 25325 | 0.291 |
| 25331 | 0.453 |
| 25332 | 0.400 |
| 25333 | 0.387 |
| 25334 | 0.334 |
| 25335 | 0.279 |
| 25341 | 0.373 |
| 25342 | 0.328 |
| 25343 | 0.316 |
| 25344 | 0.264 |
| 25345 | 0.211 |
| 25351 | 0.253 |
| 25352 | 0.218 |
| 25353 | 0.209 |
| 25354 | 0.160 |
| 25355 | 0.109 |
| 25411 | 0.486 |
| 25412 | 0.455 |
| 25413 | 0.447 |
| 25414 | 0.385 |
| 25415 | 0.320 |
| 25421 | 0.441 |
| 25422 | 0.397 |
| 25423 | 0.386 |
| 25424 | 0.332 |
| 25425 | 0.276 |
| 25431 | 0.430 |
| 25432 | 0.383 |
| 25433 | 0.371 |
| 25434 | 0.319 |
| 25435 | 0.265 |
| 25441 | 0.352 |
| 25442 | 0.311 |
| 25443 | 0.301 |
| 25444 | 0.251 |



| TT 1/1 C/ /#T #1 \ | XIO. |
|---------------------------|-------|
| Health State (5L profile) | US |
| 25445 | 0.199 |
| 25451 | 0.234 |
| 25452 | 0.203 |
| 25453 | 0.195 |
| 25454 | 0.148 |
| 25455 | 0.099 |
| 25511 | 0.425 |
| 25512 | 0.405 |
| 25513 | 0.400 |
| 25514 | 0.341 |
| 25515 | 0.280 |
| 25521 | 0.391 |
| 25522 | 0.359 |
| 25523 | 0.350 |
| 25524 | 0.299 |
| 25525 | 0.247 |
| 25531 | 0.383 |
| 25532 | 0.347 |
| 25533 | 0.338 |
| 25534 | 0.289 |
| 25535 | 0.238 |
| 25541 | 0.308 |
| 25542 | 0.278 |
| 25543 | 0.270 |
| 25544 | 0.223 |
| 25545 | 0.174 |
| 25551 | 0.194 |
| 25552 | 0.173 |
| 25553 | 0.168 |
| 25554 | 0.108 |
| 25555 | 0.078 |
| 31111 | 0.854 |
| 31112 | 0.833 |
| 31112 | 0.833 |
| 31114 | 0.827 |
| | 0.688 |
| 31115 | |
| 31121 | 0.819 |
| 31122 | 0.783 |
| 31123 | 0.774 |
| 31124 | 0.643 |
| 31125 | 0.508 |
| 31131 | 0.810 |
| 31132 | 0.771 |
| 31133 | 0.761 |
| 31134 | 0.632 |
| 31135 | 0.499 |
| 31141 | 0.669 |
| 31142 | 0.637 |
| 31143 | 0.628 |
| 31144 | 0.522 |
| 31145 | 0.412 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 31151 | 0.456 |
| 31152 | 0.435 |
| 31153 | 0.429 |
| 31154 | 0.357 |
| 31155 | 0.282 |
| 31211 | 0.845 |
| 31212 | 0.810 |
| 31213 | 0.801 |
| 31214 | 0.670 |
| 31215 | 0.535 |
| 31221 | 0.796 |
| 31222 | 0.748 |
| 31223 | 0.735 |
| 31224 | 0.613 |
| 31225 | 0.486 |
| 31231 | 0.784 |
| 31232 | 0.732 |
| 31233 | 0.719 |
| 31234 | 0.598 |
| 31235 | 0.473 |
| 31241 | 0.650 |
| 31242 | 0.604 |
| 31243 | 0.593 |
| 31244 | 0.495 |
| 31245 | 0.393 |
| 31251 | 0.448 |
| 31252 | 0.413 |
| 31253 | 0.403 |
| 31254 | 0.340 |
| 31255 | 0.273 |
| 31311 | 0.843 |
| 31312 | 0.804 |
| 31313 | 0.794 |
| 31314 | 0.666 |
| 31315 | 0.533 |
| 31313 | 0.791 |
| 31321 | 0.739 |
| 31322 | 0.735 |
| 31323 | 0.723 |
| 31324 | 0.480 |
| 31331 | 0.778 |
| 31332 | 0.723 |
| 31333 | 0.708 |
| 31334 | 0.590 |
| 31335 | 0.467 |
| 31341 | 0.645 |
| 31342 | 0.597 |
| 31343 | 0.584 |
| 31344 | 0.488 |
| 31345 | 0.389 |
| 31351 | 0.446 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 31352 | 0.407 |
| 31353 | 0.397 |
| 31354 | 0.335 |
| 31355 | 0.271 |
| 31411 | 0.769 |
| 31412 | 0.736 |
| 31413 | 0.728 |
| 31414 | 0.618 |
| 31415 | 0.504 |
| 31421 | 0.723 |
| 31422 | 0.676 |
| 31423 | 0.664 |
| 31424 | 0.563 |
| 31425 | 0.457 |
| 31431 | 0.711 |
| 31432 | 0.662 |
| 31432 | 0.649 |
| 31434 | 0.549 |
| 31435 | 0.445 |
| 31441 | 0.594 |
| 31442 | 0.551 |
| 31442 | 0.539 |
| 31444 | 0.339 |
| 31445 | 0.433 |
| 31443 | 0.308 |
| 31451 | 0.417 |
| 31453 | 0.375 |
| 31454 | 0.315 |
| 31455 | 0.252 |
| 31511 | 0.619 |
| 31512 | 0.598 |
| 31513 | 0.592 |
| 31514 | 0.520 |
| 31515 | 0.445 |
| 31521 | 0.584 |
| 31522 | 0.549 |
| 31523 | 0.540 |
| 31524 | 0.476 |
| 31525 | 0.410 |
| 31531 | 0.575 |
| 31532 | 0.537 |
| 31533 | 0.527 |
| 31534 | 0.465 |
| 31535 | 0.401 |
| 31541 | 0.488 |
| 31542 | 0.457 |
| 31543 | 0.449 |
| 31544 | 0.389 |
| 31545 | 0.326 |
| 31551 | 0.358 |
| 31552 | 0.337 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 31553 | 0.331 |
| 31554 | 0.274 |
| 31555 | 0.214 |
| 32111 | 0.816 |
| 32112 | 0.780 |
| 32113 | 0.770 |
| 32114 | 0.640 |
| 32115 | 0.505 |
| 32121 | 0.766 |
| 32122 | 0.716 |
| 32123 | 0.704 |
| 32124 | 0.582 |
| 32125 | 0.455 |
| 32131 | 0.753 |
| 32132 | 0.701 |
| 32133 | 0.687 |
| 32134 | 0.567 |
| 32135 | 0.443 |
| 32141 | 0.619 |
| 32142 | 0.573 |
| 32143 | 0.561 |
| 32144 | 0.464 |
| 32145 | 0.364 |
| 32151 | 0.418 |
| 32152 | 0.382 |
| 32152 | 0.372 |
| 32154 | 0.372 |
| 32154 | 0.244 |
| 3213 | 0.792 |
| 32211 | 0.743 |
| 32212 | 0.743 |
| | 0.608 |
| 32214 | |
| 32215 | 0.482 |
| 32221 | 0.729 |
| 32222 | 0.666 |
| 32223 | 0.650 |
| 32224 | 0.536 |
| 32225 | 0.419 |
| 32231 | 0.714 |
| 32232 | 0.647 |
| 32233 | 0.630 |
| 32234 | 0.518 |
| 32235 | 0.403 |
| 32241 | 0.586 |
| 32242 | 0.527 |
| 32243 | 0.511 |
| 32244 | 0.422 |
| 32245 | 0.330 |
| 32251 | 0.395 |
| 32252 | 0.346 |
| 32253 | 0.333 |



| Health State (5L profile) | US |
|---------------------------|----------------|
| 32254 | 0.278 |
| 32254<br>32255 | 0.278 |
| 32311 | 0.786 |
| 32312 | 0.734 |
| 32313 | 0.720 |
| 32314 | 0.600 |
| 32315 | 0.476 |
| 32321 | 0.720 |
| 32322 | 0.654 |
| 32323 | 0.636 |
| 32324 | 0.525 |
| 32325 | 0.410 |
| 32331 | 0.704 |
| 32332 | 0.634 |
| 32333 | 0.616 |
| 32334 | 0.506 |
| 32335 | 0.393 |
| 32341 | 0.578 |
| 32342 | 0.515 |
| 32343 | 0.499 |
| 32344 | 0.412 |
| 32345 | 0.322 |
| 32351 | 0.389 |
| 32352 | 0.337 |
| 32353 | 0.323 |
| 32354 | 0.323 |
| 32355 | 0.276 |
| 32411 | 0.213 |
| 32411 | |
| | 0.672 |
| 32413 | 0.659<br>0.558 |
| 32414 | |
| 32415 | 0.454 |
| 32421 | 0.658 |
| 32422 | 0.597 |
| 32423 | 0.581 |
| 32424 | 0.489 |
| 32425 | 0.392 |
| 32431 | 0.643 |
| 32432 | 0.579 |
| 32433 | 0.562 |
| 32434 | 0.471 |
| 32435 | 0.377 |
| 32441 | 0.533 |
| 32442 | 0.475 |
| 32443 | 0.460 |
| 32444 | 0.385 |
| 32445 | 0.307 |
| 32451 | 0.367 |
| 32452 | 0.319 |
| 32453 | 0.307 |
| 32454 | 0.255 |
| 32 13 1 | 0.233 |



| II I/I C/ / (FI PI) | TIG. |
|---------------------------|-------|
| Health State (5L profile) | US |
| 32455 | 0.202 |
| 32511 | 0.581 |
| 32512 | 0.545 |
| 32513 | 0.535 |
| 32514 | 0.472 |
| 32515 | 0.407 |
| 32521 | 0.531 |
| 32522 | 0.482 |
| 32523 | 0.469 |
| 32524 | 0.414 |
| 32525 | 0.357 |
| 32531 | 0.519 |
| 32532 | 0.466 |
| 32533 | 0.452 |
| 32534 | 0.399 |
| 32535 | 0.344 |
| 32541 | 0.440 |
| 32542 | 0.393 |
| 32543 | 0.381 |
| 32544 | 0.330 |
| 32545 | 0.277 |
| 32545 | 0.320 |
| 32552 | 0.284 |
| 32553 | 0.274 |
| 32554 | 0.226 |
| 32555 | 0.226 |
| 33111 | 0.808 |
| 33112 | 0.769 |
| 33113 | 0.759 |
| 33114 | 0.630 |
| 33115 | 0.497 |
| 33121 | 0.755 |
| 33122 | 0.703 |
| 33123 | 0.689 |
| 33124 | 0.569 |
| 33125 | 0.445 |
| 33131 | 0.742 |
| 33132 | 0.687 |
| 33133 | 0.672 |
| 33134 | 0.554 |
| 33135 | 0.432 |
| 33141 | 0.609 |
| 33142 | 0.561 |
| 33143 | 0.548 |
| 33144 | 0.453 |
| 33145 | 0.354 |
| 33151 | 0.410 |
| 33152 | 0.371 |
| 33153 | 0.361 |
| 33154 | 0.300 |
| 33155 | 0.236 |
| 33133 | 0.250 |



| Haaldh Chair (#1 @1.\ | TIC |
|---------------------------|-------|
| Health State (5L profile) | US |
| 33211 | 0.782 |
| 33212 | 0.729 |
| 33213 | 0.716 |
| 33214 | 0.596 |
| 33215 | 0.471 |
| 33221 | 0.716 |
| 33222 | 0.650 |
| 33223 | 0.633 |
| 33224 | 0.521 |
| 33225 | 0.405 |
| 33231 | 0.700 |
| 33232 | 0.630 |
| 33233 | 0.612 |
| 33234 | 0.502 |
| 33235 | 0.389 |
| 33241 | 0.574 |
| 33242 | 0.511 |
| 33243 | 0.495 |
| 33244 | 0.408 |
| 33245 | 0.317 |
| 33251 | 0.384 |
| 33252 | 0.332 |
| 33253 | 0.319 |
| 33254 | 0.265 |
| 33255 | 0.210 |
| 33311 | 0.775 |
| 33312 | 0.720 |
| 33312 | 0.720 |
| 33314 | 0.703 |
| 33315 | 0.387 |
| 33313 | 0.463 |
| 33322 | |
| 33322 | 0.637 |
| | 0.619 |
| 33324 | 0.509 |
| 33325 | 0.395 |
| 33331 | 0.689 |
| 33332 | 0.616 |
| 33333 | 0.597 |
| 33334 | 0.490 |
| 33335 | 0.378 |
| 33341 | 0.565 |
| 33342 | 0.499 |
| 33343 | 0.482 |
| 33344 | 0.397 |
| 33345 | 0.309 |
| 33351 | 0.378 |
| 33352 | 0.323 |
| 33353 | 0.308 |
| 33354 | 0.257 |
| 33355 | 0.204 |
| 33411 | 0.709 |



| Hoolth State (51 Cla) | US |
|---------------------------|-------|
| Health State (5L profile) | |
| 33412 | 0.659 |
| 33413 | 0.646 |
| 33414 | 0.546 |
| 33415 | 0.443 |
| 33421 | 0.645 |
| 33422 | 0.581 |
| 33423 | 0.565 |
| 33424 | 0.474 |
| 33425 | 0.379 |
| 33431 | 0.630 |
| 33432 | 0.562 |
| 33433 | 0.545 |
| 33434 | 0.456 |
| 33435 | 0.363 |
| 33441 | 0.520 |
| 33442 | 0.460 |
| 33443 | 0.444 |
| 33444 | 0.371 |
| 33445 | 0.295 |
| 33451 | 0.356 |
| 33452 | 0.306 |
| 33453 | 0.293 |
| 33454 | 0.244 |
| 33455 | 0.192 |
| 33511 | 0.573 |
| 33511 | 0.534 |
| 33512 | 0.524 |
| 33514 | 0.324 |
| 33515 | 0.399 |
| 33521 | 0.521 |
| 33522 | 0.468 |
| 33523 | 0.454 |
| 33524 | 0.401 |
| 33525 | 0.346 |
| 33531 | 0.508 |
| 33532 | 0.452 |
| 33533 | 0.437 |
| 33534 | 0.386 |
| 33535 | 0.333 |
| 33541 | 0.430 |
| 33542 | 0.380 |
| 33543 | 0.368 |
| 33544 | 0.318 |
| 33545 | 0.267 |
| 33551 | 0.312 |
| 33552 | 0.273 |
| 33553 | 0.263 |
| 33554 | 0.216 |
| 33555 | 0.167 |
| 34111 | 0.739 |
| 34112 | 0.704 |
| J 1112 | 0.701 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 34113 | 0.695 |
| 34114 | 0.580 |
| 34115 | 0.461 |
| 34121 | 0.690 |
| 34122 | 0.642 |
| 34123 | 0.629 |
| 34124 | 0.523 |
| 34125 | 0.413 |
| 34131 | 0.678 |
| 34132 | 0.627 |
| 34133 | 0.613 |
| 34134 | 0.509 |
| 34135 | 0.401 |
| 34141 | 0.556 |
| 34142 | 0.512 |
| 34143 | 0.500 |
| 34144 | 0.413 |
| 34145 | 0.324 |
| 34151 | 0.374 |
| 34152 | 0.339 |
| 34153 | 0.330 |
| 34154 | 0.270 |
| 34155 | 0.207 |
| 34133 | 0.717 |
| 34212 | 0.668 |
| 34213 | 0.656 |
| 34213 | 0.550 |
| 34214 | 0.330 |
| 34213 | 0.439 |
| 34221 | 0.653 |
| 34222 | 0.577 |
| 34223 | 0.377 |
| 34224 | 0.479 |
| 34225 | 0.639 |
| 34232 | 0.574 |
| 34233 | 0.557 |
| 34234 | 0.461 |
| 34235 | 0.362 |
| 34241 | 0.525 |
| 34242 | 0.466 |
| 34243 | 0.451 |
| 34244 | 0.373 |
| 34245 | 0.291 |
| 34251 | 0.352 |
| 34252 | 0.304 |
| 34253 | 0.292 |
| 34254 | 0.240 |
| 34255 | 0.186 |
| 34311 | 0.711 |
| 34312 | 0.660 |
| 34313 | 0.646 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 34314 | 0.542 |
| 34315 | 0.434 |
| 34321 | 0.646 |
| 34322 | 0.581 |
| 34323 | 0.564 |
| 34324 | 0.468 |
| 34325 | 0.369 |
| 34331 | 0.630 |
| 34332 | 0.561 |
| 34333 | 0.543 |
| 34334 | 0.450 |
| 34335 | 0.352 |
| 34341 | 0.517 |
| 34342 | 0.455 |
| 34343 | 0.439 |
| 34344 | 0.363 |
| 34345 | 0.284 |
| 34351 | 0.347 |
| 34352 | 0.296 |
| 34353 | 0.282 |
| 34354 | 0.232 |
| 34355 | 0.180 |
| 34411 | 0.654 |
| 34412 | 0.608 |
| 34413 | 0.596 |
| 34414 | 0.506 |
| 34415 | 0.413 |
| 34421 | 0.594 |
| 34422 | 0.535 |
| 34423 | 0.519 |
| 34424 | 0.438 |
| 34425 | 0.436 |
| 34423 | 0.533 |
| 34431 | |
| 34432 | 0.516 |
| | 0.500 |
| 34434 | 0.421 |
| 34435 | 0.338 |
| 34441 | 0.478 |
| 34442 | 0.422 |
| 34443 | 0.407 |
| 34444 | 0.340 |
| 34445 | 0.270 |
| 34451 | 0.326 |
| 34452 | 0.280 |
| 34453 | 0.268 |
| 34454 | 0.219 |
| 34455 | 0.169 |
| 34511 | 0.537 |
| 34512 | 0.502 |
| 34513 | 0.493 |
| 34514 | 0.433 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 34515 | 0.370 |
| 34521 | 0.489 |
| 34522 | 0.440 |
| 34523 | 0.428 |
| 34524 | 0.375 |
| 34525 | 0.321 |
| 34531 | 0.477 |
| 34532 | 0.425 |
| 34533 | 0.411 |
| 34534 | 0.361 |
| 34535 | 0.309 |
| 34541 | 0.400 |
| 34542 | 0.354 |
| 34543 | 0.343 |
| 34544 | 0.294 |
| 34545 | 0.244 |
| 34551 | 0.283 |
| 34552 | 0.248 |
| 34553 | 0.239 |
| 34554 | 0.193 |
| 34555 | 0.145 |
| 35111 | 0.522 |
| 35112 | 0.501 |
| 35113 | 0.495 |
| 35114 | 0.423 |
| 35115 | 0.348 |
| 35121 | 0.487 |
| 35122 | 0.452 |
| 35123 | 0.443 |
| 35124 | 0.379 |
| 35125 | 0.313 |
| 35131 | 0.478 |
| 35132 | 0.440 |
| 35133 | 0.430 |
| 35134 | 0.368 |
| 35135 | 0.304 |
| 35141 | 0.391 |
| 35142 | 0.360 |
| 35143 | 0.352 |
| 35144 | 0.292 |
| 35145 | 0.229 |
| 35151 | 0.261 |
| 35152 | 0.240 |
| 35152 | 0.234 |
| 35154 | 0.177 |
| 35155 | 0.117 |
| 35211 | 0.514 |
| 35212 | 0.479 |
| 35212 | 0.469 |
| 35213 | 0.406 |
| 35214 | 0.339 |
| JJZ1J | 0.337 |



| Haaldh CA-4- (#T Pl A | TIO |
|---------------------------|-------|
| Health State (5L profile) | US |
| 35221 | 0.465 |
| 35222 | 0.416 |
| 35223 | 0.403 |
| 35224 | 0.348 |
| 35225 | 0.290 |
| 35231 | 0.452 |
| 35232 | 0.400 |
| 35233 | 0.387 |
| 35234 | 0.334 |
| 35235 | 0.278 |
| 35241 | 0.372 |
| 35242 | 0.327 |
| 35243 | 0.315 |
| 35244 | 0.264 |
| 35245 | 0.210 |
| 35251 | 0.252 |
| 35252 | 0.217 |
| 35253 | 0.208 |
| 35254 | 0.159 |
| 35255 | 0.108 |
| 35311 | 0.512 |
| 35312 | 0.473 |
| 35312 | 0.463 |
| 35313 | 0.403 |
| 35314 | 0.401 |
| 35313 | 0.337 |
| 35322 | 0.407 |
| 35323 | 0.393 |
| 35324 | 0.340 |
| 35325 | 0.285 |
| 35331 | 0.446 |
| 35332 | 0.391 |
| 35333 | 0.376 |
| 35334 | 0.325 |
| 35335 | 0.272 |
| 35341 | 0.368 |
| 35342 | 0.319 |
| 35343 | 0.307 |
| 35344 | 0.257 |
| 35345 | 0.206 |
| 35351 | 0.250 |
| 35352 | 0.212 |
| 35353 | 0.202 |
| 35354 | 0.155 |
| 35355 | 0.106 |
| 35411 | 0.483 |
| 35412 | 0.450 |
| 35413 | 0.441 |
| 35414 | 0.381 |
| 35415 | 0.318 |
| 35415 | 0.436 |
| 33721 | 0.730 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 35422 | 0.389 |
| 35423 | 0.377 |
| 35424 | 0.325 |
| 35425 | 0.271 |
| 35431 | 0.424 |
| 35432 | 0.374 |
| 35433 | 0.361 |
| 35434 | 0.312 |
| 35435 | 0.260 |
| 35441 | 0.347 |
| 35442 | 0.304 |
| 35443 | 0.293 |
| 35444 | 0.245 |
| 35445 | 0.195 |
| 35451 | 0.231 |
| 35452 | 0.198 |
| 35452 | 0.190 |
| 35454 | 0.144 |
| 35455 | 0.097 |
| 35511 | 0.424 |
| 35512 | 0.403 |
| 35512 | 0.397 |
| 35513 | 0.339 |
| 35515 | 0.339 |
| 35513 | 0.389 |
| 35522 | 0.353 |
| 35523 | 0.333 |
| | 0.344 |
| 35524 | |
| 35525<br>25521 | 0.244 |
| 35531 | 0.380 |
| 35532 | 0.341 |
| 35533 | 0.331 |
| 35534 | 0.284 |
| 35535 | 0.235 |
| 35541 | 0.305 |
| 35542 | 0.273 |
| 35543 | 0.265 |
| 35544 | 0.219 |
| 35545 | 0.172 |
| 35551 | 0.193 |
| 35552 | 0.171 |
| 35553 | 0.165 |
| 35554 | 0.122 |
| 35555 | 0.077 |
| 41111 | 0.824 |
| 41112 | 0.804 |
| 41113 | 0.798 |
| 41114 | 0.663 |
| 41115 | 0.523 |
| 41121 | 0.790 |
| 41122 | 0.755 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 41123 | 0.747 |
| 41124 | 0.620 |
| 41125 | 0.489 |
| 41131 | 0.781 |
| 41132 | 0.744 |
| 41133 | 0.734 |
| 41134 | 0.609 |
| 41135 | 0.480 |
| 41141 | 0.643 |
| 41142 | 0.612 |
| 41143 | 0.604 |
| 41144 | 0.501 |
| 41145 | 0.394 |
| 41151 | 0.436 |
| 41152 | 0.415 |
| 41153 | 0.410 |
| 41154 | 0.339 |
| 41155 | 0.264 |
| 41211 | 0.816 |
| 41212 | 0.782 |
| 41213 | 0.773 |
| 41214 | 0.647 |
| 41215 | 0.516 |
| 41221 | 0.769 |
| 41222 | 0.721 |
| 41223 | 0.708 |
| 41224 | 0.590 |
| 41225 | 0.468 |
| 41223 | 0.468 |
| 41231 | 0.737 |
| 41232 | 0.692 |
| 41233 | 0.692 |
| 41234 | 0.576 |
| 41255 | 0.436 |
| 41242 | 0.581 |
| 41243 | 0.570 |
| 41244 | 0.475 |
| 41245 | 0.376 |
| 41251 | 0.429 |
| 41252 | 0.394 |
| 41253 | 0.386 |
| 41254 | 0.322 |
| 41255 | 0.256 |
| 41311 | 0.814 |
| 41312 | 0.777 |
| 41313 | 0.767 |
| 41314 | 0.643 |
| 41315 | 0.514 |
| 41321 | 0.763 |
| 41322 | 0.712 |
| 41323 | 0.699 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 41324 | 0.583 |
| 41325 | 0.462 |
| 41331 | 0.751 |
| 41332 | 0.696 |
| 41333 | 0.682 |
| 41334 | 0.568 |
| 41335 | 0.450 |
| 41341 | 0.621 |
| 41342 | 0.574 |
| 41343 | 0.561 |
| 41344 | 0.468 |
| 41345 | 0.371 |
| 41351 | 0.427 |
| 41352 | 0.389 |
| 41353 | 0.380 |
| 41354 | 0.318 |
| 41355 | 0.254 |
| 41411 | 0.744 |
| 41412 | 0.711 |
| 41413 | 0.703 |
| 41414 | 0.596 |
| 41415 | 0.485 |
| 41413 | 0.483 |
| 41421 | |
| | 0.653 |
| 41423 | 0.641 |
| 41424 | 0.542 |
| 41425 | 0.439 |
| 41431 | 0.687 |
| 41432 | 0.638 |
| 41433 | 0.625 |
| 41434 | 0.529 |
| 41435 | 0.428 |
| 41441 | 0.572 |
| 41442 | 0.530 |
| 41443 | 0.519 |
| 41444 | 0.437 |
| 41445 | 0.351 |
| 41451 | 0.398 |
| 41452 | 0.366 |
| 41453 | 0.358 |
| 41454 | 0.298 |
| 41455 | 0.236 |
| 41511 | 0.599 |
| 41512 | 0.578 |
| 41513 | 0.573 |
| 41514 | 0.501 |
| 41515 | 0.427 |
| 41521 | 0.565 |
| 41522 | 0.531 |
| 41523 | 0.522 |
| 41524 | 0.459 |
| T1 <i>32</i> T | U.TJ9 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 41525 | 0.393 |
| 41531 | 0.556 |
| 41532 | 0.519 |
| 41533 | 0.509 |
| 41534 | 0.448 |
| 41535 | 0.384 |
| 41541 | 0.470 |
| 41542 | 0.439 |
| 41543 | 0.431 |
| 41544 | 0.372 |
| 41545 | 0.310 |
| 41551 | 0.340 |
| 41552 | 0.320 |
| 41553 | 0.314 |
| 41554 | 0.257 |
| 41555 | 0.198 |
| 41555 | 0.198 |
| 42112 | 0.752 |
| 42112 | 0.743 |
| 42113 | 0.743 |
| 42115 | 0.486 |
| 42121 | 0.738 |
| 42122 | 0.690 |
| 42123 | 0.677 |
| 42124 | 0.560 |
| 42125 | 0.437 |
| 42131 | 0.726 |
| 42132 | 0.674 |
| 42133 | 0.661 |
| 42134 | 0.545 |
| 42135 | 0.425 |
| 42141 | 0.595 |
| 42142 | 0.550 |
| 42143 | 0.539 |
| 42144 | 0.444 |
| 42145 | 0.346 |
| 42151 | 0.399 |
| 42152 | 0.364 |
| 42153 | 0.355 |
| 42153 | 0.333 |
| 42154 | 0.292 |
| 42133 | 0.227 |
| 42211 | |
| | 0.716 |
| 42213 | 0.704 |
| 42214 | 0.586 |
| 42215 | 0.464 |
| 42221 | 0.703 |
| 42222 | 0.641 |
| 42223 | 0.624 |
| 42224 | 0.515 |
| 42225 | 0.402 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 42231 | 0.687 |
| 42232 | 0.622 |
| 42233 | 0.605 |
| 42234 | 0.498 |
| 42235 | 0.386 |
| 42241 | 0.563 |
| 42242 | 0.505 |
| 42243 | 0.490 |
| 42244 | 0.403 |
| 42245 | 0.314 |
| 42251 | 0.377 |
| 42252 | 0.329 |
| 42253 | 0.316 |
| 42254 | 0.262 |
| 42255 | 0.205 |
| 42311 | 0.759 |
| 42312 | 0.707 |
| 42313 | 0.694 |
| 42314 | 0.578 |
| 42315 | 0.459 |
| 42313 | 0.439 |
| 42321 | 0.629 |
| 42323 | 0.612 |
| 42324 | 0.504 |
| 42325 | 0.393 |
| 42331 | 0.678 |
| 42332 | 0.609 |
| 42333 | 0.591 |
| 42334 | 0.486 |
| 42335 | 0.377 |
| 42341 | 0.555 |
| 42342 | 0.494 |
| 42343 | 0.477 |
| 42344 | 0.393 |
| 42345 | 0.306 |
| 42351 | 0.372 |
| 42352 | 0.320 |
| 42353 | 0.307 |
| 42354 | 0.254 |
| 42355 | 0.200 |
| 42411 | 0.694 |
| 42412 | 0.648 |
| 42413 | 0.636 |
| 42413 | 0.636 |
| 42414 | 0.338 |
| 42421 | 0.635 |
| 42422 | 0.575 |
| 42423 | 0.559 |
| 42424 | 0.469 |
| 42425 | 0.376 |
| 42431 | 0.620 |



| TT TIT CO. ( /MT MX ) | TIO. |
|---------------------------|-------|
| Health State (5L profile) | US |
| 42432 | 0.557 |
| 42433 | 0.540 |
| 42434 | 0.452 |
| 42435 | 0.361 |
| 42441 | 0.512 |
| 42442 | 0.455 |
| 42443 | 0.441 |
| 42444 | 0.367 |
| 42445 | 0.291 |
| 42451 | 0.349 |
| 42452 | 0.303 |
| 42453 | 0.291 |
| 42454 | 0.240 |
| 42455 | 0.187 |
| 42511 | 0.562 |
| 42512 | 0.527 |
| 42513 | 0.518 |
| 42514 | 0.455 |
| 42515 | 0.390 |
| 42521 | 0.513 |
| 42522 | 0.465 |
| 42523 | 0.452 |
| 42524 | 0.432 |
| 42525 | 0.341 |
| 42525 | 0.501 |
| 42531 | |
| | 0.449 |
| 42533 | 0.436 |
| 42534 | 0.383 |
| 42535 | 0.329 |
| 42541 | 0.422 |
| 42542 | 0.377 |
| 42543 | 0.365 |
| 42544 | 0.314 |
| 42545 | 0.261 |
| 42551 | 0.303 |
| 42552 | 0.268 |
| 42553 | 0.259 |
| 42554 | 0.210 |
| 42555 | 0.160 |
| 43111 | 0.779 |
| 43112 | 0.741 |
| 43113 | 0.732 |
| 43114 | 0.607 |
| 43115 | 0.478 |
| 43121 | 0.728 |
| 43122 | 0.677 |
| 43123 | 0.663 |
| 43124 | 0.547 |
| 43125 | 0.427 |
| 43131 | 0.715 |
| 43132 | 0.660 |
| T3132 | 0.000 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 43133 | 0.646 |
| 43134 | 0.533 |
| 43135 | 0.414 |
| 43141 | 0.585 |
| 43142 | 0.538 |
| 43143 | 0.525 |
| 43144 | 0.433 |
| 43145 | 0.336 |
| 43151 | 0.391 |
| 43152 | 0.353 |
| 43153 | 0.344 |
| 43154 | 0.282 |
| 43155 | 0.219 |
| 43211 | 0.754 |
| 43212 | 0.703 |
| 43213 | 0.690 |
| 43214 | 0.574 |
| 43215 | 0.454 |
| 43221 | 0.689 |
| 43222 | 0.625 |
| 43223 | 0.608 |
| 43224 | 0.500 |
| 43225 | 0.389 |
| 43223 | 0.673 |
| 43231 | 0.605 |
| 43232 | 0.587 |
| 43233 | 0.482 |
| 43235 | 0.372 |
| 43241 | 0.551 |
| 43242 | 0.489 |
| 43243 | 0.473 |
| 43244 | 0.389 |
| 43245 | 0.301 |
| 43251 | 0.367 |
| 43252 | 0.316 |
| 43253 | 0.302 |
| 43254 | 0.249 |
| 43255 | 0.195 |
| 43311 | 0.748 |
| 43312 | 0.693 |
| 43313 | 0.679 |
| 43314 | 0.566 |
| 43315 | 0.448 |
| 43321 | 0.680 |
| 43322 | 0.612 |
| 43323 | 0.594 |
| 43324 | 0.488 |
| 43325 | 0.379 |
| 43331 | 0.663 |
| 43332 | 0.591 |
| 43333 | 0.573 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 43334 | 0.469 |
| 43335 | 0.362 |
| 43341 | 0.542 |
| 43342 | 0.477 |
| 43343 | 0.461 |
| 43344 | 0.378 |
| 43345 | 0.293 |
| 43351 | 0.361 |
| 43352 | 0.306 |
| 43353 | 0.292 |
| 43354 | 0.241 |
| 43355 | 0.189 |
| 43411 | 0.684 |
| 43412 | 0.635 |
| 43413 | 0.623 |
| 43414 | 0.526 |
| 43415 | 0.426 |
| 43421 | 0.622 |
| 43422 | 0.559 |
| 43423 | 0.543 |
| 43424 | 0.455 |
| 43425 | 0.363 |
| 43431 | 0.606 |
| 43432 | 0.540 |
| 43433 | 0.523 |
| 43434 | 0.437 |
| 43435 | 0.347 |
| 43441 | 0.500 |
| 43442 | 0.440 |
| 43443 | 0.425 |
| 43444 | 0.353 |
| 43445 | 0.279 |
| 43451 | 0.339 |
| 43452 | 0.290 |
| 43453 | 0.277 |
| 43454 | 0.228 |
| 43455 | 0.177 |
| 43511 | 0.554 |
| 43512 | 0.516 |
| 43513 | 0.507 |
| 43514 | 0.445 |
| 43515 | 0.382 |
| 43521 | 0.503 |
| 43522 | 0.452 |
| 43523 | 0.438 |
| 43524 | 0.385 |
| 43525 | 0.330 |
| 43531 | 0.490 |
| 43532 | 0.435 |
| 43533 | 0.421 |
| 43534 | 0.370 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 43535 | 0.318 |
| 43541 | 0.412 |
| 43542 | 0.364 |
| 43543 | 0.352 |
| 43544 | 0.303 |
| 43545 | 0.252 |
| 43551 | 0.295 |
| 43552 | 0.257 |
| 43553 | 0.248 |
| 43554 | 0.201 |
| 43555 | 0.152 |
| 44111 | 0.712 |
| 44112 | 0.678 |
| 44113 | 0.669 |
| 44114 | 0.558 |
| 44115 | 0.442 |
| 44121 | 0.664 |
| 44122 | 0.618 |
| 44123 | 0.605 |
| 44124 | 0.502 |
| 44125 | 0.395 |
| 44131 | 0.653 |
| 44132 | 0.602 |
| 44133 | 0.589 |
| 44134 | 0.488 |
| 44135 | 0.384 |
| 44141 | 0.534 |
| 44142 | 0.490 |
| 44143 | 0.479 |
| 44144 | 0.394 |
| 44145 | 0.306 |
| 44151 | 0.355 |
| 44152 | 0.322 |
| 44153 | 0.313 |
| 44154 | 0.253 |
| 44155 | 0.190 |
| 44133 | 0.190 |
| 44211 | 0.644 |
| 44212 | 0.632 |
| 44214 | 0.529 |
| 44215<br>44221 | 0.422 |
| 44221 | 0.630 |
| | 0.570 |
| 44223 | 0.554 |
| 44224 | 0.459 |
| 44225 | 0.361 |
| 44231 | 0.615 |
| 44232 | 0.551 |
| 44233 | 0.535 |
| 44234 | 0.442 |
| 44235 | 0.346 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 44241 | 0.503 |
| 44242 | 0.446 |
| 44243 | 0.431 |
| 44244 | 0.355 |
| 44245 | 0.276 |
| 44251 | 0.335 |
| 44252 | 0.288 |
| 44253 | 0.276 |
| 44254 | 0.224 |
| 44255 | 0.170 |
| 44311 | 0.686 |
| 44312 | 0.636 |
| 44313 | 0.622 |
| 44314 | 0.521 |
| 44315 | 0.417 |
| 44321 | 0.622 |
| 44322 | 0.558 |
| 44323 | 0.541 |
| 44324 | 0.449 |
| 44325 | 0.352 |
| 44331 | 0.606 |
| 44332 | 0.539 |
| 44333 | 0.521 |
| 44334 | 0.430 |
| 44335 | 0.336 |
| 44341 | 0.496 |
| 44342 | 0.435 |
| 44343 | 0.419 |
| 44344 | 0.345 |
| 44345 | 0.268 |
| 44351 | 0.330 |
| 44352 | 0.279 |
| 44353 | 0.266 |
| 44354 | 0.217 |
| 44355 | 0.165 |
| 44411 | 0.631 |
| 44412 | 0.586 |
| 44413 | 0.574 |
| 44414 | 0.487 |
| 44415 | 0.396 |
| 44421 | 0.572 |
| 44422 | 0.514 |
| 44423 | 0.499 |
| 44424 | 0.419 |
| 44425 | 0.337 |
| 44431 | 0.558 |
| 44432 | 0.496 |
| 44433 | 0.480 |
| 44434 | 0.403 |
| 44435 | 0.322 |
| 44441 | 0.458 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 44442 | 0.403 |
| 44443 | 0.389 |
| 44444 | 0.323 |
| 44445 | 0.255 |
| 44451 | 0.309 |
| 44452 | 0.264 |
| 44453 | 0.252 |
| 44454 | 0.204 |
| 44455 | 0.154 |
| 44511 | 0.518 |
| 44512 | 0.485 |
| 44513 | 0.476 |
| 44514 | 0.416 |
| 44515 | 0.353 |
| 44521 | 0.471 |
| 44522 | 0.424 |
| 44523 | 0.411 |
| 44524 | 0.360 |
| 44525 | 0.306 |
| 44531 | 0.460 |
| 44532 | 0.409 |
| 44533 | 0.395 |
| 44534 | 0.346 |
| 44535 | 0.294 |
| 44541 | 0.382 |
| 44542 | 0.338 |
| 44543 | 0.327 |
| 44544 | 0.279 |
| 44545 | 0.229 |
| 44551 | 0.266 |
| 44552 | 0.233 |
| 44553 | 0.224 |
| 44554 | 0.178 |
| 44555 | 0.178 |
| 45111 | 0.502 |
| 45112 | 0.302 |
| 45112 | 0.476 |
| 45115 | 0.476 |
| 45114 | 0.330 |
| 45121<br>45122 | 0.468 |
| 45122 | 0.434 |
| 45123 | 0.425 |
| 45124 | 0.362 |
| 45125 | 0.296 |
| 45131 | 0.459 |
| 45132 | 0.422 |
| 45133 | 0.412 |
| 45134 | 0.351 |
| 45135 | 0.287 |
| 45141 | 0.373 |
| 45142 | 0.342 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 45143 | 0.334 |
| 45144 | 0.275 |
| 45145 | 0.213 |
| 45151 | 0.243 |
| 45152 | 0.223 |
| 45153 | 0.217 |
| 45154 | 0.160 |
| 45155 | 0.101 |
| 45211 | 0.495 |
| 45212 | 0.460 |
| 45213 | 0.452 |
| 45214 | 0.388 |
| 45215 | 0.322 |
| 45221 | 0.447 |
| 45222 | 0.399 |
| 45223 | 0.387 |
| 45224 | 0.332 |
| 45225 | 0.274 |
| 45231 | 0.435 |
| 45232 | 0.384 |
| 45233 | 0.370 |
| 45234 | 0.318 |
| 45235 | 0.263 |
| 45241 | 0.355 |
| 45242 | 0.311 |
| 45243 | 0.299 |
| 45244 | 0.248 |
| 45245 | 0.195 |
| 45251 | 0.235 |
| 45252 | 0.201 |
| 45253 | 0.193 |
| 45254 | 0.144 |
| 45255 | 0.093 |
| 45311 | 0.493 |
| 45312 | 0.455 |
| 45313 | 0.446 |
| 45314 | 0.384 |
| 45315 | 0.320 |
| 45321 | 0.441 |
| 45322 | 0.390 |
| 45323 | 0.377 |
| 45324 | 0.324 |
| 45325 | 0.269 |
| 45331 | 0.429 |
| 45332 | 0.374 |
| 45333 | 0.360 |
| 45334 | 0.309 |
| 45335 | 0.257 |
| 45341 | 0.350 |
| 45342 | 0.303 |
| 45343 | 0.291 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 45344 | 0.242 |
| 45345 | 0.191 |
| 45351 | 0.233 |
| 45352 | 0.196 |
| 45353 | 0.187 |
| 45354 | 0.140 |
| 45355 | 0.091 |
| 45411 | 0.464 |
| 45412 | 0.432 |
| 45413 | 0.424 |
| 45414 | 0.364 |
| 45415 | 0.302 |
| 45421 | 0.418 |
| 45422 | 0.373 |
| 45423 | 0.361 |
| 45424 | 0.310 |
| 45425 | 0.256 |
| 45431 | 0.407 |
| 45432 | 0.358 |
| 45433 | 0.345 |
| 45434 | 0.296 |
| 45435 | 0.245 |
| 45441 | 0.243 |
| 45441 | |
| | 0.288 |
| 45443 | 0.277 |
| 45444 | 0.229 |
| 45445 | 0.180 |
| 45451 | 0.215 |
| 45452 | 0.183 |
| 45453 | 0.175 |
| 45454 | 0.129 |
| 45455 | 0.082 |
| 45511 | 0.406 |
| 45512 | 0.386 |
| 45513 | 0.380 |
| 45514 | 0.323 |
| 45515 | 0.263 |
| 45521 | 0.372 |
| 45522 | 0.337 |
| 45523 | 0.328 |
| 45524 | 0.280 |
| 45525 | 0.229 |
| 45531 | 0.363 |
| 45532 | 0.325 |
| 45533 | 0.316 |
| 45534 | 0.269 |
| 45535 | 0.220 |
| 45541 | 0.289 |
| 45542 | 0.258 |
| 45543 | 0.250 |
| 45544 | 0.205 |
| L 43344 | 0.203 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 45545 | 0.158 |
| 45551 | 0.177 |
| 45552 | 0.156 |
| 45553 | 0.150 |
| 45554 | 0.108 |
| 45555 | 0.064 |
| 51111 | 0.442 |
| 51112 | 0.429 |
| 51113 | 0.426 |
| 51114 | 0.349 |
| 51115 | 0.268 |
| 51121 | 0.416 |
| 51122 | 0.396 |
| 51123 | 0.391 |
| 51124 | 0.318 |
| 51125 | 0.242 |
| 51131 | 0.409 |
| 51132 | 0.388 |
| 51133 | 0.382 |
| 51134 | 0.310 |
| 51135 | 0.235 |
| 51141 | 0.318 |
| 51142 | 0.300 |
| 51143 | 0.295 |
| 51144 | 0.227 |
| 51145 | 0.156 |
| 51151 | 0.181 |
| 51152 | 0.168 |
| 51153 | 0.165 |
| 51154 | 0.102 |
| 51155 | 0.037 |
| 51211 | 0.442 |
| 51212 | 0.422 |
| 51213 | 0.417 |
| 51214 | 0.344 |
| 51215 | 0.268 |
| 51221 | 0.409 |
| 51222 | 0.377 |
| 51223 | 0.368 |
| 51224 | 0.303 |
| 51225 | 0.235 |
| 51231 | 0.400 |
| 51232 | 0.365 |
| 51232 | 0.366 |
| | 0.336 |
| 51234 | |
| 51235 | 0.226 |
| 51241 | 0.313 |
| 51242 | 0.284 |
| 51243 | 0.276 |
| 51244 | 0.215 |
| 51245 | 0.150 |



| Health State (5L profile) | US |
|---------------------------|-------|
| 51251 | 0.181 |
| 51252 | 0.161 |
| 51253 | 0.156 |
| 51254 | 0.097 |
| 51255 | 0.036 |
| 51311 | 0.442 |
| 51312 | 0.421 |
| 51313 | 0.415 |
| 51314 | 0.343 |
| 51315 | 0.268 |
| 51321 | 0.407 |
| 51322 | 0.372 |
| 51323 | 0.363 |
| 51324 | 0.299 |
| 51325 | 0.233 |
| 51331 | 0.398 |
| 51332 | 0.360 |
| 51333 | 0.350 |
| 51334 | 0.288 |
| 51335 | 0.224 |
| 51341 | 0.311 |
| 51342 | 0.280 |
| 51343 | 0.272 |
| 51344 | 0.272 |
| 51345 | 0.211 |
| 51351 | 0.149 |
| 51352 | 0.160 |
| 51353 | 0.154 |
| 51354 | 0.096 |
| 51355 | 0.036 |
| 51411 | 0.410 |
| 51412 | 0.391 |
| 51413 | 0.386 |
| 51414 | 0.317 |
| 51415 | 0.245 |
| 51421 | 0.378 |
| 51422 | 0.347 |
| 51423 | 0.340 |
| 51424 | 0.277 |
| 51425 | 0.213 |
| 51431 | 0.369 |
| 51432 | 0.337 |
| 51433 | 0.328 |
| 51434 | 0.268 |
| 51435 | 0.205 |
| 51441 | 0.285 |
| 51442 | 0.258 |
| 51443 | 0.251 |
| 51444 | 0.193 |
| 51445 | 0.132 |
| 51451 | 0.158 |
| • | |



| Health State (5L profile) | US |
|---------------------------|--------|
| 51452 | 0.140 |
| 51453 | 0.135 |
| 51454 | 0.080 |
| 51455 | 0.023 |
| 51511 | 0.344 |
| 51512 | 0.331 |
| 51513 | 0.327 |
| 51514 | 0.264 |
| 51515 | 0.199 |
| 51521 | 0.318 |
| 51522 | 0.297 |
| 51523 | 0.292 |
| 51524 | 0.233 |
| 51525 | 0.173 |
| 51531 | 0.311 |
| 51532 | 0.289 |
| 51533 | 0.283 |
| 51534 | 0.226 |
| 51535 | 0.166 |
| 51535 | 0.232 |
| 51542 | 0.232 |
| 51543 | 0.213 |
| | 0.208 |
| 51544 | |
| 51545 | 0.099 |
| 51551 | 0.112 |
| 51552 | 0.099 |
| 51553 | 0.096 |
| 51554 | 0.047 |
| 51555 | -0.003 |
| 52111 | 0.413 |
| 52112 | 0.392 |
| 52113 | 0.387 |
| 52114 | 0.314 |
| 52115 | 0.238 |
| 52121 | 0.379 |
| 52122 | 0.346 |
| 52123 | 0.338 |
| 52124 | 0.272 |
| 52125 | 0.204 |
| 52131 | 0.371 |
| 52132 | 0.335 |
| 52133 | 0.325 |
| 52134 | 0.262 |
| 52135 | 0.196 |
| 52141 | 0.283 |
| 52142 | 0.253 |
| 52143 | 0.246 |
| 52144 | 0.184 |
| 52145 | 0.120 |
| 52151 | 0.151 |
| 52152 | 0.131 |



| Health State (5L profile) | US |
|---------------------------|--------|
| 52153 | 0.126 |
| 52154 | 0.068 |
| 52155 | 0.007 |
| 52211 | 0.406 |
| 52212 | 0.373 |
| 52213 | 0.364 |
| 52214 | 0.299 |
| 52215 | 0.231 |
| 52221 | 0.359 |
| 52222 | 0.313 |
| 52223 | 0.301 |
| 52224 | 0.244 |
| 52225 | 0.185 |
| 52231 | 0.347 |
| 52232 | 0.298 |
| 52233 | 0.285 |
| 52234 | 0.230 |
| 52235 | 0.173 |
| 52241 | 0.266 |
| 52242 | 0.223 |
| 52243 | 0.212 |
| 52244 | 0.159 |
| 52245 | 0.104 |
| 52251 | 0.144 |
| 52252 | 0.112 |
| 52253 | 0.112 |
| 52254 | 0.052 |
| 52255 | -0.001 |
| 52311 | 0.404 |
| 52312 | 0.368 |
| 52313 | 0.358 |
| 52314 | 0.295 |
| 52315 | 0.230 |
| 52321 | 0.354 |
| 52322 | 0.305 |
| 52323 | 0.292 |
| 52324 | 0.237 |
| 52325 | 0.180 |
| 52331 | 0.341 |
| 52332 | 0.289 |
| 52333 | 0.275 |
| 52334 | 0.222 |
| 52335 | 0.167 |
| 52341 | 0.262 |
| 52342 | 0.216 |
| 52343 | 0.204 |
| 52344 | 0.153 |
| 52345 | 0.100 |
| 52351 | 0.143 |
| 52352 | 0.107 |
| 52353 | 0.097 |



| Harlah Chata (FT Pla) | US |
|---------------------------|--------|
| Health State (5L profile) | |
| 52354 | 0.049 |
| 52355 | -0.002 |
| 52411 | 0.374 |
| 52412 | 0.344 |
| 52413 | 0.336 |
| 52414 | 0.274 |
| 52415 | 0.210 |
| 52421 | 0.330 |
| 52422 | 0.286 |
| 52423 | 0.275 |
| 52424 | 0.221 |
| 52425 | 0.165 |
| 52431 | 0.319 |
| 52432 | 0.272 |
| 52433 | 0.259 |
| 52434 | 0.208 |
| 52435 | 0.154 |
| 52441 | 0.240 |
| 52442 | 0.200 |
| 52443 | 0.189 |
| 52444 | 0.140 |
| 52445 | 0.088 |
| 52451 | 0.123 |
| 52452 | 0.092 |
| 52453 | 0.084 |
| 52454 | 0.037 |
| 52454 | -0.012 |
| 52433 | 0.314 |
| 52511 | 0.294 |
| 52513 | 0.289 |
| 52514 | 0.230 |
| 52515 | 0.170 |
| 52521 | 0.280 |
| 52522 | 0.248 |
| 52523 | 0.239 |
| 52524 | 0.189 |
| 52525 | 0.136 |
| 52531 | 0.272 |
| 52532 | 0.236 |
| 52533 | 0.227 |
| 52534 | 0.178 |
| 52535 | 0.128 |
| 52541 | 0.196 |
| 52542 | 0.167 |
| 52543 | 0.159 |
| 52544 | 0.112 |
| 52545 | 0.064 |
| 52551 | 0.083 |
| 52552 | 0.062 |
| 52553 | 0.057 |
| 52554 | 0.013 |
| | 0.015 |



| Health State (5L profile) | US |
|---------------------------|--------|
| 52555 | -0.032 |
| 53111 | 0.407 |
| 53112 | 0.385 |
| 53113 | 0.379 |
| 53114 | 0.307 |
| 53115 | 0.232 |
| 53121 | 0.372 |
| 53122 | 0.336 |
| 53123 | 0.327 |
| 53124 | 0.263 |
| 53125 | 0.197 |
| 53131 | 0.363 |
| 53132 | 0.324 |
| 53133 | 0.314 |
| 53134 | 0.252 |
| 53135 | 0.188 |
| 53141 | 0.276 |
| 53142 | 0.244 |
| 53143 | 0.236 |
| 53144 | 0.176 |
| 53145 | 0.113 |
| 53151 | 0.145 |
| 53152 | 0.124 |
| 53153 | 0.118 |
| 53154 | 0.061 |
| 53155 | 0.001 |
| 53211 | 0.398 |
| 53212 | 0.363 |
| 53212 | 0.353 |
| 53213 | 0.333 |
| 53215 | 0.224 |
| 53213 | 0.349 |
| 53222 | 0.349 |
| 53222 | |
| | 0.287 |
| 53224 | 0.232 |
| 53225 | 0.175 |
| 53231 | 0.337 |
| 53232 | 0.284 |
| 53233 | 0.271 |
| 53234 | 0.218 |
| 53235 | 0.162 |
| 53241 | 0.257 |
| 53242 | 0.211 |
| 53243 | 0.199 |
| 53244 | 0.148 |
| 53245 | 0.094 |
| 53251 | 0.137 |
| 53252 | 0.102 |
| 53253 | 0.092 |
| 53254 | 0.043 |
| 53255 | -0.008 |



| Health State (5L profile) | US |
|---------------------------|--------|
| 53311 | 0.396 |
| 53312 | 0.357 |
| 53313 | 0.347 |
| 53314 | 0.286 |
| 53315 | 0.222 |
| 53321 | 0.343 |
| 53322 | 0.291 |
| 53323 | 0.277 |
| 53324 | 0.224 |
| 53325 | 0.169 |
| 53331 | 0.330 |
| 53332 | 0.275 |
| 53333 | 0.260 |
| 53334 | 0.209 |
| 53335 | 0.156 |
| 53341 | 0.252 |
| 53342 | 0.203 |
| 53343 | 0.191 |
| 53344 | 0.141 |
| 53345 | 0.090 |
| 53351 | 0.135 |
| 53352 | 0.096 |
| 53353 | 0.086 |
| 53354 | 0.039 |
| 53355 | -0.010 |
| 53411 | 0.367 |
| 53412 | 0.334 |
| 53412 | 0.325 |
| 53413 | 0.323 |
| 53414 | 0.203 |
| 53413 | 0.203 |
| 53421 | 0.320 |
| 53423 | 0.261 |
| 53424 | 0.210 |
| 53425 | 0.156 |
| 53431 | 0.308 |
| 53432 | 0.259 |
| 53433 | 0.246 |
| 53434 | 0.196 |
| 53435 | 0.144 |
| 53441 | 0.232 |
| 53442 | 0.188 |
| 53443 | 0.177 |
| 53444 | 0.129 |
| 53445 | 0.079 |
| 53451 | 0.116 |
| 53452 | 0.083 |
| 53453 | 0.074 |
| 53454 | 0.028 |
| 53455 | -0.019 |
| 53511 | 0.308 |



| Haaldh Chada (#1 @1.\ | US |
|---------------------------|--------|
| Health State (5L profile) | |
| 53512 | 0.287 |
| 53513 | 0.281 |
| 53514 | 0.224 |
| 53515 | 0.164 |
| 53521 | 0.273 |
| 53522 | 0.238 |
| 53523 | 0.229 |
| 53524 | 0.180 |
| 53525 | 0.129 |
| 53531 | 0.264 |
| 53532 | 0.226 |
| 53533 | 0.216 |
| 53534 | 0.169 |
| 53535 | 0.120 |
| 53541 | 0.189 |
| 53542 | 0.158 |
| 53543 | 0.149 |
| 53544 | 0.104 |
| 53545 | 0.057 |
| 53551 | 0.077 |
| 53552 | 0.055 |
| 53552 | 0.049 |
| 53553 | 0.006 |
| 53555 | -0.038 |
| 55555 | 0.368 |
| 54111 | 0.368 |
| | 0.348 |
| 54113 | |
| 54114 | 0.273 |
| 54115 | 0.200 |
| 54121 | 0.335 |
| 54122 | 0.303 |
| 54123 | 0.295 |
| 54124 | 0.232 |
| 54125 | 0.167 |
| 54131 | 0.327 |
| 54132 | 0.292 |
| 54133 | 0.283 |
| 54134 | 0.222 |
| 54135 | 0.159 |
| 54141 | 0.242 |
| 54142 | 0.213 |
| 54143 | 0.206 |
| 54144 | 0.147 |
| 54145 | 0.086 |
| 54151 | 0.114 |
| 54152 | 0.094 |
| 54153 | 0.089 |
| 54154 | 0.034 |
| 54155 | -0.024 |
| 54211 | 0.361 |
| 54211 | 0.330 |
| J7414 | 0.550 |



| Health State (5L profile) | US |
|---------------------------|--------|
| 54213 | 0.321 |
| 54214 | 0.259 |
| 54215 | 0.194 |
| 54221 | 0.316 |
| 54222 | 0.271 |
| 54223 | 0.259 |
| 54224 | 0.205 |
| 54225 | 0.149 |
| 54231 | 0.305 |
| 54232 | 0.256 |
| 54233 | 0.244 |
| 54234 | 0.192 |
| 54235 | 0.138 |
| 54241 | 0.226 |
| 54242 | 0.184 |
| 54243 | 0.173 |
| 54244 | 0.123 |
| 54245 | 0.071 |
| 54251 | 0.107 |
| 54252 | 0.076 |
| 54253 | 0.068 |
| 54253 | 0.008 |
| 54254 | -0.030 |
| 54255 | 0.360 |
| 54312 | 0.325 |
| 54313 | 0.316 |
| 54314 | 0.256 |
| 54315 | 0.193 |
| 54321 | 0.311 |
| 54322 | 0.263 |
| 54323 | 0.251 |
| 54324 | 0.198 |
| 54325 | 0.144 |
| 54331 | 0.299 |
| 54332 | 0.248 |
| 54333 | 0.234 |
| 54334 | 0.184 |
| 54335 | 0.132 |
| 54341 | 0.222 |
| 54342 | 0.177 |
| 54343 | 0.166 |
| 54344 | 0.117 |
| 54345 | 0.067 |
| 54351 | 0.106 |
| 54352 | 0.071 |
| 54353 | 0.062 |
| 54354 | 0.016 |
| 54355 | -0.032 |
| 54335 | 0.332 |
| 54412 | 0.332 |
| 54413 | 0.303 |
| J <del>11</del> 13 | 0.293 |



| Haddle CA-4- (FT PL.) | FIG |
|---------------------------|--------|
| Health State (5L profile) | US |
| 54414 | 0.236 |
| 54415 | 0.175 |
| 54421 | 0.289 |
| 54422 | 0.246 |
| 54423 | 0.235 |
| 54424 | 0.185 |
| 54425 | 0.132 |
| 54431 | 0.278 |
| 54432 | 0.232 |
| 54433 | 0.220 |
| 54434 | 0.172 |
| 54435 | 0.121 |
| 54441 | 0.202 |
| 54442 | 0.163 |
| 54443 | 0.153 |
| 54444 | 0.106 |
| 54445 | 0.057 |
| 54451 | 0.088 |
| 54452 | 0.059 |
| 54453 | 0.051 |
| 54454 | 0.006 |
| 54455 | -0.040 |
| 54455 | 0.276 |
| 54511 | 0.276 |
| | 0.257 |
| 54513 | |
| 54514 | 0.197 |
| 54515 | 0.140 |
| 54521 | 0.243 |
| 54522 | 0.212 |
| 54523 | 0.204 |
| 54524 | 0.156 |
| 54525 | 0.106 |
| 54531 | 0.235 |
| 54532 | 0.201 |
| 54533 | 0.192 |
| 54534 | 0.146 |
| 54535 | 0.098 |
| 54541 | 0.162 |
| 54542 | 0.134 |
| 54543 | 0.126 |
| 54544 | 0.082 |
| 54545 | 0.037 |
| 54551 | 0.053 |
| 54552 | 0.033 |
| 54553 | 0.027 |
| 54554 | -0.013 |
| 54555 | -0.055 |
| 54555 | 0.247 |
| 55112 | 0.234 |
| 55113 | 0.234 |
| 55114 | 0.230 |
| 33114 | 0.107 |



| Health State (5L profile) | US |
|---------------------------|--------|
| 55115 | 0.102 |
| 55121 | 0.221 |
| 55122 | 0.200 |
| 55123 | 0.195 |
| 55124 | 0.136 |
| 55125 | 0.076 |
| 55131 | 0.214 |
| 55132 | 0.192 |
| 55133 | 0.186 |
| 55134 | 0.129 |
| 55135 | 0.069 |
| 55141 | 0.135 |
| 55142 | 0.116 |
| 55143 | 0.111 |
| 55144 | 0.057 |
| 55145 | 0.002 |
| 55151 | 0.016 |
| 55152 | 0.003 |
| 55153 | -0.001 |
| 55154 | -0.050 |
| 55155 | -0.100 |
| 55211 | 0.247 |
| 55212 | 0.227 |
| 55212 | 0.227 |
| 55214 | 0.163 |
| 55215 | 0.103 |
| 55221 | 0.214 |
| 55222 | 0.181 |
| 55223 | 0.173 |
| 55224 | 0.122 |
| 55225 | 0.069 |
| 55231 | 0.205 |
| 55232 | 0.170 |
| 55233 | 0.160 |
| 55234 | 0.111 |
| 55235 | 0.060 |
| 55241 | 0.129 |
| 55242 | 0.100 |
| 55243 | 0.092 |
| 55244 | 0.045 |
| 55245 | -0.004 |
| 55251 | 0.015 |
| 55252 | -0.005 |
| 55253 | -0.010 |
| 55254 | -0.054 |
| 55255 | -0.100 |
| 55311 | 0.247 |
| 55312 | 0.226 |
| 55313 | 0.220 |
| 55314 | 0.162 |
| 55315 | 0.102 |
| 33313 | 0.102 |



| Health State (5L profile) | US |
|---------------------------|--------|
| 55321 | 0.212 |
| 55322 | 0.176 |
| 55323 | 0.167 |
| 55324 | 0.118 |
| 55325 | 0.067 |
| 55331 | 0.203 |
| 55332 | 0.164 |
| 55333 | 0.154 |
| 55334 | 0.107 |
| 55335 | 0.058 |
| 55341 | 0.128 |
| 55342 | 0.096 |
| 55343 | 0.088 |
| 55344 | 0.042 |
| 55345 | -0.005 |
| 55351 | 0.015 |
| 55352 | -0.006 |
| 55353 | -0.012 |
| 55354 | -0.055 |
| 55355 | -0.100 |
| 55411 | 0.224 |
| 55412 | 0.206 |
| 55413 | 0.201 |
| 55414 | 0.146 |
| 55415 | 0.089 |
| 55421 | 0.192 |
| 55422 | 0.162 |
| 55423 | 0.162 |
| | 0.134 |
| 55424 | |
| 55425 | 0.057 |
| 55431 | 0.184 |
| 55432 | 0.151 |
| 55433 | 0.142 |
| 55434 | 0.096 |
| 55435 | 0.049 |
| 55441 | 0.111 |
| 55442 | 0.084 |
| 55443 | 0.077 |
| 55444 | 0.033 |
| 55445 | -0.012 |
| 55451 | 0.002 |
| 55452 | -0.016 |
| 55453 | -0.021 |
| 55454 | -0.061 |
| 55455 | -0.103 |
| 55511 | 0.178 |
| 55512 | 0.165 |
| 55513 | 0.162 |
| 55514 | 0.113 |
| 55515 | 0.063 |
| 55521 | 0.152 |
| | , |



| Health State (5L profile) | US |
|---------------------------|--------|
| 55522 | 0.132 |
| 55523 | 0.127 |
| 55524 | 0.083 |
| 55525 | 0.037 |
| 55531 | 0.145 |
| 55532 | 0.124 |
| 55533 | 0.118 |
| 55534 | 0.075 |
| 55535 | 0.030 |
| 55541 | 0.078 |
| 55542 | 0.060 |
| 55543 | 0.055 |
| 55544 | 0.015 |
| 55545 | -0.026 |
| 55551 | -0.024 |
| 55552 | -0.037 |
| 55553 | -0.040 |
| 55554 | -0.074 |
| 55555 | -0.109 |



## 9.10. Abbreviations

| Abbreviation | Definition |
|---|---|
| ADL | Activities of daily living |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| APMP | Abuse Potential Monitoring Plan |
| AST | Aspartate aminotransferase |
| BLQ | Below limit of quantification |
| BUN | Blood urea nitrogen |
| C <sub>max</sub> | Maximum observed plasma concentration |
| cAMP | Cyclic adenosine monophosphate |
| CFR | Code of Federal Regulations |
| CI | Confidence interval |
| CGI-I | Clinical Global Impressions - Improvement |
| CGI-S | Clinical Global Impressions – Severity of Illness |
| CIOMS | Council for International Organizations of Medical Sciences |
| COMT | Catechol-O-methyltransferase |
| CONSORT | Consolidated Standards of Reporting Trials |
| СРК | Creatine phosphokinase |
| C-QT | Concentration-QT |
| CSR | Clinical study report |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CVL-751 | Tavapadon |
| D1Rs | Dopamine D1-like receptors |
| D2/D3R | Dopamine D2 and D3 receptor subtypes |
| DNA | Deoxyribonucleic acid |
| DSM-5 | Diagnostic and Statistical Manual of Mental Disorders, 5th Edition |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| ЕОТ | End of treatment |
| EQ-5D-5L | EuroQol 5 Dimension 5 Level |
| ESAMs | Events subject to additional monitoring |



| ESS | Epworth Sleepiness Scale |
|---|---|
| ET | Early termination |
| EU | European Union |
| EudraCT | European Union Drug Regulating Authorities Clinical Trials Database |
| FAS | Full analysis set |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GGT | Gamma-glutamyl transferase |
| HbsAg | Hepatitis B surface antigen |
| HCV | Hepatitis C virus |
| HDL-C | High-density lipoprotein cholesterol |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | Human immunodeficiency virus |
| ICD | Impulsive control disorder |
| ICE | Intercurrent event |
| ICF | Informed consent form |
| ICH | International Conference on Harmonisation |
| IEC | Independent Ethics Committee |
| IMP | Investigational medicinal product |
| IOP | Intraocular pressure |
| IRB | Institutional Review Board |
| ITT | Intent-to-treat |
| IVRS/IWRS | Interactive Voice Response System/Interactive Web Response System |
| LDL-C | Low-density lipoprotein cholesterol |
| L-Dopa | Levodopa |
| LLN | Lower limit of normal |
| LLOQ | Lower limit of quantification |
| LSMean | Least square mean |
| MAO | Monoamine oxidase |
| MAO-B | Monoamine oxidase B |
| MAR | Missing at random |
| MCAR | Missing completely at random |
| MNAR | Missing not at random |
| MCV | Mean corpuscular volume |



| MDS-UPDRS | Movement Disorder Society – Unified Parkinson's Disease Rating Scale |
|---|---|
| MedDRA | Medical Dictionary for Regulatory Activities |
| MHIs | Medication handling irregularities |
| mITT | Modified intent-to-treat |
| MMRM | Mixed Model for Repeated Measures |
| MoCA | Montreal Cognitive Assessment |
| PD | Parkinson's disease |
| PDQ-39 | 39-Item Parkinson's Disease Questionnaire |
| PGIC | Patient Global Impression of Change |
| PK | Pharmacokinetic |
| QD | Once daily |
| QTcF | QT interval corrected for heart rate by Fridericia's formula |
| QUIP-RS | Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease – Rating Scale |
| RBC | Red blood cell |
| RNA | Ribonucleic acid |
| SAE | Serious adverse event |
| TEAE | Treatment-emergent adverse event |
| THC | Tetrahydrocannabinol |
| TQT | Thorough QT |
| TSH | Thyroid-stimulating hormone |
| ULN | Upper limit of normal |
| VAS | Visual analog scale |
| WBC | White blood cell |